Emulation of the effects of oral semaglutide on cardiovascular outcomes in individuals with type 2 diabetes: PIONEER6 trial

NCT06659679

23<sup>rd</sup> April 2025

# 1. Title Page

| Title | Emulation of the effects of oral semaglutide on cardiovascular outcomes in individuals with type 2 diabetes: PIONEER6 trial (NCT02692716) |
|---|---|
| Research question & Objectives | The PIONEER6 trial aims to evaluate the effect of oral semaglutide versus placebo on |
| | MACE outcomes (CV death, nonfatal MI or nonfatal stroke) among individuals with |
| | type 2 diabetes. |
| Protocol version | Version 4 |
| Last update date | 23st April 2025 |
| Contributors | Primary investigator contact information: |
| | Dr. Shirley Wang |
| | Swang1@bwh.harvard.edu |
| | Contributor names: |
| | Shirley Wang, Sushama Kattinakere Sreedhara, Elyse DiCesare |
| | Sushama implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform. |
| Study registration | Site: <text></text> |
| | Identifier: <text></text> |
| Sponsor | Organization: Food and Drug Administration |
| | Contact: Dianne Paraoan |
| | dianne.paraoan@fda.hhs.gov |
| Conflict of interest | Dr. Wang has consulted for Veracity Healthcare Analytics, Exponent Inc, and MITRE |
| | and FFRDC for Centers for Medicare and Medicaid for unrelated work. |

# Table of contents

| 1. Title Page | 1 |
|---|---|
| 2. Abstract | 3 |
| 3. Amendments and updates | 3 |
| 4. Rationale and background | 5 |
| 5. Research question and objectives | |
| Table 1 Primary and secondary research questions and objective | |
| 6. Research methods | |
| 6.1. Study design | 7 |
| 6.2. Study design diagram | 8 |
| 6.3. Setting | 9 |
| 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population | |
| 6.3.2 Context and rationale for study inclusion criteria: | |
| 6.3.3 Context and rationale for study exclusion criteria | |
| 6.4. Variables | |
| 6.4.1 Context and rationale for exposure(s) of interest | |
| 6.4.2 Context and rationale for outcome(s) of interest | |
| 6.4.3 Context and rationale for follow up | |
| Table 2. Operational Definitions of Follow Up | |
| 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) | |
| Table 3. Operational Definitions of Covariates | |
| 6.5. Data analysis | |
| Table 4. Primary, secondary, and subgroup analysis specification | |
| Table 5. Sensitivity analyses – rationale, strengths and limitations | |
| 6.6. Data sources | |
| 7.6.1 Context and rationale for data sources | |
| Table 6. Metadata about data sources and software | |
| 6.7. Data management | |
| 6.8. Quality control | |
| 6.9. Study size and feasibility | |
| 7. Limitation of the methods | 31 |
| 8. Protection of human subjects | 31 |
| 9. References | |
| 10. Appendices | |
| 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment | |
| 2 Code algorithms. | |
| 3 Flowchart for cohort assembly | |
| 4 1st feasibility assessment | 32 |

| 5 2nd feasibility assessment | 32 |
|--------------------------------------------------------|----|
| 6 Balance Assessment - PS Distribution and C-Statistic | 32 |
| 7 Balance Assessment - Table 1 | 32 |

### 2. Abstract

This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the PIONEER6 trial described below. Although many features of the trial cannot be directly replicated in healthcare claims data, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization cannot be emulated in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The PIONEER6 trial, is a is a non-inferiority trial to evaluate the effects of oral semaglutide versus placebo in terms of cardiovascular safety (CV death, nonfatal MI, or nonfatal stroke) in patients with type 2 diabetes.

The database study designed to emulate PIONEER6 will be a new-user active comparative study, where we compare the effect of oral semaglutide versus sitagliptin on MACE outcome among patients with T2DM. Sitagliptin was selected to act as an active-comparator proxy for placebo. Sitagliptin and the class of dipeptidyl peptidase-4 (DPP-4) inhibitors have been demonstrated not to have an effect on MACE in a series of RCTs, and they are used in similar stages of disease/line of therapy as semaglutide, as well as being similarly costly.

The study will use three data sources: Optum Clinformatics, Merative Marketscan, and Medicare.

Optum: Study period between 20<sup>th</sup> Sept 2019 – 29<sup>th</sup> February 2024 Marketscan: Study period between 20<sup>th</sup> Sept 2019 - 31<sup>st</sup> Dec 2022 Medicare: Study period between 20<sup>th</sup> Sept 2019 – 31<sup>st</sup> Dec 2020

# 3. Amendments and updates

| Version date | Version number | Section of protocol Amendment or update | | Reason |
|---|---|---|---|---|
| 19 <sup>th</sup> Aug 2024 | 2 | 6.4, 6.5, Table 2-4,<br>appendices 5-8 | Inclusion Exclusion Criteria: Adding TIRZEPATIDE to the list of other GLP1, Stroke definition to include only Ischemic stroke Outcome: | Better algorithms for exclusion criteria and outcome |

| | | | Stroke definition to include only Ischemic stroke Added covariates for PS adjustment | To operationally define covariates and adjust for confounding Pre-planned data check |
|---|---|---|---|---|
| | | | Power and feasibility (balance checks) post PS matching added in appendices 5, 6 and table 1 | Power calculation indicates that there will be sufficient power with 1:1 matching To pre-specify sensitivity |
| | | | Changed primary analysis from PS fine-stratification weights to 1:1 PS matching Added planned sensitivity analyses | analyses |
| 16 <sup>th</sup> December<br>2024 | 2.1 | Appendices | Added the FDA protocol review dates for first and second feasibility | The protocol review dates by the FDA were not documented in the previous version. |
| 10 <sup>th</sup> March<br>2025 | 3 | Appendices | Covariate code algorithms for Pap smear, COPD, pneumonia, and diabetic nephropathy were corrected. | Errors in the implementation of covariate code algorithms for Pap smear, COPD, pneumonia, and diabetic nephropathy were identified. |
| 17 <sup>th</sup> April 2025 | 5 | Negative control outcomes | Added Hernia and Lumbar radiculopathy | Given the ongoing discussion around semaglutide and its potential association with non-arteritic anterior ischemic optic neuropathy (NAION) as a negative control outcome, we wanted to include alternative negative control outcomes. |

# 4. Rationale and background

The purpose of this protocol is to describe the emulation of the PIONEER6 trial (NCT02692716). Market availability of oral Semaglutide began on 19th September 2019.¹ The trial enrolled 3,183 participants between January and August 2017. The trial design was event-driven to collect 122 events, with an assumption of 3% event rate in both arms over a period of 7 months, which would result in 90% power, to rule out 80% excess cardiovascular risk to assess non-inferiority.².³

# 5. Research question and objectives

#### Table 1 Primary and secondary research questions and objective

# A. Primary research question and objective

| Objective: | To evaluate the effect of oral semaglutide versus sitagliptin (proxy for placebo) on MACE outcomes (CV death, nonfatal MI, or nonfatal stroke). |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will be superior to sitagliptin at preventing MACE |
| Population (mention key inclusion-exclusion criteria): | The study population includes patients with Type 2 Diabetes (Type2DM), >=50 years with established cardiovascular disease OR >=60 years with subclinical cardiovascular disease. Patients were excluded if they had type 1 diabetes, secondary or gestational diabetes, recent use of GLP-1, pramlitinide, or DPP4-I, had a history of diabetic ketoacidosis, pancreatitis, recent myocardial infarction, stroke, hospitalization for unstable angina or transient ischemic attack; heart failure class IV, personal or family history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma, chronic hemodialysis or peritoneal dialysis, end stage liver disease, malignant neoplasm within 5 years, current or recent pregnancy, proliferative retinopathy or maculopathy requiring treatment, history of major stomach surgeries |
| Exposure: | Oral Semaglutide |
| Comparator: | Sitagliptin |
| Outcome: | Major adverse cardiac event (MACE), including myocardial infarction, stroke, and all cause death |
| Time (when follow up begins and ends): | 1 days after cohort entry date until the first of outcome, disenrollment, end of study period, 365 days after cohort entry date, discontinuation (30 days grace and risk window), switch between the arms, |

| | start of any other GLP1 agonists (including injectable Semaglutide), Other DPP4 or Pramlintide, Nursing home admission |
|---|---|
| Setting: | Patients may be treated in outpatient settings. The outcome will be measured from inpatient hospitalizations and/or death. |
| Main measure of effect: | Hazard ratio |

# B. Secondary research question 1 and objective

| Objective: | To evaluate the effect of oral semaglutide versus sitagliptin on negative control outcomes, includi cataract surgery, B. hernia and C. lumbar radiculopathy |
|---|---|
| Hypothesis: | We hypothesize that semaglutide will not have a different effect than sitagliptin |
| Population (mention key inclusion-exclusion criteria): | The study population includes patients with Type 2 Diabetes (Type2DM), >=50 years with established cardiovascular disease OR >=60 years with subclinical cardiovascular disease. |
| | Patients were excluded if they had type 1 diabetes, secondary or gestational diabetes, recent use of GLP-1, pramlitinide, or DPP4-I, had a history of diabetic ketoacidosis, pancreatitis, recent myocardial infarction, stroke, hospitalization for unstable angina or transient ischemic attack; heart failure class IV, personal or family history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma, chronic hemodialysis or peritoneal dialysis, end stage liver disease, malignant neoplasm within 5 years, current or recent pregnancy, proliferative retinopathy or maculopathy requiring treatment, history of major stomach surgeries. In addition, patients were excluded for baseline hernia or lumbar radiculopathy when the negative outcome was hernia or lumbar radiculopathy respectively. |
| Exposure: | Oral semaglutide |
| Comparator: | Sitagliptin |
| Outcome: | Separate analyses were run for cataract surgery, hernia, and lumbar radiculopathy |
| Time (when follow up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, death, 365 days after cohort entry date, discontinuation (30 days grace and risk window), switch between the arms, start of any other GLP1 agonists (including injectable semaglutide) |
| Setting: | Patients may be treated in outpatient settings. The outcome will be measured from outpatient procedure codes |

| Main measure of effect: | Hazard ratio |
|-------------------------|--------------|

# 6. Research methods

#### 6.1. Study design

Research design (e.g. cohort, case-control, etc.): New user active comparator cohort study

Rationale for study design choice: For drug safety evaluations, a cohort study of new initiators is a powerful design that may be able to address confounding by indication. It accomplishes this, in large part, through judicious selection of an appropriate active-comparator group.<sup>4,5</sup> While selection of an appropriate comparator in the design phase is crucial, cohort studies often require additional adjustment of measurable confounders. A common method for adjusting for confounding is via a propensity score (PS).

#### 6.2. Study design diagram



Note: The CV disease inclusion may include acute MI codes but any acute MI in the 60 days is excluded. History of heart failure is an inclusion criterion, but heart failure class IV is excluded.

#### 6.3. Setting

#### 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population

Time 0 in the database study was defined to emulate randomization to treatment oral semaglutide versus sitagliptin in the clinical trial design. See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

#### 6.3.2 Context and rationale for study inclusion criteria:

Study inclusion criteria were defined to emulate the inclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in Appendix 3.

#### 6.3.3 Context and rationale for study exclusion criteria

Study exclusion criteria were defined to emulate the exclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in Appendix 3.

#### 6.4. Variables

#### 6.4.1 Context and rationale for exposure(s) of interest

The exposure and comparator were defined to emulate the agents compared for the trial, Oral Semaglutide versus Sitagliptin (proxy for placebo). See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

### Algorithm to define duration of exposure effect:

Assuming the effect of the drugs lasts for 30 days after the days' supply finishes, we allow 30 days gap between the dispensing (grace period) and also add 30 days extension at the end of days' supply of the last dispensing (exposure risk window).

### 6.4.2 Context and rationale for outcome(s) of interest

The primary outcome for the database study was defined to emulate the primary outcome for the trial of MACE. In the trial, this was a combination of myocardial infarction, stroke, and cardiovascular death. In our emulation, due to inability to capture cause of death, our modified MACE outcome was measured as inpatient myocardial infarction, inpatient stroke, and all-cause mortality. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. Optum includes death information from the inpatient discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. MarketScan includes information from the inpatient discharged dead status up until 2016. Medicare includes information from the inpatient discharged dead status, NDI cause of death, and social security death master file. The positive predictive value for the myocardial infarction outcome algorithm using ICD-9 codes was observed to be 88.4% and 94% in validation studies.<sup>6,7</sup> The PPV for the ischemic stroke outcome algorithm was 88% and 95% in validation studies using ICD9

codes.<sup>6,8</sup> The ICD9 code algorithms were mapped to ICD10 codes and reviewed by a clinician, but the performance of the mapped codes was not further validated.

Secondary outcomes from the trial that will be evaluated include:

- 1. Myocardial infarction
- 2. Stroke
- 3. All cause death

Control outcomes of interest include:

- 1. Cataract surgery. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.
- 2. Hernia. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.
- 3. Lumbar radiculopathy. This is a negative control outcome where no difference in effect is expected for semaglutide versus sitagliptin.

#### 6.4.3 Context and rationale for follow up

Both on-treatment (OT) and intention-to-treat (ITT) analyses will be conducted. Adherence in clinical practice is expected to be much worse than in the trial, therefore the OT analysis will be the primary analysis. The OT analysis targets the relative hazard of outcomes while on treatment and may more closely emulate the effect observed in highly adherent trial participants.

Table 2. Operational Definitions of Follow Up

| Follow up start | Day 1 | |
|---|---|---|
| Follow up end <sup>1</sup> | Select all that apply | Specify |
| Date of outcome | Yes | |
| Date of death | Yes | Part of the outcome |
| End of observation in data | Yes | Date of disenrollment |
| Day X following index date<br>(specify day) | Yes | Day 365 |
| End of study period (specify date) | Yes | Different dates for different databases (Optum: 29th Feb 2024, Marketscan Dec 31st 2022, Medicare Dec 31st 2020) |
| End of exposure (specify operational details, | Yes | 30 days grace window and 30 days risk window |

| e.g. stockpiling algorithm, grace period) | | |
|---|---|---|
| Date of add to/switch from exposure (specify algorithm) | Yes | Date of augmentation or switching from an exposure to a comparator and vice versa. |
| Other date (specify) | Yes | Censor upon starting any other GLP1 agonists, including injectable Semaglutide, Other DPP4 inhibitors or Pramlintide, Nursing home admission |

<sup>&</sup>lt;sup>1</sup> Follow up ends at the first occurrence of any of the selected criteria that end follow up.

# 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications)

We identified a series of covariates that were likely confounders due to being strong risk factors for the primary outcome that were associated with choice of treatment. These include demographics, disease severity related variables, comorbid conditions, comedications, frailty, healthcare utilization and markers of health seeking behaviour.

Table 3. Operational Definitions of Covariates

| Characteristic | Conceptual<br>Definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to<br>study<br>populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Age | Cohort entry year – year of birth, (last observed value in the baseline) | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Gender | Male, Female<br>(last observed<br>value in the<br>baseline) | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Region | Northeast, Midwest/North central, South, West (last observed value in the baseline) | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Year of Cohort<br>Entry | 2019 (Sept-Dec),<br>2020 (Jan-March),<br>2020 (April-June),<br>2020 (July-Sept),<br>2020 (Oct-Dec),<br>2021 (Jan-Dec),<br>2022 (Jan-Dec), | Categorical | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | n/a |


| Characteristic | Conceptual<br>Definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | sources in<br>Appendix 8 |
| Thiazolidinediones | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| SGLT-2i | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Alpha-glucosidase inhibitors | | Binary | [-180, -1] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| ACEs/ARBs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Thiazides | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Beta-blockers | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Calcium channel<br>blockers | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Loop diuretics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Other diuretics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual<br>Definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Nitrates | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Hear failure<br>medications<br>(Digoxin +<br>Entresto +<br>Ivabradine) | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anti-arrhythmics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| COPD/asthma medications | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Statins | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Other lipid-<br>lowering drugs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Antiplatelet agents | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Oral<br>anticoagulants | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| NSAIDs | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Oral corticosteroids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral Semaglutide | n/a | Investigator review of codes, |

| Characteristic | Conceptual<br>Definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | sources in |
| Bisphosphonates | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Appendix 8 Investigator review of codes, sources in Appendix 8 |
| Opioids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anti-depressants | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Gabapentinoids | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Benzodiazepines | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Anxiolytics/hypnot ics | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Medications for dementia | | Binary | [-180, 0] | n/a | generic | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Combined comorbidity score | Comorbidity score ranging from -2 to 26 | Continuous | [-180, 0] | Any | ICD10-CM | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | | Gagne, Joshua J<br>et al. <sup>9,10</sup> |
| Frailty score | | Continuous | [-180, 0] | Any | ICD10-CM | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | | Kim et al. <sup>11</sup> |

| Characteristic | Conceptual<br>Definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Unique generic<br>medicines | | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Unique brand medicines | | Continuous | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Hospitalizations<br>[-90, 0] | | Binary | [-90, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Hospitalizations<br>[-180, 0] | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| ED visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Office visits | | Continuous | [-180, 0] | OP | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Endocrinologist visit | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Cardiologist visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Internal medicine/family medicine visits | | Binary | [-180, 0] | n/a | n/a | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Electrocardiogram<br>s | | Binary | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide | n/a | Investigator review of codes, |

| Characteristic | Conceptual<br>Definitions | Type of variable | Assessment window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | sources in<br>Appendix 8 |
| Echocardiograms | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| HbA1c tests received | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Glucose tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Lipid tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Creatinine tests ordered | | Continuous | [-180, 0] | Any | CPT/HCPCS | Any | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Bone mineral density test | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Basic or<br>comprehensive<br>metabolic blood<br>chem test | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Mammogram | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Pap smear | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

| Characteristic | Conceptual<br>Definitions | Type of<br>variable | Assessment<br>window | Care<br>Settings¹ | Code Type <sup>2</sup> | Diagnosis<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics/ validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| PSA | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Flu vaccine/<br>Pneumococcal<br>vaccine | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |
| Telemedicine | | Binary | [-180, 0] | n/a | CPT/HCPCS | n/a | Exposure: Oral<br>Semaglutide<br>Reference:<br>Sitagliptin | n/a | Investigator<br>review of codes,<br>sources in<br>Appendix 8 |

 $<sup>^{1}</sup>$ IP = inpatient, OP = outpatient, ED = emergency department, OT = other, n/a = not applicable

# 6.5. Data analysis

#### 6.5.1 Context and rationale for analysis plan

The study will use a propensity score (PS) based fine-stratification weighting method with 50 strata<sup>7</sup>. The PS will be estimated as the probability of initiating oral Semaglutide versus Sitagliptin given the baseline patient characteristics using multivariable logistic regression models. 50 strata will be created based on the distribution of PS in oral Semaglutide treated patients, and weighted Sitagliptin initiators proportional to the distribution of oral Semaglutide initiators in the PS stratum. As diagnostics for PS models, the study will evaluate distributional overlap, weight distribution, and covariate balance using standardized differences post-weighting. The study will estimate the hazard ratio for oral Semaglutide versus Sitagliptin inhibitor on MACE outcome in the weighted population using a Cox proportional hazards model.

Table 4. Primary, secondary, and subgroup analysis specification

#### A. Primary analysis

<sup>&</sup>lt;sup>2</sup>See appendix for listing of clinical codes for each study parameter

<sup>&</sup>lt;sup>3</sup> Specify whether a diagnosis code is required to be in the primary position (main reason for encounter)

| Hypothesis: | Oral Semaglutide might decrease risk of MACE outcome compared to Sitagliptin |
|---|---|
| Exposure contrast: | Oral Semaglutide vs Sitagliptin |
| Outcome: | MACE |
| Analytic software: | Aetion, STATA 17, SAS 9.4, R.4.4.0 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | n/a |

# B. Secondary Analysis 1

| Hypothesis: | Oral semaglutide has no effect on risk of negative control outcomes compared to sitagliptin. Negative control outcomes |
|---|---|
| | include: A. cataract surgery, B. hernia, C. lumbar radiculopathy |
| Exposure contrast: | Oral semaglutide vs sitagliptin |
| Outcome: | Separate analyses were run for each negative control outcome, including cataract surgery, hernia and lumbar radiculopathy |
| Analytic software: | Aetion, STATA 17, SAS 9.4, R.4.4.0 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Operations adjustes out as other | Name weather and avertide velocity and details of his prints would invalid a way on the company weathing (a weathing a locality we |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score matching (specify matching algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |

| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
|---|---|
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present |
| Subgroup Analyses | List all subgroups |
| | n/a |

Table 5. Sensitivity analyses – rationale, strengths and limitations

| | What is being varied? How? | Why?<br>(What do you expect to<br>learn?) | Strengths of the sensitivity analysis compared to the primary | Limitations of the sensitivity analysis compared to the primary |
|---|---|---|---|---|
| Re-weighted population distribution | We will re-weight the population distribution of the pooled database study cohorts to reflect that of the RCT if that information is made public prior to publication of our results. | We will learn about potential effect modification due to different distributions of key characteristics such as age/sex in the RCT versus the database study. | The population distributions will be more aligned. | The measurement of these population characteristics may be measured differently in the RCT vs database study, with different levels of specificity and sensitivity. |
| Negative control<br>outcomes, including<br>cataract surgery,<br>hernia, lumbar<br>radiculopathy | We evaluate negative control outcomes of cataract surgery, hernia, and lumbar radiculopathy, where no causal effect is expected from semaglutide or sitagliptin | We will evaluate the potential impact of residual confounding on this outcome for which there is not expected to be a causal effect | The evaluates the robustness of<br>the interpretation of the primary<br>analysis by evaluating the<br>potential magnitude of<br>unmeasured confounding | This analysis assumes that the confounding structure is the same or similar for the negative control outcome as the outcome of interest |
| PS-adjustment<br>method | Instead of 1:1 PS matching, we will use PS fine stratification weights. The analytic cohort will be asymmetrically trimmed at 1% of the tails. The analytic cohort will be weighted to estimate the average effect in the treated (ATT). Each exposed patient will be assigned a weight = 1. | Use of fine-stratification<br>weights will have more power<br>than 1:1 matching | More power to estimate ATT | More complex to understand than simple 1:1 match, potentially less closely balanced |

| | Each comparator patient will be assigned a weight = $\frac{\binom{Nexposed\ in\ strata\ i}{Ntotal\ exposed}}{\binom{Nunexposed\ in\ strata\ i}{Ntotal\ unexposed}}$ | | | |
|---|---|---|---|---|
| Apply benchmark, expand, calibrate (BenchExCal) sensitivity and tipping point analysis | We will use the observed difference in result from emulation of SUSTAIN6 to recalibrate the result from the database study emulation of PIONEER6. We will conduct a tipping point analysis with a range of plausible estimates of the expected difference. | We expect to learn about the performance of BenchExCal in an example where we emulate an RCT for an expanded indication and an RCT result for the expanded indication is available. | The analysis will calibrate the primary result based on expected differences due to bias and/or design emulation differences and propagate uncertainty regarding the impact of these factors into the frequentist primary result | The ability to appropriately calibrate the result depends on how "close" the clinical context is between the initial and expanded indication. The approach assumes that the net effect of bias and design emulation differences is the similar. |

#### 6.6. Data sources

#### 7.6.1 Context and rationale for data sources

**Reason for selection:** The study will be conducted in 3 US health care claims databases: Optum Clinformatics (2019-Feb 2024), Merative Marketscan (2019-2022) and Medicare (a sample that includes all patients with diabetes or heart failure diagnosis, 2019-2020).

Strengths of data source(s): Each data source contains deidentified, longitudinal, date-stamped information on patient enrollment, demographics, inpatient/outpatient diagnosis and procedures, admission and discharge dates, and medication dispensation. The death data is captured in the Optum database from inpatient discharge status, social security death master file, and deaths scraped from obituaries or other sources. The death data in MarketScan is captured from the social security death master file and inpatient discharge status. It is recognized that the social security death master file has high specificity and positive predictive value for deaths. While this data resource has under captured deaths since 2011, the capture of deaths is not expected to be differential between compared exposure groups. The death data is captured in the Medicare database from inpatient discharge status, and social security death master file. 12-14

Limitations of data source(s): Patient healthcare encounters are only observable when they are enrolled in an insurance plan that contributes to the database. Patients may change insurance plans for multiple reasons. Both Optum Clinformatics and Merative MarketScan are primarily employer based insurance databases where patients may disenroll with job changes. Patients in Medicare may move in and out of fee-for-service plans. We are excluding person-time in health maintenance organization (HMO) plans due to concerns about the completeness of capture of diagnoses and procedures. This means that we require patients to be enrolled in Medicare parts AB and D during the baseline assessment window and censor patients if they switch to part C. In claims data, dispensing data for inpatient medication is unavailable. Diagnoses reflect billing practices, therefore algorithms (preferably validated) are needed for accurate phenotyping of patient conditions. Services that are not covered by insurance do not appear in the data. The trial evaluated cardiovascular deaths, however we will evaluate all cause death in the emulation because most deaths in this cohort of patients at high cardiovascular risk will be related to cardiovascular reasons, the cause of death is not recorded for databases not linked to NDI, and the performance of NDI at identifying cardiovascular causes of death may be suboptimal.<sup>14</sup>

Data source provenance/curation: Information about Optum Clinformatics and Merative MarketScan can be found in data dictionaries and user guides that are provided to clients. Information about Medicare data provenance and curation can be found on the ResDac website.<sup>15</sup>

Table 6. Metadata about data sources and software

| | Data 1 | Data 2 | Data 3 |
|---|---|---|---|
| Data Source(s): | Optum Clinformatics | Merative Marketscan | Medicare |
| Study Period: | 20th Sept 2019-29th Feb 2024 | 20th Sept 2019-31st Dec 2022 | 20th Sept 2019- 31st Dec 2020 |
| Eligible Cohort Entry Period: | 20th Sept 2019-29th Feb 2024 | 20th Sept 2019-31st Dec 2022 | 20 <sup>th</sup> Sept 2019- 31st Dec 2020 |
| Data Version (or date of last update): | April 2024 | Mortality Cut Set A<br>Received 2024-03-01 | DUA 59286_Received 2023-10-<br>17 |
| Data sampling/extraction criteria: | n/a | n/a | Patients with a diabetes or heart failure diagnosis |
| Type(s) of data: | Administrative healthcare claims | Administrative healthcare claims | Administrative healthcare claims |
| Data linkage: | n/a | n/a | Linkage to National Death Index |
| Conversion to CDM*: | n/a | n/a | n/a |
| Software for data management: | Aetion Evidence Platform® (2024) | Aetion Evidence Platform® (2024) | Aetion Evidence Platform® (2024) |

<sup>\*</sup>CDM = Common Data Model

#### 6.7. Data management

<u>Tracking data:</u> The Data Use Agreement (DUA) Custodian (Principal Investigator) and the Division Operations Manager (Winta Tekle) are responsible for receiving and creating a record of new data associated with the given request. The Operations Manager is responsible for all indexing and archiving of documents and electronic media related to data that the Division receives and will log data location, data contents, and associated DUA and Institutional Review Board (IRB) numbers in the Division's centralized tracking system.

<u>Handling and storage:</u> In-scope data will be stored utilizing Mass General Brigham approved information systems – i.e., Division servers and Mass General Brigham network storage.

<u>Archiving</u>: Data retention and any removal will be executed by the Division Operations Manager (Winta Tekle) and Data Manager (Todd MacGarvey). The Division follows Mass General Brigham enterprise record retention policies and follow the terms of the agreement through which the in-scope data was received.

Information security: The Division follows Mass General Brigham's Enterprise Information Security Program (EISP). The EISP helps by providing assurance that Mass General Brigham information and information systems are protected from unauthorized access, use, disclosure, duplication, modification, or destruction in order to maintain their confidentiality, integrity, and availability. To that end, the EISP policies, standards and procedures create an information security framework that is aligned with the recommendations of the International Organization for Standardization's (ISO) publication 27001 and the National Institute of Standards and Technology's (NIST) publication 800-53 Family of Controls and MGB regulatory and legal requirements (as a HIPAA covered entity).

Mass General Brigham workforce members are required to complete new workforce privacy and information security training upon hire and annually thereafter. Refresh training is provided as appropriate. Mass General Brigham workforce members are required to review and sign a Confidentiality Agreement upon hire and annually thereafter. Additionally, we follow Enterprise Information Security and Privacy policies, including Managing Workforce Members Information Security Responsibilities Policy, which was developed to help assure that Mass General Brigham workforce members are competent and eligible to support the information security responsibilities associated with their role. Mass General Brigham workforce, including Division staff, are required to comply with Enterprise Information Security and Privacy Policies.

<u>Facilities:</u> The research team uses a highly secure, state-of-the-art, computing facility housed at Mass General Brigham's Corporate Data Centers in Needham and Marlborough, Massachusetts as well as Amazon Web Services (AWS). We maintain redundant storage for maximal data integrity and high-speed data access.

The Division uses Mass General Brigham corporate provisioned servers to analyze and store data in connection with this project. There are strict access controls enforced by technical means to ensure that only study staff who have been approved to conduct data analyses and contracted data engineers are able to access data (e.g., Mass General Brigham Authentication (Active Directory) utilized; auditing, logging, and monitoring enabled; firewalls enabled; etc.). All Division servers used in this study are accessible to only authorized staff only through the MGB network and utilizing VPN as appropriate (i.e., users must be on the network and logged into VPN to access). Mass General Brigham has a network information security monitoring team and in-scope servers are enrolled in enterprise security tools (e.g., vulnerability scanning service, antivirus, etc.).

The Division also uses AWS. In-scope AWS services / resources have undergone review and assessment by Mass General Brigham's Information Security Risk Assessment Team/ InfoSec Risk Management Team as required and in alignment with NIST 800-30: Guide for Conducting Risk Assessments. In-scope AWS servers are for our exclusive use (reserved instances), are covered under our organization's Business Associate Agreement with AWS. In-scope servers are housed in anonymous facilities that are not branded as AWS facilities. Physical access is strictly controlled both at the perimeter and at building ingress points by professional security staff utilizing video surveillance, intrusion detection systems, and other electronic means.

Security attributes and controls for the Division's use of in-scope AWS in connection with this project include: encryption at rest and in transit (industry standard AES-256 encryption, SSL/TSL), anti-malware, latest OS updates and patches as well as anti-virus; multi-factor authentication (MFA), Identity and Access Management, including SSO; auditing and logging; principle of least privilege, including for traffic and ports (e.g., deny all default configurations), use of VPC enabled Step functions, etc.; separation between environments; minimum necessary (out of the box AWS roles are not used as they can be overly permissive); all data would reside in the US domestic regions – use only US east HIPAA compliant region; performance monitoring enabled and reviewed as per internal processes; passwords compliant with enterprise password policy and, as appropriate, more protective password requirements; etc. Our Division's AWS use is also subject to ongoing evaluation and monitoring as well – e.g., vulnerability scanning and management, access review, etc.

A data file list will be maintained in Amazon S3 and tracked through Cloudtrail and Cloudwatch. Reporting of data file availability for any file stored in an S3 bucket will be controlled by MGB.

Amazon EC2, Amazon EBS, and Amazon VPC are integrated with AWS CloudTrail, a service that provides a record of actions taken by a user, role, or an AWS service in Amazon EC2, Amazon EBS, and Amazon VPC. CloudTrail captures all API calls for Amazon EC2, Amazon EBS, and Amazon VPC as events, including calls from the console and from code calls to the APIs. MGB IT/security staff have full access to CloudTrail to ensure that CloudTrail monitoring is available at all times. Amazon CloudWatch Events delivers a near-real-time stream of system events that describe changes in AWS resources. Amazon CloudTrail can log, continuously monitor, and retain account activity related to actions across the MGB AWS infrastructure. CloudTrail provides event history of MGB AWS account activity. This event history simplifies security analysis, resource change tracking, and troubleshooting and complies with requirements to ensure the data file inventory is controlled by MGB.

Backups: Backups are created using industry recognized Cryptographic mechanisms (e.g., 256-bit AES encryption) as appropriate and required. Data are backed up within the MGB network from the MGB Needham data center to the MGB Marlborough data center via replication/mirroring and volume-level snapshots.\_AWS Backup supports both instance-level backups as Amazon Machine Images (AMIs) and volume-level backups as separate snapshots based on the resource tags. AMIs allow MGB IT and security staff to create backups of all S3 and EC2 instances. This backup approach allows elimination of EC2 instances when access to CMS data files is no longer needed. Use of temporary instances will allow highest security control to be applied regarding for whom and when CMS data files are accessible.

In addition to the safeguards listed above, the Division follows enterprise privacy and information security policies and maintains internally procedures in connection with this project to safeguard the data in connection with this project as appropriate and required including: Physical Security and Environmental Controls for Electronic Information Policy; IT Access Control Standards for Users policy; Safeguarding Fax Copiers Printers Telephone Use and Pagers; Physical Removal and Transport of Protected Health Information and Personal Information policy, etc.

# 6.8. Quality control

Senior Programmers and Research Specialists perform QA/QC on raw or common data model converted data via SAS/R/Aetion software. The protocol will be iteratively developed and pre-specified data checks including feasibility counts and balance on baseline covariates will be conducted with outputs reviewed by both MGB and FDA team members. Team members will review code lists to ensure fidelity to intended algorithms

# 6.9. Study size and feasibility

First feasibility assessment: Details of power calculations after applying eligibility criteria and matching on ages, sex and comorbidity score are available in appendix 4.

Second feasibility assessment: Details of power calculations after matching or weighting on all predefined propensity score variables are available in appendix 5..

Propensity score distribution plots with c-statistics are available in appendix 6. Table 1 showing prevalence of baseline characteristics and standardized differences in distribution are available in appendix 7.

### 7. Limitation of the methods

As we are using secondary data and the data were not collected for research, some important variables may not be collected or will be measured imperfectly. We have selected validated algorithms when possible and we have created proxies for important variables that are not directly captured in the data to reduce confounding by unmeasured factors. One measurement difference is for the primary outcome, where for the RCT, MACE was defined as stroke, myocardial infarction, and cardiovascular death, whereas in our database study, it is defined as stroke, myocardial infarction, and all cause death.

When comparing results from an RCT to a database study that emulates the design, we assume that the findings from the single RCT are internally valid which is not guaranteed.

Although we plan to emulate the important features of each RCT as closely as possible in healthcare claims, there may be some elements of RCT design that are not emulable with a database study, which means that the study generating RWE and the RCT will address slightly different clinical questions. For example, in routine clinical practice, adherence to treatment is typically not as high as it is in an RCT with strong measures in place to encourage adherence to the study protocol. This means that there is more discontinuation and short-term medication use in the patients identified in claims databases than trial participants.

Apparent agreement between RCT and database study results could occur if the effects of multiple factors (chance, emulation differences, bias) cancel each other out.

# 8. Protection of human subjects

This study has been approved by the Brigham and Women's Hospital Institutional Review Board.

# 9. References

- 1. Novo Nordisk Receives FDA Approval of OZEMPIC® (semaglutide) Injection For the Treatment of Adults with Type 2 Diabetes. <a href="https://www.prnewswire.com/news-releases/novo-nordisk-receives-fda-approval-of-ozempic-semaglutide-injection-for-the-treatment-of-adults-with-type-2-diabetes-300567052.html#:~:text=OZEMPIC%C2%AE%20(semaglutide)%20injection%200.5%20mg%20or%201%20mg%20was,adults%20with%20type%202%20diabetes. PR Newswire.
- 2. ClinicalTrials.gov. Trial to Evaluate Cardiovascular and Other Long-term Outcomes With Semaglutide in Subjects With Type 2 Diabetes (SUSTAIN™ 6). National Institutes of Health. Accessed April 30, 2024. <a href="https://www.clinicaltrials.gov/study/NCT01720446">https://www.clinicaltrials.gov/study/NCT01720446</a>
- 3. Husain M, Birkenfeld AL, Donsmark M, et al. Oral Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. *N Engl J Med*. Aug 29 2019;381(9):841-851. doi:10.1056/NEJMoa1901118
- 4. Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. *Pharmacoepidemiol Drug Saf.* Aug 2010;19(8):858-68. doi:10.1002/pds.1926
- 5. Ray WA. Evaluating Medication Effects Outside of Clinical Trials: New-User Designs. *American Journal of Epidemiology*. November 1, 2003 2003;158(9):915-920. doi:10.1093/aje/kwg231

- 6. Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. *Pharmacoepidemiol Drug Saf*. Jun 2010;19(6):596-603. doi:10.1002/pds.1924
- 7. Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. *Am Heart J*. Jul 2004;148(1):99-104. doi:10.1016/j.ahj.2004.02.013
- 8. Tirschwell DL, Longstreth WT, Jr. Validating administrative data in stroke research. *Stroke*. Oct 2002;33(10):2465-70. doi:10.1161/01.str.0000032240.28636.bd
- 9. Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. *J Clin Epidemiol*. Jul 2011;64(7):749-59. doi:10.1016/j.jclinepi.2010.10.004
- 10. Sun JW, Rogers JR, Her Q, et al. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. *Med Care*. Dec 2017;55(12):1046-1051. doi:10.1097/mlr.000000000000824
- 11. Kim D, Schneeweiss S, Glynn R, Lipsitz L, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. *Journals of Gerontology: Medical Sciences*. 2017;73:980-987. doi:10.1093/gerona/glx229
- 12. Jarosek S. Death Information in the Research Identifiable Medicare Data. Accessed June 17, 2024. <a href="https://resdac.org/articles/death-information-research-identifiable-medicare-data">https://resdac.org/articles/death-information-research-identifiable-medicare-data</a>
- 13. Hill ME, Rosenwaike I. The Social Security Administration's Death Master File: The Completeness of Death Reporting at Older Ages. *Social Security Bulletin*. 2002;64(1):45-51.
- 14. Olubowale OT, Safford MM, Brown TM, et al. Comparison of Expert Adjudicated Coronary Heart Disease and Cardiovascular Disease Mortality With the National Death Index: Results From the REasons for Geographic And Racial Differences in Stroke (REGARDS) Study. *J Am Heart Assoc*. May 3 2017;6(5)doi:10.1161/jaha.116.004966
- 15. Research Data Assistance Center (ResDAC). https://resdac.org/. Centers for Medicare & Medicaid Services (CMS).

# 10. Appendices

See accompanying excel file.

- 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1

# **Appendices**

- 1 Target Trial Framework, Operational Definitions and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate algorithm sources

| | (add trialname here) trial definitions | (Optum) | (Medicare) | (MarketScan) | Notes/Questions | Color coding |
|---|---|---|---|---|---|---|
| atment assignment (time<br>0, index date | Parallel, randomized (treatment A vs B) double blind, double-dummy | Non-randomized initiation of treatment A vs B<br>(first eligible entry to study population after applying inclusion-<br>exclusion criteria) | Non-randomized initiation of treatment A vs B<br>(first eligible entry to study population after applying inclusion-<br>exclusion criteria) | Non-randomized initiation of treatment A vs B<br>(first eligible entry to study population after applying inclusion-<br>exclusion criteria) | | |
| Exposur | Semaglutide (oral 3mg, 7mg 14mg; target dose of 14mg) | Code type: Generic name with route of administration/NDC code/Brand name Care setting: N/A Diagnosis position: N/A Washout Window; 1:80, -1] Incident with respect tos:emaglutide and sitagliptin in any formulation and any strength Assessement window; N/A Source of algorithme: N/A Measurement characteristics: N/A | Code type: Generic name with route of administration/NDC code/Brand name Care setting N/A Diagnosis position: N/A Washout window; 1:80, -1] Inclident with respect tossemaglutide and sitagliptin in any formulation and any strength Assessement window: N/A Source of algorithm: N/A Measurement characteristics: V/A | Code type: Generic name with route of administration/NDC code/Brand name Care setting: N/A Diagnosis position: N/A Washout window; 1:80, -1] Incident with respect tossemaglutide and sitagliptin in any formulation and any strength Assessement window: N/A Source of algorithm: N/A Measurement characteristics: V/A | We defined oral semaglutide using generic name with route of administration, ndc codes and also brand name | Good proxy definition |
| Comparato | Placebo | Code type: Generic name Care setting: [N/A] Diagnosis position: N/A Weshout Window: 1.30 - 1.1 Incident with respect to:semaglutide and sitagliptin in any formulation and any strength Assessment window: N/A Source of algorithms/N/A Messurement characteristics: I/A | Code type: Generic name Care setting; No. 19/A Diagnosis position: 1/A Washout Window(1:40: -1] Incident with respect to:semaglutide and sitagliptin in any formulation and any strength Assessment window: 1/A Source of algorithm: 1/A Messurement characteristics: 1/A | Code type: Generic name Care setting; No.18/A Diagnosis position: 1/A Washout widnow(1:4801] Incident with respect to:semaglutide and sitagliptin in any formulation and any strength Assessment window: 1/VA Source of algorithmist/A Messurement chearacteristicst/VA | We used stagliptin as an active comparator proxy for<br>placebo. We allowed stagliptin alone or in<br>combination pills with metformin only. | Moderate proxy definition |
| Primary Outcom | MACE, Defined as Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-<br>fatal Stroke | Code type:DX Care setting: inpatient Diagnosis position:Primary for Stroke, Any for MI Weahout Window: Source of algorithms:PROMISE team Measurement characteristics:PPV for MI using ICD9 codes was 88.4% and 54% [Inttps://pubmed.ncbi.nlm.nih.gov/20140892/ and Inttps://pubmed.ncbi.nlm.nih.gov/12516798/1] PPV for ischemic stroke using ICD9 codes was 88% and 95% [Inttps://pubmed.ncbi.nlm.nih.gov/12364739/ and Inttps://pubmed.ncbi.nlm.nih.gov/12364739/ and Inttps://pubmed.ncbi.nlm.nih.gov/12364739/ and Inttps://pubmed.ncbi.nlm.nih.gov/120140892/1 Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | loods type: IX Corn setting in patient Diegnoels position: Primary for Stroke, Any for MI Washout window: Source of algorithm: PROMISE team Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94% [https://pubmed.ncbi.mim.in.gov/20140832/ and https://pubmed.ncbi.mim.in.gov/20140832/ and https://pubmed.ncbi.mim.in.gov/12014739/ and https://pubmed.ncbi.mim.in.gov/1204739/ and https://pubmed.ncbi.mim.in.gov/1204739/ and https://pubmed.ncbi.mim.in.gov/1204739/ and https://pubmed.ncbi.mim.in.gov/20140892/] Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | loods type:IX Core setting inpatient Diegnoels position:Primary for Stroke, Any for MI Washout window: Source of algorithm:PROMISE team Measurement characteristics: PV for MI using ICD9 codes was 88.4% and 94% PV for MI using ICD9 codes was 88.4% and 94% [https://pubmed.ncbi.mim.in.gov/20140892/ and https://pubmed.ncbi.mim.in.gov/20140893/ PV for ischemic stroke using ICD9 codes was 88% and 95% [https://pubmed.ncbi.mim.in.gov/12364739/ and https://pubmed.ncbi.mim.in.gov/12364739/ and https://pubmed.ncbi.mim.in.gov/20140892/] Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. | Optum death includes information from the inpatient discharged dead status, social security death master file, and deaths scraped from obtainers or other sources. MarketScan includes information from the inpatient discharged dead status up until 2016. Medicare includes information from the inpatient discharged dead status, NDI cause of death, and social security death master file. | Poorly measured in database but not critic for the analysis |
| Follow up star | Randomization date | One day after date of initiation of treatment A vs B | One day after date of initiation of treatment A vs B | One day after date of initiation of treatment A vs B | | Poorly measured and important for the analysis |
| Follow up end | Time Frame: Maximum treatment duration is dependent on event rates and is estimated to be no longer than 19 months +5 weeks of follow-up period. | Earliest of: Outcome, End of observation in data, end of data/study period, 19 months + 5 weeks, discontinuation (30 days grace window and risk-window), switch within or between GLP and DPP4 or add pramlintide, disenrollment, nursing home stay | Earliest of: Outcome, End of observation in data, end of data/study period, 19 months + 5 weeks, discontinuation (30 days grace window and risk-window), switch within or between GLP and DPP4 or add pramlintide, disenrollment, nursing home stay | Earliest of: Outcome, End of observation in data, end of data/study period, 19 months + 5 weeks, discontinuation (30 days grace window and risk-window), switch within or between GLP and DPP4 or add pramlintide, disenrollment, nursing home stay | | |
| Causal estiman<br>Effect estimation | Modified intention-to-treat | On-treatment | On-treatment | On-treatment | | - |
| inclusion criteria | | Applied before/after selection of Index dat@efore | Applied before/after selection of Index dat@efore | | | - |
| 1 | Type 2 DM | Applied Detrory arter assection or index dateserore Assessment window(;180, 0) Code type:DX Core setting: Any Diagnosis position:Any Source of algorithmsPROMISE team Measurement characteristicsti/A | Applied petroty arter selection or index dateserore Assessment windows [180, 0] Code type:DX Core settling: Any Diagnosis position: Any Source of algorithm:PROMISE team Measurement cheracteristics:V/A | Applied before/after selection of Index databetore Assessment windows [-180, 0] Code type:DX Care setting: Any Diagnosis poetition:Any Source of algorithm:PROMISE team Measurement cherarcteristics/V/A | | |
| 2a or 21 | | Applied before/after selection of Index dat@efore | Applied before/after selection of Index dat@efore | Applied before/after selection of Index dat@efore | | 1 |
| 22 | Age above or equal to 50 years at screening and clinical evidence of cardiovascular disease. Established CVD as one of the following: | Assessment window.[0, 0] Code type:n/a Care setting: n/a Diagnosts postton:n/a Source of algorithmen/a Measurement characteristicstv/A | Assessment window:[0, 0] Code type:n/a Care setting: n/a Diagnosis position:n/a Source of algorithm:n/a Measurement characteristics/ti/A | Assessment window:[0, 0] Code type:n/a Care setting: n/a Diagnosis position:n/a Source of algorithm:n/a Measurement characteristics!\/A | | |
| 2a: | prior myocardial infarction | Applied before/after selection of Index date/efore Assessment window(=180, 0) Code type:DX Core setting: Any Diagnosis position:Any Source of algorithmsPROMISE team Measurement characteristics:1/A | Applied before/after selection of Index detelerore Assessment windows [-180, 0] Code type:DX Core setting: Any Diagnosis position: Any Source of algorithm:PROMISE team Measurement characteristics:V/A | Applied before/after selection of index detainfore Assessment windows [-180, 0] Code type:DX Care setting: Any Diagnosis position: Any Source of algorithm:PROMISE team Measurement characteristics:V/A | | |
| 2aú | prior stroke or prior transient ischemic attack | Applied before/wfiter selection of Index date@efore Assessment window(=180, 0) Code type:DX Core setting: Any Diagnosis position:Any Source of algorithmsPROMISE team Measurement characteristicst/A | Applied before/after selection of index datelefore<br>Assessment windows (=180, 0)<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics:V/A | Applied before/after selection of index detelerore Assessment windows (=180, 0) Code type:DX Core setting: Any Diagnosis position: Any Source of algorithm:PROMISE team Messurement characteristics:*//A | | |
| <b>2</b> a3 | prior coronary, carottid or peripheral arterial revascularization | Applied before/after selection of Index dat@efore<br>Assessment Window:[-180, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team, Investigator review of<br>codes<br>Measurement characteristics:N/A | Applied before/after selection of index date/efore<br>Assessment window:[1.80, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team, Investigator review of codes<br>Measurement characteristics:\/A | Applied before/after selection of Index date/efore<br>Assessment window:[1.80, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team, Investigator review of codes<br>Measurement characteristics:\(\frac{1}{2}\)/A | | |
| 24 e | | Applied before/after selection of index datelefore Assessment windows:[-180, 0] Code type:PX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics!\/A Can't measure in claims | Applied before/after selection of index dates fore<br>Assessment window:[-180, 0]<br>Code type:PX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of elgorithm:PROMISE team<br>Measurement characteristics!\/A | Applied before/after selection of Index datesefore Assessment windows.[-180, 0] Code type:PX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics:\(^{1}\)/A Can't measure in claims | Part of this is captured in the above inclusion or<br>We also added peripheral vascular disease and<br>coronary atherosclerosis codes to be inclusive |
|---|---|---|---|---|---|
| e | istory of symptomatic coronary heart disease documented by e.g. positive<br>vercise stress test or any cardiac imaging or unstable angina with ECG changes | | | | |
| 6 es | symptomatic cardiac ischemia documented by positive nuclear imaging test or<br>xercise test or stress echo or any cardiac imaging | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| <b>7</b> cl | hronic heart failure New York Heart Association (NYHA) class II-III | Applied before/after selection of index detelefore Assessment windows [-180, 0] Code type.DX Care setting: Any Diagnosis position: Any Source of algorithm:PROMISE team Measurement characteristics: I/A | Applied before/after selection of index detelerore<br>Assessment windows [-180, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics:I/A | Applied before/after selection of Index datelefore<br>Assessment windown[-180, 0]<br>Code type.DX<br>Care setting: Any<br>Diagnosis position: Any<br>Source of algorithm: PROMISE team<br>Measurement characteristics: V/A | We defined by using heart failure codes (patient<br>type 4 heart failure are excluded so hopefully the<br>help with capturing patients with milder heart fa<br>this class) |
| 8 CI | hronic renal impairment, documents by estimated eGFR < 60 ml/min/1.73 m2<br>er MDRD | Applied before/after selection of index detelefore Assessment windows(=180, 0) Code type:DX Care setting: Any Diagnosis position:Any Source of algorithms:PROMISE team Measurement cheracteristics:V/A | Applied before/after selection of Index databefore<br>Assessment window; [180, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics:V/A | Applied before/after selection of Index datasefore<br>Assessment windows.[-180, 0]<br>Code type.DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithms:PROMISE team<br>Measurement characteristics:V/A | We defined it by CKD 3-4 |
| 2ь | with subclinical evidence of cardiovascular disease. | Applied before/after selection of Index date/efore<br>Assessment window:(0, 0)<br>Code type:r/g<br>Care setting: n/a<br>Diagnosia poetition:r/a<br>Source of algorithm:n/a<br>Measurement characteristics:r/a | Applied before/after selection of Index date/efore Assessment window:[0, 0] Code type:n/a Care setting: n/a Diagnosis poetition:n/a Source of algorithm:n/a Measurement characteristics:n/a | Applied before/after selection of index datasefore<br>Assessment window(0, 0)<br>Code type:n/a<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithm:n/a<br>Measurement characteristics:n/a | |
| <b>1</b> pe | ersistent microalbuminuria (30–299 mg/g) or proteinuria | Applied before/after selection of index datelefore Assessment windows:[-180, 0] Code type::DX Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement otherarcteristics://a | Applied before/after selection of index datelefore<br>Assessment window:[-180, 0]<br>Oxde type:DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics://a | Applied before/effer selection of Index det&efore<br>Assessment windows.[-180, 0]<br>Cade type.DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of signifitant-PROMISE team<br>Measurement characteristics:r/a | |
| b2 hy | ypertension and left ventricular hypertrophy by electrocardiogram or imaging | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| | ft ventricular systolic or diastolic dysfunction by imaging | Can't measure in claims Applied before/after selection of index detalefore Assessment window;[-180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithmishvestigator review of codes Measurement characteristics://a | Can't measure in claims Applied before/after selection of Index detalefore Assessment windows[:180, 0] Code type:DX Care setting: Any Diagnosis position:Any Source of algorithm:investigator review of codes Measurement characteristics:1/a | Can't measure in claims Applied before/after selection of Index datasefore Assessment windows[-180, 0] Code type.DX Care setting: Any Diagnosis position:Any Source of algorithm:investigator review of codes Measurement characteristics:1/a | |
| | ype 1 diabetes mellitus, Secondary diabetes, Gestational diabetes | Applied before/after selection of Index datelefore Assessment windows:[-180, 0] Oode type:UN Care setting: Any Diagnosis position:Any Source of algorithm:PROMISE team Measurement of haracteristics!V/A | Applied before/after selection of index datelefore<br>Assessment windows:[-180, 0]<br>Out bype:0X<br>Care setting: Any<br>Diagnosis potition:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics!y/A | Applied before/after selection of Index dat@efore<br>Assessment windown[-180, 0]<br>Code byse.10%<br>Care setting: Any<br>Disgnosis position:Any<br>Source of signothins:PROMISE team<br>Measurement characteristics:V/A | Secondary diabetes, Gestational diabetes are the additional criteria added |
| | se of glucagon-like peptide-1 (GLP-1) receptor agonist (exenatide, liraglutide, or<br>ther) or pramlintide within 90 days prior to screening | Applied before/after selection of index datablefore Assessment windows(=180, 0) Code type:Generic Care setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristics:n/a | Applied before/after selection of Index databefore<br>Assessment window.[-180, 0]<br>Code type:Generic<br>Care setting: n/a<br>Diagnosis position://a<br>Source of algorithm:PROMISE team<br>Measurement obaracteristics://a | Applied before/after selection of Index dateefore Assessment window.[-180, 0] Code type.Generic Care setting.n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement obsarvateristics:n/a | we are doing 180 days look back |
| | se of any dipeptidyl peptidase 4 (DPP-IV) inhibitor within 30 days prior to<br>creening | Applied before/after selection of Index detalefore Assessment windows(=180, 0) Code type:Generic Care settling: "/a" Diagnosis position: "/a" Source of algorithm:PROMISE team Measurement characteristics: "/a | Applied before/after selection of Index detelerore<br>Assessment window. [180, 0]<br>Code type:Generic<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithm:PROMISE team<br>Measurement characteristics:1/a | Applied before/after selection of Index datasefore<br>Assessment window.[-180, 0]<br>Code type.Generic<br>Care setting. n/a<br>Diagnosis position:n/a<br>Source of algorithm=ROMISE team<br>Measurement characteristics:n/a | we are doing 180 days look back |
| н | istory of diabetic ketoacidosis | Applied before/after selection of index datelefore Assessment windows[-90, 0] Code type:DX Core setting: n/a Diagnosis position:n/a Source of algorithm:PROMISE team Measurement characteristics:n/a | Applied before/after selection of index dates/ore<br>Assessment windows[:90, 0]<br>Code type:DX<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithm:PROMISE team<br>Measurement characteristics:y/a | Applied before/after selection of Index dateefore<br>Assessment windows.[-90, 0]<br>Code type:DX<br>Care setting: n/a<br>Disgross position:n/a<br>Source of algorithm-PROMISE team<br>Measurement characteristics:n/a | 90 days assessment window based on SUSTAIN criteria |
| н | istory of chronic pancreatitis or idiopathic acute pancreatitis | Applied before/after selection of index date/efore<br>Assessment windows:[-180, 0]<br>Code type::DX<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithms:PGMISE team<br>Measurement characteristics:)/a | Applied before/after selection of index date/efore<br>Assessment windows:[-180, 0]<br>Odd type:DX<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithm:PROMISE team<br>Measurement characteristics:n/a | Applied before/after selection of Index datesfore<br>Assessment windows.[-180, 0]<br>Code type:DX<br>Care setting: n/a<br>Diagnosis position:n/a<br>Source of algorithm:PROMISE team<br>Measurement characteristica;/a | |

| | A - Wall of the Conference of the Lands of the Conference of the C | A - H - A b - A A A A A A - | A - U - d b - d (-db l db d l - d d - t - c - / | |
|---|---|---|---|---|
| Any of the following: myocardial infarction, stroke, or hospitalization for unstable angina or transient ischemic attack within the past 60 days prior to screening | Applied before/after selection of index datalefore Assessment window;[-60, 0] Code type:DX Care setting: Inpatient Diagnosis position:Any Source of algorithms:PROMISE team Measurement characteristics:r/a | Applied before/after selection of index datelefore<br>Assessment window; [-6, 0]<br>Code type:DX<br>Care setting: Inpatient<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics://a | Applied before/after selection of Index datelefore Assessment window; (-6,0,0) Code type: DX Care setting: Inpatient Diagnosis position:Any Source of algorithm:PROMISE team Measurement characteristics://a | |
| Currently planned coronary, carotid or peripheral artery revascularisation | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| Chronic heart failure New York Heart Association (NYHA) class IV | Applied before/after selection of index datate/ore Assessment windows(-180, 0) Code type:Dx, PX, Core esting: PP, Any Diagnosis position:Any Source of algorithms*PROMISE team Measurement characteristics:n/a | Applied before/after selection of index dates/ore Assessment window;(-180, 0) Code type:DX, PX Care setting: IP, Any Diagnosis position:Any Source of algorithms:PROMISE team Measurement characteristics://a | Applied before/after selection of Index datelerore Assessment window(:180, 0) Code type: DX, PX Care setting: IP, Any Diagnosis position:Any Source of algorithms:PAOMISE team Measurement characteristics://a | We defined this as heat failure codes in inpatient setting with oxygen use code on the same day |
| Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medulary thyroid carcinoma | Applied before/after selection of Index datalefore Assessment windows [-180, 0] Code type:DX Care setting: Inpatient Diagnosis position:Any Source of alignithms*PROMISE team Measurement characteristics:n/a | Applied before/after selection of index dateerfore<br>Assessment window; 138, 0]<br>Ode type:DX<br>Care setting: Inpatient<br>Diagnosis position:Any<br>Source of algorithms (MISE team<br>Measurement oharacteristics://a | Applied before/after selection of Index dat@efore Assessment window(:180, 0) Code type: DX Care setting: Inpatient Diagnosis position:Any Source of algorithms/PAOMISE team Measurement characteristics:y/a | |
| Chronic hemodialysis or chronic peritoneal dialysis | Applied before/after selection of index datalefore Assessment windows(-180, 0) Code type:Dx, PX Care setting: Inpatient Diagnosis position:Any Source of algorithms*PROMISE team Measurement of haracteristics:r/a | Applied before/after selection of Index dates/fore<br>Assessment window; [-180, 0]<br>Code type:DX, PX<br>Care setting: Inpatient<br>Diagnosis position:Any<br>Source of algorithms/PROMISE team<br>Measurement characteristics://a | Applied before/after selection of Index datelerore Assessment window(:180, 0) Code type: DX, PX Care setting: Inpatient Diagnosis position:Any Source of algorithms:PAOMISE team Measurement characteristics://a | We defined using CKD5/ESRD/Dialysis/Renal transplant code |
| End-stage liver disease, defined as the presence of acute or chronic liver disease and recent history of one or more of the following: ascites, encephalopathy, variceal bleeding, billriohia > 2.0 mg/d, albumin lew 3.5 g/d, potrormbin time 24 seconds prolonged, international normalized ratio >1.7 or prior liver transplant | https://pubmed.ncbi.nlm.nih.gov/34256144/ Measurement characteristics: | Applied before/after selection of Index data: Before<br>Assessment window(-180, 0)<br>Code type:DX, PX, RX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:<br>https://pubmed.ncbi.nlm.nih.gov/22674685/ and<br>https://pubmed.ncbi.nlm.nih.gov/34256144/<br>Messurement oharacteristics: | Applied before/after selection of Index date: Before<br>Assessment window(:180, 0)<br>Code type: DX, PX, RX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of signathum:<br>https://pubmed.ncbi.nlm.nih.gov/242674685/ and<br>https://pubmed.ncbi.nlm.nih.gov/24266144/<br>Messurement observations: | According to<br>https://pubmed.ncbi.nlm.nih.gov/22674685/, ESLD in<br>claims can be defined using Cirrohosis +<br>Decompensation event.<br>Decompensation event<br>we used the ICD9/ICD10 codes from the above study<br>and https://pubmed.ncbi.nlm.nih.gov/34256144/, to<br>define the codes required for Cirrhosis and<br>Decompensation events |
| A prior solid organ transplant or awaiting solid organ transplant | Applied before/after selection of index datalefore Assessment windows(=180, 0) Code typecDX, PX Care setting: inpatient Diagnosis position:Any Source of algorithms/PROMISE team Measurement characteristics:r/a | Applied before/after selection of index dateerfore<br>Assessment window; (-180, 0)<br>Code type: DX, PX<br>Care setting: Inpatient<br>Diagnosis position: Any<br>Source of algorithms<br>Measurement characteristics: // a | Applied before/after selection of Index dat@efore<br>Assessment window(:180, 0)<br>Code type: DX, PX<br>Cale setting: Inpatient<br>Diagnosis position:Any<br>Source of algorithm:PROMISE team<br>Measurement characteristics://a | |
| Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer) | Applied before/after selection of Index dat@efore Assessment windows(=1825, 0) Code type:DX Care setting: Any Diagnosis position:Any Diagnosis position:Any Source of algorithms?PROMISE team Measurement characteristics:n/a | Applied before/after selection of Index dat@efore<br>Assessment windows[-1825, 0]<br>Code type:DX<br>Care setting: Any<br>Diagnosis postton:Any<br>Source of algorithms/POMISE team<br>Measurement characteristics://a | Applied before/after selection of Index dat@efore<br>Assessment windows(-1825, 0]<br>Code type: DX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of algorithm:PAOMISE team<br>Measurement characteristics:y/a | |
| Any acute condition or exacerbation of chronic condition that would in the investigator's opinion interfere with the initial trial visit schedule and procedures | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice) | Applied before/after selection of Index datalefore Assessment windows(=180, 0) Code type:Dx, PX, Core esting: AP, Diagnosis position:Am, Diagnosis position:Am, Messurement characteristics:n/a | Applied before/after selection of Index dateerfore<br>Assessment window:[-180, 0]<br>Ode type:DX, PX<br>Care setting: Any<br>Diagnosis position:Any<br>Sugnosis position:Any<br>Measurement characteristics://a | Applied before/after selection of Index dat@efore Assessment window(:180, 0) Code type: DX, PX Care setting: Any Diagnosis position:Any Source of algorithmsPregnancy team Measurement characteristics://a | |
| Known or suspected hypersensitivity to trial products or related products Previous participation in this trial. | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| | Can't measure in claims Can't measure in claims | Can't measure in claims Can't measure in claims | Can't measure in claims Can't measure in claims | |
| Receipt of any investigational medicinal product within 90 days prior to screening | | | | |
| Any other factor likely to limit protocol compliance or reporting of adverse event at<br>the discretion of the investigator | Can't measure in claims | Can't measure in claims | Can't measure in claims | |
| the discretion of the investigator Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to screening or within the period between screening and randomization | Applied before/after selection of Index dat&efore Assessment window;[-90, 0] Code type:PX Care setting: Any Diagnosis position:Any Source of algorithm:EAD-2 Measurement characteristics:1/a | Applied before/after selection of Index dat@efore Assessment windows[:90, 0] Code type:PX Care setting: Any Diagnosis position:Any Source of algorithm:tEAD-2 Measurement characteristics:1/a | Applied before/after selection of Index date/efore<br>Assessment windowc[-90, 0]<br>Code type:PX<br>Care setting: Any<br>Diagnosis position:Any<br>Source of signothm:EAD-2<br>Measurement characteristics:r/a | We defined it by either Anti-VEGFi injections or<br>Photocoagulation |
| History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g., subtotal and total gastrectomy, sieeve gastrectomy, gastric bypass surgery) | Applied before/after selection of Index datasefore Assessment windows[Start of all available data, 0] Code type;PX Care setting:Any Source of algorithm:PROMISE team Measurement characteristicary/a | Applied before/after selection of Index datelerore Assessment window: [Start of all available data, 0] Code type:P. Care setting:Any Diagnosis position:Any Source of algorithm-RPOMISE team Measurement characteristics://a | Applied before/after selection of index dataerfore<br>Assessment window:[Start of all available data, 0]<br>Code Spect?<br>Care setting:Any<br>Diagnosis position:Any<br>Source of algorithms:PROMISE team<br>Measurement characteristics://a | |
| Age OR Gender Missing | Applied before/after selection of Index dataeriore Assessment windows(=180, 0) Code typen/a Core osting: n/a Diagnosis position:n/a Source of algorithms Measurement characteristics:n/a | Applied before/after selection of Index detectore Assessment window:[-180, 0] Ode type:r/a Care setting: r/a Diagnosis position:r/a Source of sigorithm: Measurement characteristics:r/a | Applied before/after selection of Index dat@efore<br>Assessment windows(:180, 0)<br>Code type:://a<br>Care setting:://a<br>Diagnosis position:://a<br>Source of signothm:<br>Measurement characteristics:://a | Additional criteria |

| Applied before/efter selection Assessment windows[180, Code types) is charged by the code types is charged by the code types is charged by the code types is charged by the code types is charged by the code types is code types in the code types is code to the code types in the code types in the code types is code to the code types in t | Assessment window:[-180, 0] Assessment window:[-180, 0] Code type:Discharge Status Code, CPT/HCPCS Provider Category Code Care setting:Any | Assessment window:[-180, 0] | Additional criteria |
|---|---|---|---|
|---|---|---|---|


DRUG OR CHEMICAL INDUCED DIABETES MELLITUS WITH NEUROLOGICAL COMPLICATIONS WITH DIABETIC AUTONOMIC (POLY)NEUROPATHY

DPP4i, GLP-1, Pramlintide component

DPP4, GLP-1, Pramilitude component DPP4, GLP-1, Pramilitude CDP-1, Pram


II/Stroke/Unstable angina/TIA (inpatient) component II/Stroke/Unstable angina/TIA (inpatient) component /II/Stroke/Unstable angina/TIA (inpatient) component II/Stroke/Unstable angina/TIA (inpatient) component II/Stroke/Unstable angina/TIA (inpatient) component /II/Stroke/Unstable angina/TIA (inpatient) component /II/Stroke/Unstable angina/TIA (inpatient) component II/Stroke/Unstable angina/TIA (inpatient) component /II/Stroke/Unstable angina/TIA (inpatient) component /II/Stroke/Unstable angina/TIA (inpatient) component /II/Stroke/Unstable angina/TIA (inpatient) component

eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component

eart failure class IV component must overlap with oxygen use component

leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component

eart failure class IV component must overlap with oxygen use component

eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component

eart failure class IV component must overlap with oxygen use component

leart failure class IV component must overlap with oxygen use component

eart failure class IV component must overlap with oxygen use component

eart failure class IV component must overlap with oxygen use componen

eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component eart failure class IV component must overlap with oxygen use component leart failure class IV component must overlap with oxygen use component


END-STAGE RENAL DISEASE (ESRD) RELATED SERVICES FOR DIALYSIS LESS THAN A FULL MONTH OF SERVICE, PER DAY; FOR PATIENTS 12-19


component
End stage liver disease (Cirrhosis overlap with Decompensation event) End stage liver disease (Cirrhosis overlap with Decompensation event) component End stage liver disease (Cirrhosis overlap with Decompensation event) component
End stage liver disease (Cirrhosis overlap with Decompensation event) component End stage liver disease (Cirrhosis overlap with Decompensation event) End stage liver disease (Cirrhosis overlap with Decompensation event) component End stage liver disease (Cirrhosis overlap with Decompensation event) component End stage liver disease (Cirrhosis overlap with Decompensation event) component
End stage liver disease (Cirrhosis overlap with Decompensation event) End stage liver disease (Cirrhosis overlap with Decompensation event) component End stage liver disease (Cirrhosis overlap with Decompensation event) component End stage liver disease (Cirrhosis overlap with Decompensation event) component
End stage liver disease (Cirrhosis overlap with Decompensation event) component
End stage liver disease (Cirrhosis overlap with Decompensation event)

component

End stage liver disease (Cirrhosis overlap with Decompensation event)


```
COLLIDANA DI TROCAS DI RETRINO CERRAL ARREY

COLLIDANA DEI TROCAS DI RETRINO CERRAL ARREY

COLLIDANA DEI TROCAS DI PARI ARRES CERRALA, ARREY

COLLIDANA DEI TROCAS DI PARI ARRES CERRALA, ARREY

COLLIDANA DEI TROCAS DI RETRINO ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI CRESSI DI PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PARI ARRES PARI ARRES PARI ARRES

COLLIDANA DEI TROCAS DI PARI ARRES PA
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                     CD-10

Rominian Stockes

Rominian Sto
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                           166.1
166.11
166.12
166.13
166.19
166.2
166.2
166.21
166.23
166.29
166.3
166.3
166.9
20
41
42
21
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                          Modern (Charles)

Modern (Char
```

# Flowchart for Cohort Assembly

Link to Aetion reports:

Semaglutide oral vs Sitagliptin

Marketscan-

https://bwh-dope.aetion.com/project/2322/cohort/59481/116372/comparative/basics 8/2/24

Optum

https://bwh-dope.aetion.com/project/2321/cohort/59483/116374/comparative/basics 8/2/24

Medicare-

https://bwh-dope.aetion.com/project/2323/cohort/59485/116376/comparative/basics 8/2/24

| | | Optum<br>(Sept 20, 2019 and Feb 29, 2024) | | Marketscan<br>(Sept 20, 2019 and December 31,<br>2021) | | are<br>ad December<br>20) |
|---|---|---|---|---|---|---|
| | Less Excluded | • | | Remaining | Less Excluded | Remaining |
| | Patients | Patients | Patients | Patients | Patients | Patients |
| Patients in dataset | | 93,159,383 | | 119,592,975 | | 28,874,258 |
| Patient with cohort entry criteria (Exposure: Semaglutide oral, Refrence: Sitaglitpin) | | | | | | |
| Date of dispensing is cohort entry date (CED, 0,0) | | 430,611 | | 338,596 | | 598,543 |
| Excluded due to insufficient enrollment (30 day gap allowed) (-180, 0) | -63,623 (15%) | 366,988 | -33,728 (10%) | 304,868 | -132,618 (22%) | 465,925 |
| Exclude due to prior use of reference (-180, -1) | -216,331 (59%) | 150,657 | -214,382 (70%) | 90,486 | -400,547 (86%) | 65,378 |
| Exclude due to prior use of reference (-180, -1) | -58,267 (39%) | 92,390 | -39,790 (44%) | 50,696 | -3,934 (6%) | 61,444 |
| Excluded because patient qualified in >1 exposure category | -24 (<1%) | 92,366 | -9 (<1%) | 50,687 | -4 (<1%) | 61,440 |
| Excluded based on Inclusion: Type 2 DM (-180, 0) | -5,932 (6%) | 86,434 | -6,322 (12%) | 44,365 | -1,374 (2%) | 60,066 |
| Excluded based on Inclusion: >=50 years with established CVD OR >=60 years with subclinical CVD (-180, 0) | | | | | . , , | * |
| Exclude if patient is between 50 and 60 years of age without established CVD | -4,631 (5%) | 81,803 | -10,219 (23%) | 34,146 | -0 (<1%) | 60,066 |
| Exclude if patient is greater than or equal to 60 years of age without established or subclinical CVD | -26,643 (33%) | 55,160 | -10,559 (31%) | 23,587 | -21,316 (35%) | 38,750 |
| Excluded based on Age (<=49 years) | -3,461 (6%) | 51,699 | -8,665 (37%) | 14,922 | -0 (<1%) | 38,750 |
| Excluded based on Exclusion: Use of Sitagliptin/Semaglutide [any formulations/combinations] (-180, -1) | -3,464 (7%) | 48,235 | -1,123 (8%) | 13,799 | -3,691 (10%) | 35,059 |
| Excluded based on Exclusion: Type 1 DM (-180, 0) | -545 (1%) | 47,690 | -196 (1%) | 13,603 | -657 (2%) | 34,402 |
| Excluded based on Exclusion: Gestational DM (-180, 0) | -0 (<1%) | 47,690 | -0 (<1%) | 13,603 | -0 (<1%) | 34,402 |
| Excluded based on Exclusion: Secondary DM (-180, 0) | -497 (1%) | 47,193 | -129 (<1%) | 13,474 | -581 (2%) | 33,821 |
| Excluded based on Exclusion: Pramlintide, Other DPP4i/GLP1 (-180, 0) | -1,935 (4%) | 45,258 | -602 (4%) | 12,872 | -1,536 (5%) | 32,285 |
| Excluded based on Exclusion: Diabetic ketoacidosis (-90, 0) | -82 (<1%) | 45,176 | -25 (<1%) | 12,847 | -74 (<1%) | 32,211 |
| Excluded based on Exclusion: History of pancreatitis (-180, 0) | -105 (<1%) | 45,071 | -24 (<1%) | 12,823 | -115 (<1%) | 32,096 |
| Excluded based on Exclusion: MI/Stroke/Angina/TIA (-60, 0) | -529 (1%) | 44,542 | -262 (2%) | 12,561 | -628 (2%) | 31,468 |
| Excluded based on Exclusion:Heart failure class IV (-180, 0) | -119 (<1%) | 44,423 | -21 (<1%) | 12,540 | -0 (<1%) | 31,468 |
| Excluded based on Exclusion: History of MEN-2 (-180, 0) | -0 (<1%) | 44,423 | -0 (<1%) | 12,540 | -1 (<1%) | 31,467 |
| Excluded based on Exclusion: End-stage renal disease (-180, 0) | -336 (<1%) | 44,087 | -91 (<1%) | 12,449 | -408 (1%) | 31,059 |
| Excluded based on Exclusion: End stage liver disease (-180, 0) | -51 (<1%) | 44,036 | -11 (<1%) | 12,438 | -68 (<1%) | 30,991 |
| Excluded based on Exclusion: Organ transplant (-180, 0) | -28 (<1%) | 44,008 | -13 (<1%) | 12,425 | -29 (<1%) | 30,962 |
| Excluded based on Exclusion: Cancer (-1825, 0) | -2,383 (5%) | 41,625 | -612 (5%) | 11,813 | -3,099 (10%) | 27,863 |
| Excluded based on Exclusion: Pregnancy (-180, 0) | -1 (<1%) | 41,624 | -1 (<1%) | 11,812 | -3 (<1%) | 27,860 |
| Excluded based on Exclusion: Proliferative retinopathy or maculopathy (-90, 0) | -252 (<1%) | 41,372 | -73 (<1%) | 11,739 | -231 (<1%) | 27,629 |
| Excluded based on Exclusion: Nursing home stay (-180, 0) | -379 (<1%) | 40,993 | -18 (<1%) | 11,721 | -635 (2%) | 26,994 |
| Excluded based on Exclusion: Bariatric surgery (all avail data, 0) | -45 (<1%) | 40,948 | -54 (<1%) | 11,667 | -54 (<1%) | 26,940 |
| Excluded based on Exclusion: Missing Age (-180, 0) | -0 (<1%) | 40,948 | -0 (<1%) | 11,667 | -0 (<1%) | 26,940 |
| Excluded based on Exclusion: Missing Gender (-180, 0) | -1 (<1%) | 40,947 | -0 (<1%) | 11,667 | -0 (<1%) | 26,940 |
| Patients in Exposure Group | | 11,103 | | 2,515 | | 1,153 |
| Patients in Referent Group | | 29,844 | | 9,152 | | 25,787 |
| Total Patients | | 40,947 | | 11,667 | | 26,940 |

| | | - COLOR | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | - | - | | - | | | - |
| | 46774 | auti's | 6+8 | 100 | 1642 | 1-1 | HCM2 | TT NE | 1.1 |
| metar (68) | 1400 (680), 79/00 | \$100 (80.00,7500) | 6+8 | 6620 (6030,7620) | enterior and | 1-1 | See (Teas seed) | Section (Text) | 1.1 |

| | No. | | The state of |
|---|---|---|---|
| | | 750 | - |
| Number of patients dropped as<br>incomplete upper. | 0 | 0 | 0 |
| Number of patients that stat not<br>impin follow-up | 100 | 29 | |
| Number of patients in analysis<br>rathers | 40,845 | 11,638 | 26,860 |
| | 1112 | 240 | |
| | | 1,201.84 | |
| Number of patients in group:<br>Reference Staglistin | 26,774 | 9,126 | 26,712 |
| Sunter of patients in group<br>Survives Semestatist and | 11,071 | 2,812 | 1,148 |

| iyad isint iyada | 188 (68, 268) | 118 (18, 268) | EUR [58, 000] |
|---|---|---|---|
| D. Proposition Consuming to the | - | • | |
| | | 100 | |
| Const | | Yeles | - |
| | | | 424-13.84 |
| | 344 (0.8%) | | 66 (0.2%) |
| To dept. grant & this workers) | 24,714 (63.2%) | 6,386 (66.4%) | 10,060 (37.4%) |
| Maximum Indian say time (2011 steps) | 6,628 (36.24) | T-936-(EE-61) | 4,733 (6.6%) |
| Coll of patient amalinant | 3,028 (7.4%) | 1,882 (13.7%) | 720 (3.7%) |
| Panistin, Ohr-SPA, G.P.L<br>Hamistin, Ohr-SPA, G.P.L<br>Halling In Earney + Kursing home | 3,208 (7.8%) | 732 (6.3%) | E-601 (6.1%) |

| - | | | | | | | |
|---|---|---|---|---|---|---|---|
| Number of patients, matched | | furnise of patients | | distributed for materials | | Number of patients matched | |
| Nelsonar | 58,151 | Selevene | 58,151 | Selevanos | 58,014 | Selevence | 95.0 |
| | | | | | | | 40 |
| Risk per 1,000 patients | 27.84 | Risk per 1,000 patients. | 27.84 | dala per 1,000<br>palaria | 27.84 | Risk per I,000 partents | 21 |
| Central All Eryn ACT | 9.76 | Genised HE from NCT | 6.6 | Concret HR from RCT | 0.86 | Grained HR how RCT | _ |
| tida Custed | 2.00 | Service Colors | 0.00 | tary 2 costs | 0.00 | fatur 2 scient | |
| Survive of events expected | 2016.0 | Surviver of exercis | 2096.6 | Number of Avents | 2006.6 | Sunter of events, experted | 201 |
| | | | - | | | | |
| Number of patents matched | | Sumber of patients<br>matched | | Number of patients<br>matched | | Number of patients matched | |
| Patienerus | 14,10 | | 14,112 | Selevense | 14.03 | Televise | |
| | | Daniel | | Sancel | | Europe | 10.0 |
| | | Risk per X,000 patients. | 27.64 | fish per 5,000<br>outliers | 27.64 | Mais per 1,000 patients | 21 |
| flish per 1,000 patients | 27.64 | | | | | | |
| Daziel of the NCT | 9.75 | Section 18 Four SCT | | Desired HR hard RCT | | Section 14th horse BCT | |
| | 9.75 | Sector of Four NCT<br>Spin (2 name) | | Spins (Faller) | | Sphar Gradesh | |
| Daziel of the NCT | 9.75 | | | | 0.00 | | |

The second secon

| <br>- | - | - 100 i |
|---------------|---------------|---------------|
| 116 (68, 268) | 118 (68, 268) | 118 (NR, 206) |

| | | Trees | - Hoters |
|---|---|---|---|
| Number of patients in<br>full colors | 40,847 | 11,647 | 26,660 |
| Standar of patients,<br>depped as incomplete<br>cases. | 0 | | 0 |
| Standar of patients<br>that sixt not legin<br>below up | 100 | 29 | ac . |
| Number of patients in<br>analytic colors | 40,845 | 11,638 | 24,860 |
| Number of events | 1182 | 243 | 826 |
| Number of person. | 16,716.60 | 1,203.86 | 10,847.60 |
| Sunder of patients in<br>group Entereum<br>Stantage | 29,776 | 9,126 | 29,712 |
| Number of patients in<br>group Expenses<br>Semeglatein and | 11,071 | 2,812 | 1,148 |
| Risk per 1,000 | 28.2 | 20.62 | 30.71 |
| Nation per 1,000 | 61.55 | 46.12 | TH.33 |

| | | - | |
|---|---|---|---|
| | 1,182 (2.8%) | 262 (2.2%) | 828 (3.1%) |
| Start of an additional<br>manager | 314 (0.8%) | #1 (6.7%) | 88 (0.2%) |
| End of Index exposure<br>(30 days glace & dub<br>scordina) | 21,714 (83.2%) | 1,391 (41.4%) | 13,080 (37.4%) |
| Washingto Miller up<br>time (265 days) | 6,628 (36.2%) | 1,896 (36.6%) | 1,733 (6.8%) |
| Draft of patient data: | 4,800 (11.8%) | 1,662 (16.3%) | 11,837 (44.2%) |
| Sni of patient<br>explorers | 3,028 (7.4%) | 1,882 (13.7%) | 729 (2.7%) |
| Edia senson<br>Medications<br>(Pransistials/Other<br>OPPO/GLPS including<br>inj Sensoj + Numbry<br>home legion | 3,209 (7.8%) | 732 (6.3%) | 1,631 (6.2%) |



| | najmi (ina ana) | | (march ) | | (بعبد) خرید | | · independent |
|---|---|---|---|---|---|---|---|
| Yumber of patients,<br>matched | | Surviver of patients,<br>matched | | Sumber of patients<br>matched | | partients. | |
| | | Relevance | | Reference | | Relevence | 62,11 |
| Descri | 16,721 | Description | 14.701 | Description | 14.700 | Donald | 14.7 |
| Risk per 1,000 patients | 27.94 | Risk per 1,000 patients. | 27.84 | Rab per 1,000<br>patients | 27.84 | Rinals perv<br>1,000 percentin | 27.0 |
| Ominel HR fem RCT | 6.76 | Ominal HR term BCT | 0.8 | Organic Hill Street RCT | 0.85 | Sested HR<br>from RCT | |
| Sphe (2 sales) | 0.08 | Apha (2 sides) | 0.08 | Byte (2 sales) | 0.08 | April (2 scient) | 0.0 |
| Yumber of events<br>expected | 2047.1 | Survier of morris<br>represent | 2147.1 | Number of evenin<br>experient | 2147.1 | | 2147 |
| Property. | 1.0 | Preser. | 1.0 | Person. | 1.0 | Frame | • |
| | | | | | القضفة | | |
| Number of patients<br>matched | Andrea (L.) | Sunday of patients<br>matched | | Sunder of patients<br>matched | | Complete of<br>patients | - |
| Selector | | Selector | | Selector | 13.063 | Believes | 13.06 |
| Equipme | | Esperanti | | Equani | | Especial | 11.00 |
| Risk per 1,000 patients | 21.94 | fish per 1,000 petients | 27.84 | Rink per 1,000<br>patients | 27.84 | Rinals perv<br>1,000 patientis | 20.4 |
| | | | | TOR mort RH (enriged) | 0.85 | | |
| Ominel HR fem SCT | | Comment HR from RCT | | | | | |





## fine-stratified cstats, Optum: 0.50016



| Summary, PS distribution, Unadjusted cohort | | | | | | |
|---|---|---|---|---|---|---|
| OPTUM | Minimum Maximum Mean Median 25th pct 75th pct | | | | | |
| Reference | 1.76E-05 | 0.954 | 0.215 | 0.175 | 0.0683 | 0.324 |
| Exposure | 0.000869 | 0.948 | 0.422 | 0.415 | 0.279 | 0.56 |

| | Summary, PS distribution, 1:1 cohort | | | | | |
|---|---|---|---|---|---|---|
| OPTUM | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.000867 | 0.909 | 0.385 | 0.383 | 0.259 | 0.501 |
| Exposure | 0.000869 | 0.907 | 0.385 | 0.383 | 0.259 | 0.503 |

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| OPTUM | TUM Minimum Maximum Mean Median 25th pct 75th pct | | | | | |
| Reference | 0.0844 | 10.4 | 1 | 0.579 | 0.253 | 1.21 |
| Exposure | 1 | 1 | 1 | 1 | 1 | 1 |

## fine-stratified cstats, Marketscan: 0.50005



| Summary, PS distribution, Unadjusted cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.00000384 | 0.869 | 0.176 | 0.132 | 0.051 | 0.261 |
| Exposure | 0.00666 | 0.914 | 0.361 | 0.345 | 0.217 | 0.492 |

| Summary, PS distribution, 1:1 cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN Minimum Maximum Mean Median 25th pct 75th pct | | | | | | |
| Reference | 0.00669 | 0.799 | 0.335 | 0.324 | 0.208 | 0.45 |
| Exposure | 0.00666 | 0.798 | 0.335 | 0.324 | 0.208 | 0.451 |

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| MARKETSCAN Minimum Maximum Mean Median 25th pct 75th pct | | | | | | |
| Reference | 0.0734 | 9.29 | 1 | 0.552 | 0.0734 | 1.33 |
| Exposure 1 1 1 1 1 1 | | | | | | |

## fine-stratified cstats, Medicare: 0.49995



| Summary, PS distribution, Unadjusted cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE Minimum Maximum Mean Median 25th pct 75th pct | | | | | | |
| Reference | 0.00000806 | 0.615 | 0.0386 | 0.0139 | 0.00357 | 0.051 |
| Exposure | 0.000597 | 0.786 | 0.137 | 0.112 | 0.0589 | 0.185 |

| Summary, PS distribution, 1:1 cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.000597 | 0.575 | 0.124 | 0.105 | 0.0562 | 0.172 |
| Exposure | 0.000597 | 0.575 | 0.124 | 0.105 | 0.0562 | 0.172 |

| Summary, PS WEIGHT distribution, fine-stratifed cohort | | | | | | |
|---|---|---|---|---|---|---|
| MEDICARE | Minimum | Maximum | Mean | Median | 25th pct | 75th pct |
| Reference | 0.055 | 15.9 | 1 | 0.427 | 0.055 | 1.16 |
| Exposure | 1 | 1 | 1 | 1 | 1 | 1 |

| Variable<br>Number of patients | Optun<br>Sitagliptin - reference<br>29,741 | n: Unadjusted cohort<br>Semaglutide - exposure<br>11,050 | Stddiff | Optum<br>Stagliptin - reference<br>9,670 | 11 matched cohort<br>Semaglutide - exposure | 2467 | Optum: F<br>Stagliptis - reference<br>28,581 | Ine stratification cohort<br>Semaglutide - exposure<br>11,049 | Stddff | Market:<br>Sitagliptin - reference<br>9,100 | Semaglutide - exposure | Std dVT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age<br>mean (ud)<br>Gender | 73.69 (7.96) | 69.58 (8.00) | 0.514 | 70.60 (7.50) | 20.47 (7.75) | 0.018 | 69.76 (7.70) | £9.58 (8.00) | 0.022 | 68.26 (10.64) | 63.00 (8.44) | 0.547 |
| Female; n (%) Region Northeast; n (%) | 15421 (51.9)<br>3729 (12.5) | 5405 (48.9)<br>1007 (9.1) | 0.059 | 4779[49.4]<br>949 (9.8) | 4812 (49.8)<br>946 (9.8) | 0.005 | 14037 (49.1)<br>2624.4 (9.2) | 5405 [48.9]<br>1007.0(9.1) | 0.004 | 2081 (22.9) | 987 (39.3)<br>386 (15.4) | 0.065 |
| Midwest/North central; n (%)<br>South; n (%)<br>West: n (%) | 4827 (16.2)<br>16147 (54.3)<br>5038 (16.9) | 2051 (18.6)<br>6104 (55.2)<br>1888 (17.1) | | 1749 [18.1]<br>5317 [55.0]<br>1655 [17.1] | 1759 (18.2)<br>5328 (55.1)<br>1637 (16.9) | | 5238.7 (18.3)<br>15810.1 (55.3)<br>4907.9 (17.2) | 2051.0(18.6)<br>6104.0(55.2)<br>1887.0(17.1) | | 2932 [32.2]<br>3543 [38.9]<br>544 (6.0) | 565 (22.5)<br>1342 (53.4)<br>218 (8.7) | |
| Near of cohort entry<br>2019 (Sept-Osc); n (%)<br>2020 (Jan-March); n (%) | 1978 (6.7)<br>2042 (6.9) | 2 (0.0)<br>74 (0.7) | 0.78 | 2 (0.0) | 2 (0.0)<br>74 (0.0) | 0.024 | 69.5 (0.2)<br>214.6 (0.8) | 1.0(0.0)<br>74.0 (0.7) | 0.07 | 1136 (12.5)<br>859 (9.4) | 27 (1.1)<br>82 (2.3) | 0.703 |
| 2020 (April-June); n (N)<br>2020 (July-Sept); n (N)<br>2020 (Oct-Oec'; n (N) | 1796 (6.0)<br>1858 (6.2)<br>1737 (5.8) | 130 (1.2)<br>231 (2.1)<br>271 (3.4) | | 111 (1.1)<br>226 (2.3)<br>329 (3.5) | 130 (1.3)<br>231 (2.4)<br>361 (2.7) | | 290.1 (1.0)<br>546.2 (1.9)<br>949.8 (3.3)<br>5625.8 (19.7) | 130.0 (1.2)<br>231.0 (2.1)<br>171.0 (3.4) | | 679 (7.5)<br>818 (9.0)<br>835 (9.2) | 90 (3.6)<br>128 (5.1)<br>185 (7.4) | |
| 2021 (Jan-Dec); n (Ki)<br>2022 (Jan-Dec); n (Ki)<br>2023 (Jan-Dec); n (Ki) | 7292 (24.5)<br>6048 (20.3)<br>5887 (19.8) | 271 (2.4)<br>2204 (19.9)<br>2922 (26.4)<br>4256 (29.4) | | 2099 (21.7)<br>2633 (27.2)<br>2632 (26.7) | 2100 (21.7)<br>2594 (26.8)<br>2547 (36.7) | | \$625.8 (19.7)<br>7582.1 (26.5)<br>11158.5 (19.7)<br>1944.4 (6.8) | 2204.0 (19.9)<br>2922.0 (26.4)<br>4356.0 (29.4) | | 2673 (29.4)<br>2100 (23.1) | 919 (36.6)<br>1079 (43.0) | |
| 2024 (Jan - Feb); n (%)<br>Drug abuse or dependence; n (%)<br>Alcohol abuse or dependence; n (%) | 1113 (3.7)<br>736 (2.5)<br>435 (1.5) | 760 (6.9)<br>264 (2.4)<br>142 (1.3) | 0.006 | 2633 [27.2]<br>2633 [27.2]<br>2552 [26.7]<br>638 [6.6]<br>244 [2.5]<br>129 [1.3]<br>221 [2.3] | 631 (6.5)<br>231 (2.4)<br>122 (1.3) | 0.009 | 1944.4 (E.B)<br>663.6 (2.3)<br>365.7 (1.3) | 762.0 (6.9)<br>264.0 (2.4) | 0.004 | 121(1.3) | 23 (0.9) | 0.019 |
| Underweight or normal weight; n (%) Dierweight; n (%) Obese: n (%) | 1134(4.5)<br>1101(10.4)<br>4571(15.4) | 228 (2.1)<br>1011 (9.1)<br>2168 (19.6) | 0.136<br>0.043<br>0.112 | 221 (2.3)<br>879 (9.1)<br>1793 (18.5) | 221 (2.3)<br>916 (9.5)<br>1824 (18.9) | 0.001 | 663.6 (2.3)<br>365.7 (1.3)<br>620.9 (2.2)<br>2649.9 (9.3)<br>5687.1 (19.9) | 228.0 (2.1)<br>1011.0(9.2)<br>2168.0(19.6) | 0.008 | 232 (2.5)<br>741 (8.1)<br>866 (9.5) | 25 (1.0)<br>342 (5.7)<br>285 (11.4) | 0.118<br>0.097<br>0.06 |
| Severe obesity, n (%) Unspecified obesity, n (%) Smokingr a (%) | 2270(11.3)<br>2726(12.6)<br>6086(20.5) | 2337 (21.1)<br>2012 (18.2)<br>2143 (19.4) | 0.269<br>0.157<br>0.022 | 1792 (18.5)<br>1721 (17.8)<br>1575 (16.3)<br>1910 (19.8) | 1775 (18.4)<br>1600 (16.5)<br>1878 (19.4) | 0.008<br>0.015<br>0.007 | 5881.0 (20.4)<br>5139.4 (18.0)<br>5707.3 (20.0) | 2337.0(21.2)<br>2012.0(18.2)<br>2143.0(19.4) | 0.007<br>0.014<br>0.006 | 1015 (11.2)<br>1277 (14.0) | 642 (17.6)<br>478 (19.0)<br>220 (8.8) | 0.185<br>0.135<br>0.056 |
| Diabetic retinopathy; n (%) Diabetic neuropathy; n (%) | 2681 (9.0)<br>8803 (29.6) | 963 (8.7)<br>2035 (27.5) | 0.011<br>0.047<br>0.047 | | 843 (8.7)<br>2671 (27.6) | 0.006<br>0.018<br>0.018 | 2551.0 (8.9) | 963.0 (8.7) | 0.007<br>0.026<br>0.026 | 621 (6.8)<br>2004 (22.0) | 141 (5.6)<br>456 (18.2) | 0.05<br>0.096<br>0.096 |
| Diabetes with unspecified complications; n (%) Diabetes with other ophthalmic complications; n (%) | 8803 (29.6)<br>6391 (21.5)<br>1402 (4.7)<br>5877 (19.8) | 2429 (22.0)<br>2429 (22.0)<br>645 (4.0)<br>1903 (17.2) | 0.012<br>0.034<br>0.065 | 2749(28.4)<br>2749(28.4)<br>2135(22.1)<br>404(4.2)<br>1696(17.5) | 2118 (21.9)<br>409 (4.2) | 0.004<br>0.003<br>0.005 | 8187.7 (28.6)<br>8187.7 (28.6)<br>6277.8 (22.0)<br>1175.9 (4.1)<br>4983.9 (17.4) | 1034.0(27.5)<br>1034.0(27.5)<br>2429.0(22.0)<br>445.0 (4.0)<br>1901.0(17.2) | 0.001 | 1106 (12.2)<br>1162 (1.8) | 456(18.2)<br>385(15.3)<br>38(1.5)<br>285(11.4) | 0.092 |
| Diabetic floor + Lower extremity amputation; n (N) Skin infections; n (N) | 765 (2.6)<br>1811 (6.1) | 245 (2.2)<br>660 (6.0) | 0.023 | 590 (5.0) | 1679 (17.4)<br>207 (2.1)<br>561 (5.8) | 0.008 | 1744.1 (6.1) | 660.0 (6.0) | 0.007 | 1086 (11.9)<br>203 (2.2)<br>612 (6.7) | 28 (1.5)<br>156 (6.2) | 0.053 |
| Erectile dysfunction; n (%) Hypoglycemix; n (%) Hyperglycemia, DKA, HONK; n (%) | 726 (2.4)<br>6484 (21.8)<br>11065 (43.9) | 280 (2.4)<br>2389 (21.6)<br>5038 (45.6) | 0.059<br>0.004<br>0.023<br>0.046<br>0.029 | 216 (2.3) | 307 (3.2)<br>2088 (21.6)<br>4344 (44.9) | 0.005<br>0.002<br>0.003<br>0.012<br>0.007 | 932.4 (3.3)<br>6163.2 (21.6)<br>13178.3 (46.1) | 2389.0(21.6)<br>5028.0(45.6) | 0.01<br>0.001<br>0.01<br>0.007<br>0.009 | 199 (2-2)<br>1115 (12-3)<br>3781 (41-5) | 80 (3.2)<br>370 (14.7)<br>1164 (46.4) | 0.062<br>0.073<br>0.097<br>0.044<br>0.06 |
| Hypertension; n (%)<br>Hyperlipidemix; n (%)<br>Atrial fibrillation; n (%) | 13065 (43.9)<br>27084 (91.1)<br>24329 (81.8)<br>4678 (15.7)<br>244 (2.5) | 5038(45.6)<br>9912(89.7)<br>9163(82.9)<br>1375(12.4)<br>281 (2.5) | 0.046<br>0.029<br>0.095<br>0.003 | 2034 (21.7)<br>4258 (45.1)<br>8675 (89.7)<br>7995 (82.7)<br>1255 (13.0)<br>229 (2.5) | 8711 (90.1)<br>8019 (82.9)<br>1257 (13.0)<br>234 (2.4) | 0.012<br>0.007<br>0.001<br>0.003 | 25703.9 (89.9)<br>23793.5 (83.2)<br>3622.6 (32.7)<br>720.8 (2.5) | 9911.0(89.7)<br>9162.0(82.9)<br>1375.0(12.4)<br>281.0 (2.5) | 0.007<br>0.009<br>0.007<br>0.001 | 7957 (87.4)<br>7148 (78.5)<br>1210 (13.3)<br>200 (3.3) | 2158 (BS.9)<br>2023 (B1.0)<br>253 (20.1)<br>100 (4.0) | 0.044<br>0.06<br>0.1 |
| Acute M; n (%) Old M; n (%) Consnay atheroscienosi; n (%) | 744 (2.5)<br>2084 (7.0)<br>12438 (41.8) | 281 (2.5)<br>705 (6.4)<br>4754 (43.0) | 0.025 | 229 (2.5)<br>624 (6.5)<br>6239 (41.8) | 234 (2.4)<br>616 (6.4)<br>4080 (42.2) | 0.003 | 720.8(2.5)<br>1860.2 (6.5)<br>12221.4 (42.8) | 281.0 (2.5)<br>705.0 (6.4)<br>4754.0 (43.0) | 0.005 | 300 (3.3)<br>396 (4.4)<br>4371 (48.0) | 100 (4.0)<br>122 (4.9)<br>1318 (52.5) | 0.027<br>0.024<br>0.089 |
| Nistory of CASG/PTCA; n (N) Previous cardiac procedure; n (N) Cerebrowacular procedure; n (N) | 3859 (13.0)<br>456 (1.5) | 1378(12.5)<br>180 (1.6) | 0.015<br>0.015<br>0.008 | 1185(12.3)<br>141(1.5) | 1188 (12.3)<br>149 (1.5) | 0.005 | 3605.5 (12.6)<br>469.6 (1.6) | 1378.0(12.5)<br>180.0(1.6) | 0.005<br>0.004<br>0.001<br>0.003 | 612 (6.7)<br>202 (2.2) | 198 (7.9)<br>62 (2.5) | 0.016 |
| Ischemic stroke; n (%) PVD disposition surgery; n (%) CVD Street 2-6 - n (%) | 34 (0.1)<br>4204 (14.5)<br>5580 (18.8) | 9 (D.1)<br>1402 (12.7)<br>1749 (15.8) | 0.052<br>0.078<br>0.092 | 8 (0.1)<br>1264 (13.1)<br>1620 (16.8) | 9 (0.1)<br>1263 (13.1)<br>1586 (16.4) | 0.001<br>0.009<br>0.001 | 26.2 (0.1)<br>3728.6 (13.0)<br>4585.2 (16.0)<br>10065.7 (15.2) | 9.0 (0.1)<br>1402.0 (12.7)<br>1749.0 (15.8)<br>3827.0 (34.6) | 0.001<br>0.001<br>0.006<br>0.012 | 6 (0.1)<br>1294 (14.2)<br>1288 (14.2) | 2 (0.1)<br>287 (11.4)<br>269 (10.7) | 0.005<br>0.084<br>0.104 |
| Other cardiac dyshythmia; n (K) Cardiom yopathy; n (K) | 5580(18.8)<br>11619 (29.1)<br>6233 (21.0)<br>2431 (8.2) | 1749 [15.8]<br>2827 (24.6)<br>2066 [18.7)<br>828 (7.5) | 0.057 | 1620(16.8)<br>2456(15.7)<br>1800(18.6)<br>711 (7.4) | 1455 (15.7)<br>1814 (18.8)<br>715 (7.4) | 0.004 | 5441.9 (19.0)<br>2186.6 (7.7) | 2066.0(18.7)<br>828.0 (7.5) | 0.009 | 2385 (26.2)<br>1773 (19.5)<br>715 (7.9) | 269 (10.7)<br>548 (21.8)<br>403 (16.0)<br>209 (8.3) | 0.09 |
| COPG; n (%) Asthma; n (%) | 1043 (3.5)<br>6092 (20.5)<br>2008 (6.8) | 297 (2.7)<br>1948 (17:6)<br>819 (7:4) | 0.047<br>0.072<br>0.026 | 263 (2.7)<br>1765 (18.3)<br>711 (7.4) | 272 (2.8)<br>1749 (18.1)<br>690 (7.1) | 0.006<br>0.004<br>0.008 | 813.4(2.8)<br>5353.3 (18.7)<br>2136.5 (7.5) | 297.0 (2.7)<br>1948.0 (17.6)<br>819.0 (7.4) | 0.01<br>0.029<br>0.002 | 229 (2.5)<br>1342 (14.7)<br>455 (5.0) | 45 (1.8)<br>286 (11.4)<br>146 (5.8) | 0.05<br>0.1<br>0.036 |
| Obstructive sleep apnea; n (N) Pneumonia; n (N) CXD Stage 1-2; n (N) | 4291 (14.4)<br>1575 (5.3)<br>1778 (6.0) | 2354(21.3)<br>362(3.3)<br>583(5.3) | 0.1 | 1870 (19.3)<br>258 (2.7)<br>537 (5.6)<br>524 (5.4)<br>2 (9.0) | 1898 (19.6)<br>133 (2.4)<br>519 (5.4) | 0.007<br>0.014<br>0.008<br>0.007<br>0.008 | 6120.2 (21.4)<br>999.1 (3.5)<br>1525.7 (5.3) | 2354.0(21.3)<br>361.0 (3.3)<br>583.0 (5.3) | 0.003<br>0.013<br>0.003<br>0.008 | 1621 (17.8)<br>428 (4.8)<br>240 (2.6) | 581 (23.1)<br>75 (3.0)<br>67 (2.7) | 0.132<br>0.094<br>0.002 |
| Acute renal disease (AO); n (%)<br>Nephrotic syndrome; n (%)<br>Hypertensive nephropathy; n (%) | 7 (0,0) | 557 (5.0)<br>1 (0.0)<br>2172 (19.7)<br>7120 (54.4) | 0.011<br>0.012<br>0.092 | 524 (5.4)<br>2 (0.0)<br>1953 (20.2) | 1 (0.0) | 0.007<br>0.008<br>0.005 | 1492.5 (5.2)<br>1.9 (0.0)<br>5712.1 (20.0)<br>18685.4 (65.4) | 557.0 (5.0)<br>1.0 (0.0)<br>2172.0 (19.7)<br>7120.0 (64.4) | 0.008<br>0.003<br>0.008 | 2 (0.0) | 92 (2.7)<br>0(0.0)<br>284 (11.3)<br>1453 (57.9) | 0.17<br>0.021<br>0.106 |
| Other renal conditions; n (%)<br>Liver disease; n (%)<br>Hispathyroidism: n (%) | 8965 (23.4)<br>19505 (65.6)<br>3469 (11.7)<br>5788 (19.5) | 7120(64.4)<br>1294(11.7)<br>1949(17.6) | 0.024<br>0.001<br>0.047 | 1953(20.2)<br>6230(64.4)<br>1115(11.5)<br>1765(18.3) | 1971 (20.4)<br>6249 (64.6)<br>1120 (11.6)<br>1721 (17.8) | 0.004<br>0.002<br>0.012 | 18685.4 (65.4)<br>3351.3 (11.7)<br>5104.7 (17.9) | 7120.0(64.4)<br>1294.0(11.7)<br>1948.0(17.6) | 0.02 | \$169 (\$6.8)<br>\$08 (\$0.0)<br>\$419 (\$5.6) | 3453 (57.9)<br>232 (9.2)<br>330 (13.1) | 0.021<br>0.025<br>0.07 |
| Osteoarthritis; n (%) Fracture; n (%) | 6804 (22.9)<br>569 (1.9) | 2428(22:0)<br>153 (1:4) | 0.022<br>0.042<br>0.085 | 2127 (22.0)<br>135 (1.4) | 2110 (21.8)<br>127 (1.4) | 0.004 | 6414.6 (22.4)<br>403.3 (1.4) | 2428.0(22.0)<br>153.0(1.4) | 0.011 | 1480 (16.3)<br>152 (1.7) | 373 (14.9)<br>28 (1.1) | 0.039 |
| Ostroporosis; n (%) Depression; n (%) | 1270 (4.3)<br>1580 (5.3)<br>4928 (16.6) | 200 (2.7)<br>429 (2.9)<br>1613 (14.6)<br>1444 (13.1)<br>2777 (25.1) | 0.068 | 270 (2.8)<br>406 (4.2)<br>1416 (14.6) | 285 (2.9)<br>288 (4.0)<br>1419 (14.7) | 0.009<br>0.001<br>0.008 | 839.8(2.9)<br>1161.2 (4.1)<br>4216.2 (14.8) | 200.0 (2.7)<br>429.0 (2.9)<br>1613.0 (14.6) | 0.002<br>0.013<br>0.009<br>0.004 | 292 (3.2)<br>211 (2.3)<br>942 (10.4) | 65 (1.8)<br>64 (1.8)<br>242 (9.6)<br>243 (9.7)<br>405 (16.1) | 0.04<br>0.024<br>0.001 |
| Accesty, n (%) Sieep disorder, n (%) Dementia; n (%) | 1580 (5.3)<br>4928 (16.6)<br>3818 (12.8)<br>7516 (25.3)<br>2745 (9.2) | 397 (3.6) | 0.007<br>0.003<br>0.232 | 805 (4.2)<br>1416 (14.6)<br>1275 (13.2)<br>2378 (24.6)<br>371 (3.8) | 1248 (12.9)<br>2393 (24.7)<br>387 (4.0) | 0.004 | 1161.2 (4.1)<br>4216.2 (14.8)<br>1825.3 (12.4)<br>7380.6 (25.5)<br>1047.8 (2.7) | 1644.0(13.1)<br>2777.0(25.1)<br>197.0 (1.6) | 0.009<br>0.009<br>0.004 | 880 (9.7)<br>1523 (16.7)<br>480 (5.3) | 33 (1.3) | 0.016 |
| Delinium; n (N)<br>COVID; n (N)<br>Number of antidiabetic drugs | 700 (2.4)<br>1477 (5.0) | 95 (0.9)<br>584 (5.3) | 0.016 | 534 (5.5) | 89 (0.9)<br>508 (5.3) | 0.011 | 1484.4 (5.2) | 96.0 (0.9)<br>584.0 (5.3) | 0.001 | 193 (2.1)<br>425 (4.7) | 16 (0.6)<br>160 (6.4) | 0.127 |
| mean (sd)<br>Insulint; n (%)<br>Meglitinides; n (%) | 1.20 (0.86)<br>4842 (16.3)<br>204 (1.0) | 1.24 (0.92)<br>1909 (17.3)<br>109 (1.0) | 0.05<br>0.027<br>0.004 | 1.25 (0.88)<br>1679(17.4)<br>92(1.0) | 1.24 (0.91)<br>1633 (16.9)<br>92 (1.0) | 0.011<br>0.013<br>0.001<br>0.012 | 1.26 (0.90)<br>5247.9 (18.4)<br>280.7 (1.0)<br>9690.0 (23.9) | 1.24 (0.92)<br>1909.0 (17.3)<br>109.0 (1.0)<br>3617.0 (32.7) | 0.024<br>0.028<br>0.001<br>0.025 | 1.12 (0.86)<br>1320 (14.5)<br>113 (1.2) | 1.28 (0.91)<br>445 (17.7)<br>19 (0.8) | 0.176<br>0.068<br>0.049<br>0.03 |
| Sti 3nd gen; n (K)<br>Metformin; n (K)<br>Thiazolidinedioner; n (K) | 304 (1.0)<br>10330 (34.7)<br>15612 (52.5)<br>1988 (6.7) | 109 (1.0)<br>3617 (32.7)<br>6661 (60.3)<br>916 (8.3) | 0.004<br>0.042<br>0.158<br>0.061 | 92 (1.0)<br>3278 (33.9)<br>5751 (59.5)<br>788 (8.3) | 3223 (33.3)<br>5725 (59.2)<br>781 (8.1) | 0.005 | 17440.8 (61.0)<br>2470.5 (8.6) | 6660.0(60.3)<br>916.0 (8.3) | 0.013 | 113(1.2)<br>2737(30.1)<br>5010(55.1)<br>448(4.9) | 19 (0.8)<br>721 (28.7)<br>1634 (65.1)<br>178 (7.1) | 0.03<br>0.206<br>0.091 |
| SGLT-21; n (N) Alpha-glucoidase inhibitors; n (N) ACE + ARRic n (N) | 2930 (13.2)<br>118 (0.4)<br>20701 (69.6) | 2992 (27.1)<br>55 (0.5)<br>7880 (71.3) | 0.351<br>0.015<br>0.037 | 2367 (24.5)<br>54 (0.6)<br>6877 (71.1) | 2331 (24.1)<br>47 (0.5)<br>6904 (71.4) | 0.009<br>0.01<br>0.006 | 8110.4 (28.4)<br>164.8 (0.6)<br>20429.1 (71.5) | 2992.0 (27.1)<br>55.0 (0.5)<br>7879.0 (71.3) | 0.029<br>0.011<br>0.004 | 1400 (15.4)<br>28 (0.3)<br>6163 (67.7) | 843 (33.6)<br>10 (3.4)<br>1787 (71.2) | 0.422<br>0.015<br>0.075 |
| Thisdes; n (K) Betablocker; n (K) Calcium channel blocker; n (K) | 8040 (27.0)<br>16513 (55.5) | 3245 (29.4)<br>6049 (54.7) | 0.052 | 2828(29.2)<br>5274(54.5)<br>3532(36.5) | 2823 (29.2)<br>5295 (54.8) | 0.001 | 8400.2 (29.4)<br>15752.5 (55.1)<br>10217.4 (35.7) | 1245.0(29.4)<br>6048.0(54.7) | 0.001 | 2419 (26.6)<br>5207 (57.2) | 729 (29.0)<br>1426 (56.8) | 0.055<br>0.009<br>0.068 |
| Loop disretic; n (%) Other disretic; n (%) Nicotor: n (%) | 10964 (36.9)<br>6825 (22.9)<br>2312 (7.8)<br>2855 (9.6)<br>1079 (3.6) | 2912 (25.4)<br>2387 (21.6)<br>1041 (9.4)<br>1071 (9.7) | 0.016<br>0.03<br>0.032<br>0.059 | 2062 (21.3)<br>855 (8.8)<br>917 (9.5)<br>241 (3.5) | 2077 (21.5)<br>878 (9.1) | 0.018<br>0.004<br>0.008 | 6258.2 (21.9)<br>2715.1 (9.5)<br>2797.0 (9.8)<br>1024.7 (2.6) | 2912.0(25.4)<br>2386.0(21.6)<br>1043.0(9.4) | 0.007<br>0.007<br>0.002<br>0.002 | 3210 (35.3)<br>1928 (21.2)<br>852 (9.4) | 805 (32.1)<br>472 (18.8)<br>229 (9.1)<br>278 (11.1)<br>112 (4.5) | 0.00 |
| HF drugs [Digoxin + Entresto + Ivabadrine]; n (X) Anti-acrhythmics; n (X) | \$24 (2.8) | 292 (2.5)<br>230 (2.1) | 0.004<br>0.045 | 917 (8.5)<br>341 (3.5)<br>213 (2.2)<br>2492 (25.8) | 218 (2.5)<br>217 (2.2) | 0.002<br>0.003<br>0.001 | | 192.0 (2.5)<br>230.0 (2.1) | 0.003<br>0.002<br>0.001<br>0.006 | 972 (10.7)<br>164 (4.0)<br>277 (3.0) | 61 (2.4) | 0.022<br>0.038<br>0.004 |
| CONSTITUTION (1 PM) Stating (1 PM) Other lipid-lowering drugs; (1 PM) | 7298(24.9)<br>22642(29.5)<br>3262(11.0) | 2882 (26.1)<br>9133 (82.7)<br>1467 (13.3) | 0.045<br>0.028<br>0.081<br>0.071<br>0.012 | 7976(82.5)<br>1261(13.0) | 2494 (25.8)<br>7970 (82.4)<br>1245 (12.9) | 0.002<br>0.005<br>0.007 | | 2882.0(26.1)<br>9132.0(82.7)<br>1467.0(13.3) | 0.015 | 2012 [22.1]<br>7025 [77.2]<br>1181 [13.0] | 559 (22.3)<br>2042 (81.3)<br>389 (15.5) | 0.102 |
| Antiputer agent, n (N) Oral anticoagulants; n (N) NSAIDs; n (N) | 5022(16.9)<br>4255(14.3)<br>5128(17.2) | 1918(17.4)<br>1342(12.1)<br>2183(19.8) | 0.064 | 1617(16.7)<br>1212(12.5)<br>1879(19.4) | 1644 (17.0)<br>1214 (12.6)<br>1873 (19.4) | 0.001 | 6851.8 (17.0)<br>3516.1 (12.4)<br>5867.8 (20.5)<br>3957.0 (12.8)<br>585.0 (2.4)<br>6298.1 (22.0) | 1917.0(17.3)<br>1342.0(12.1)<br>2183.0(19.8) | 0.01<br>0.007<br>0.019 | 2045 (22.5)<br>1300 (14.3)<br>1547 (17.2) | 610 (24.3)<br>305 (12.1)<br>434 (17.3) | 0.072<br>0.043<br>0.063<br>0.002 |
| Oral conticosteroids; n (%)<br>Bisphosphonates; n (%)<br>Opioids; n (%) | 5128(17.2)<br>3853(13.0)<br>949(3.2)<br>6295(21.2) | 2182(19.8)<br>1517(12.7)<br>254(2.3)<br>2350(21.3) | 0.023<br>0.055<br>0.002 | 1879 (19.4)<br>1308 (13.5)<br>235 (2.4)<br>2078 (21.5) | 1290 (13.3)<br>244 (2.5)<br>2055 (21.3) | 0.005<br>0.006<br>0.006 | 2957.0 (13.8)<br>685.0 (2.4)<br>6298.1 (22.0) | 2183.0(19.8)<br>1517.0(13.7)<br>254.0(2.3)<br>2350.0(21.3) | 0.003<br>0.006<br>0.019 | 1292 (14.2)<br>128 (1.5)<br>1691 (18.6) | 434(17.3)<br>337(13.4)<br>23 (0.9)<br>405(16.1) | 0.023<br>0.055<br>0.065 |
| Anti-depresants; n (N) Gabapentinoids; n (N) Senzodiazepines; n (N) | 8736 (29.4)<br>6400 (21.5)<br>2828 (9.5) | 2297 (20.7)<br>2471 (22.4)<br>1009 (9.1) | 0.02<br>0.02<br>0.013 | 2959 (30.6)<br>2156 (22.3)<br>912 (9.4) | 2956 (30.6)<br>2143 (2.2)<br>882 (9.1) | 0.001<br>0.003<br>0.011 | 6698.2 (23.4)<br>2652.3 (9.3) | 2471.0(22.4)<br>1009.0(9.1) | 0.025<br>0.026<br>0.005 | 2225 (24.5)<br>1405 (15.4)<br>759 (8.3) | 623 (24.8)<br>382 (15.2)<br>198 (7.9) | 0.008<br>0.006<br>0.017 |
| Anxiolyticyhypeotics; n (%)<br>Dementia medi; n (%)<br>Comorbidity score | 2035 (6.8)<br>1520 (5.1) | 900 (8.1)<br>237 (2.1) | 0.049 | 770 (8.0)<br>245 (2.5) | 758 (7.8)<br>229 (2.4) | 0.005 | 2450.8 (8.6)<br>631.6 (2.2) | 900.0 (8.1)<br>237.0 (2.1) | 0.016 | \$47 (6.0)<br>258 (2.8) | 165 (6.6)<br>17 (0.7) | 0.022 |
| mean (ud)<br>Frailty score<br>mean (ud) | 2.81 (2.47)<br>0.18 (0.05) | 2.15 (2.15)<br>0.17 (0.05) | 0.283 | 2.22 (2.18)<br>0.17 (0.05) | 2.20 (2.17)<br>0.17 (0.05) | 0.005 | 2.20 (2.16)<br>0.17 (0.05) | 2.15 (2.15)<br>0.17 (0.05) | 0.019 | 2.10 (2.23)<br>0.17 (0.05) | 0.16 (0.04) | 0.272 |
| Unique generic medicines<br>mean (ud)<br>Unique brand medicines | 11.88 (5.21) | 12.12(5.15) | 0.046 | 12.17 (5.30) | 12.05 (5.12) | 0.021 | 12.37 (5.35) | 12.12 (5.15) | 0.047 | 11.06 (4.97) | 11.27 (4.79) | 0.643 |
| mean (sd)<br>Hospitalizations (-90, 0); n (%)<br>Hospitalizations (-180, 0); n (%) | 12:00 (5:33)<br>2692 (9:3)<br>3940 (13:2) | 12.24 (5.25)<br>418 (2.8)<br>861 (7.8) | 0.045<br>0.216<br>0.179 | 12.28 (5.40)<br>617 (4.3)<br>812 (8.4)<br>2209 (22.8) | 12.17 (5.22)<br>401 (4.1)<br>771 (8.0) | 0.022<br>0.008<br>0.016<br>0.013 | 12.49 (5.46)<br>1098.0 (3.8)<br>2302.2 (8.1) | 12.24 (5.25)<br>418.0 (3.8)<br>861.0 (7.8) | 0.047<br>0.003<br>0.01<br>0.03 | 11.18 (5.09)<br>864 (9.5)<br>1354 (54.9)<br>2831 (31.1) | 11.39 (4.87)<br>103 (4.1)<br>216 (8.6) | 0.041<br>0.215<br>0.196 |
| ED visits; n (%) Officer lists tream (sd) | 2940 (13.2)<br>8768 (29.5)<br>5.30 (4.06) | 2339 (21.2)<br>5.68 (3.99) | 0.192 | 2209 (22.8)<br>5.65 (4.42) | 771 (8.0)<br>2158 (22.3)<br>5 61 (2.8) | 0.013 | 2302.2 (8.1)<br>6407.3 (22.4)<br>5.83/5.33 | 2239.0(21.2)<br>5.68(2.99) | | 2831 (21.1)<br>5.30 (4.03) | 216 (8.6)<br>569 (22.7)<br>5 64 (5.57) | 0.191 |
| man (Lo) Cardiologist visit; n (%) Cardiologist visit; n (%) Internal medicine/family medicine visit;; n (%) | 5.30 (4.06)<br>2859 (9.6)<br>12466 (45.3)<br>27222 (91.5) | 5.68 (3.99)<br>1307 (11.8)<br>6918 (44.5)<br>10036 (90.8) | 0.095<br>0.072<br>0.015<br>0.025 | 5.65 (4.42)<br>1098 (11.4)<br>4212 (43.6)<br>8745 (90.4) | 5.61 (3.88)<br>1079 (11.2)<br>4223 (43.7)<br>8776 (60.8) | 0.005<br>0.002<br>0.011 | 5 83 (5.33)<br>2315.3 (11.6)<br>12670.7 (44.3)<br>25992.8 (80.9) | 5.68 (3.99)<br>1307.0(11.8)<br>4917.0(44.5)<br>10036.0 (90.8) | 0.002<br>0.007<br>0.003<br>0.004 | 977 (10.7)<br>4567 (50.2)<br>7903 (86.8) | 5.64 (5.57)<br>346 (13.8)<br>1242 (49.5)<br>2100 (83.6) | 0.093 |
| Electrocardiograms mean (sd) | 27222 (91.5)<br>0.78 (1.68) | 10036 (90.8)<br>0.68 (1.18) | 0.025 | 8745 (90.4)<br>0.67 (1.19) | 8776 (90.8)<br>0.68 (1.19) | 0.005 | 25992.8 (90.9)<br>0.69 (1.27) | 10036.0 (90.8)<br>0.68 (1.18) | 0.004 | 7903 (86.8)<br>1.48 (3.49) | 2100 (83.6)<br>1.10 (4.29) | 0.091 |
| schocardo<br>men (sd)<br>HbAIc tests received | 0.24 (0.53) | 0.22 (0.50) | 0.045 | 0.21 (0.51) | 0.22 (0.49) | 0.001 | 0.22 (0.51) | 0.22 (0.50) | 0.006 | 0.67 (2.57) | 0.47 (1.77) | 0.091 |
| mean (ud) Glucose tests ordered mean (ud) | 1.38(0.83)<br>0.51(2.66) | 1.48 (0.87)<br>0.41 (1.26) | 0.12 | 1.47 (0.84)<br>0.41 (1.11) | 1.46 (0.81)<br>0.41 (1.27) | 0.012 | 1.49 (0.84)<br>0.43 (1.22) | 1.48 (0.87)<br>0.41 (1.26) | 0.018 | 1.32 (1.18)<br>0.46 (1.58) | 1.39 (1.10)<br>0.40 (1.13) | 0.147 |
| Lipid tests ordered<br>mean (ud)<br>Creatinine tests ordered | 0.95 (0.80) | 1.02 (0.81) | 0.095 | 1.01 (0.78) | 1.01 (0.80) | 0.001 | 1.02 (0.80) | 1.02 (0.81) | 0.001 | 0.88 (0.99) | 1.03 (0.92) | 0.151 |
| mean (sd) Sone mineral density test; n (%) Sasic or comprehensive metabolic blood chem test: n (%) | 0.03 (0.21)<br>1256 (4.2)<br>25915 (87.1) | 0.03 (0.21)<br>502 (4.5)<br>9748 (88.2) | 0.016<br>0.016<br>0.023 | 0.03 (0.20)<br>640 (4.6)<br>8500 (87.9) | 0.03 (0.21)<br>446 (4.6)<br>8523 (88.1) | 0.012<br>0.003<br>0.007 | 0.03 (0.20)<br>1335.0 (4.7)<br>25312.1 (88.6)<br>4123.4 (14.4) | 0.03 (0.21)<br>502.0 (4.5)<br>9747.0 (88.2) | 0.006<br>0.006<br>0.011 | 0.04 (0.32)<br>188 (2.1)<br>7097 (78.0) | 0.03 (0.20)<br>65 (2.6)<br>2084 (83.0) | 0.06<br>0.035<br>0.137 |
| Mammogram; n (%) Pap smear; n (%) PSS-m (%) | 2329(11.2)<br>2777(9.3) | 1586(14.4)<br>1361(12.3) | 0.095 | 840 (4.6)<br>8500 (87.9)<br>1342 (12.9)<br>1142 (11.8)<br>1606 (16.6) | 1356 (14.0)<br>1157 (12.0) | 0.004 | 4123.4 (14.4)<br>3511.3 (12.3)<br>4878.8 (17.1) | 1586.0(14.4)<br>1361.0(12.3) | 0.002 | 752 (8.3)<br>705 (7.7) | 264 (10.5)<br>251 (10.0) | 0.077 |
| PSACTEN Flexible Signal discopy or colonoscopy or CT virtual colonoscopy, n (N) City varcina/fleximococcal varcinar n (N) | 4240 (14.3)<br>1309 (4.4)<br>6903 (23.5) | 557 (5.0)<br>5457 (27.3) | 0.079 | 485 (5.0) | 485 (5.0)<br>2180 (2.5) | 0.001 | 1483.0 (5.2) | 1892.0 (17.1)<br>557.0 (5.0)<br>5467.0 (22.3) | 0.001 | 1549 [17.0]<br>409 [4.5]<br>1092 [23.0] | \$15 (20.5)<br>132 (5.3)<br>486 (19.4) | 0.089 |
| Telemedicine; n (%) | 6991(23.5)<br>5046(17.0)<br>7093(23.8) | 2467 (22.3)<br>1830 (16.6)<br>2361 (21.4) | 0.028<br>0.011<br>0.059 | 2186(22.6)<br>1601(16.6)<br>2063(21.3) | 2180 (22.5)<br>1614 (16.7)<br>2058 (21.3) | 0.004 | 6464.5 (22.6)<br>4711.3 (16.5)<br>6201.8 (21.7) | 2467.0(22.3)<br>1830.0(16.6)<br>2360.0(21.4) | 0.007<br>0.002<br>0.008 | 1932 (21.2)<br>1932 (21.2)<br>1926 (21.2) | 486(19.4)<br>601(23.9)<br>860(18.3) | 0.065 |
| Microalbuminuria/proteinuria; n (K) | 747 (4.1)<br>1109 (4.4) | 478 (2-8)<br>(644 (5-8) | 0.065 | 536 (5.5) | 546 (5.6) | 0.004 | 1596.7 (5.6) | 644.0 (5.8) | 0.008 | 160 (4.0) | 118 (4.7) | 0.032 |
| Writing in (In)<br>Asian; n(In) | | | | | | | | | | | 1 | = |
| Mack; 6 (%) | | | | | | | | | | | + | - |

| tagliptin - refer<br>70 | Optum: 1:1 matched cohor<br>ence Semaglutide -expo | ure 2d St | Opts<br>Stagliptin - referen | em: Fine stratification coho<br>sce Semaglutide - exposu | std diff |
|---|---|---|---|---|---|
| 50 (7.50) | 20.47 (7.75) | 2011 | 28,381 | 11,049 | 200 |
| 9(49.4) | 4812 (49.8) | | 14037 (49.1) | \$405 (48.9) | 0.00 |
| (9.8)<br>9(18.1) | 946 (9.8)<br>1759 (18.2) | 0.005 | 2624.4 (9.2)<br>5238.7 (18.3) | 1007.0(9.1)<br>2051.0(18.6) | 0.00 |
| 9(18.1)<br>7(55.0)<br>5(17.1) | 1759 (18.2)<br>5328 (55.1) | | \$238.7 (18.3)<br>15810.1 (55.3) | 2051.0(18.6)<br>6104.0(55.2) | |
| | 1637 (16.9) | 0.024 | 4907.9 (17.2)<br>69.5 (0.2) | 1887.0(17.1) | 0.0 |
| (5)<br>(5)<br>(7)<br>(23)<br>(23)<br>(24)<br>(25)<br>(27)<br>(27)<br>(27)<br>(27)<br>(27)<br>(28)<br>(29)<br>(23)<br>(23)<br>(24)<br>(23)<br>(24)<br>(24)<br>(24)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(25)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(25)<br>(24)<br>(24)<br>(24)<br>(25)<br>(24)<br>(26)<br>(27)<br>(27 | 74 (0.0)<br>140 (1.3) | | 214.6 (0.8)<br>290.1 (1.0) | 74.0 (0.7)<br>130.0 (1.2) | |
| (2.3) | 231 (2.4)<br>361 (2.7) | | \$46.2 (1.9)<br>\$49.8 (3.3) | 231.0 (2.1)<br>271.0 (3.4) | |
| 9(21.7)<br>1(27.2) | 2100 (21.7)<br>2594 (26.8) | | 5625.8 (19.7)<br>7582.1 (26.5) | 2204.0 (19.9)<br>2922.0 (26.4) | |
| (6.6)<br>(2.5) | 1547 (16.7)<br>631 (6.5) | 0.009 | 11158.5 (39.7)<br>1944.4 (6.8)<br>663.672.31 | 4356.0 (39.4)<br>760.0 (6.9) | 0.00 |
| (1.3) | 231 (2:4)<br>122 (1:3)<br>221 (2:3) | 0.000 | 663.6 (2.3)<br>365.7 (1.3)<br>620.9 (2.2) | 760.0 (6.9)<br>264.0 (2.4)<br>142.0 (1.3)<br>228.0 (2.1) | 0.00 |
| (9.1)<br>2(18.5) | 916 (9.5)<br>1824 (18.9) | 0.013 | 2649.9 (9.3)<br>5687.1 (19.9) | 1011.0(9.2)<br>2168.0(19.6) | 0.00 |
| (1 (17.8)<br>(5 (16.3) | 1775 (18.4)<br>1600 (16.5) | 0.015 | 5881.0 (20.6)<br>5139.4 (18.0) | 2337.0(21.2)<br>2012.0(18.2) | 0.00 |
| (0(19.8)<br>(8.9) | 1878 (19.4)<br>843 (8.7) | 0.008 | \$707.3 (20.0)<br>2551 0 (8.9) | 2143.0(19.4)<br>963.0(8.7) | 0.05<br>0.00<br>0.02 |
| 19(28.4) | 2671 (27.6)<br>2671 (27.6)<br>2118 (21.9) | 0.018 | 8187.7 (28.6)<br>8187.7 (28.6)<br>6277.8 (22.0) | 3034.0(27.5)<br>3034.0(27.5)<br>2429.0(22.0) | 0.02 |
| (4.2) | 409 (4.2)<br>1679 (17.4) | 0.003 | 1175.9 (4.1)<br>4983.9 (17.4) | 645.0 (4.0)<br>1903.0 (17.2) | 0.00 |
| (2.2) | 207 (2.1)<br>561 (5.8) | 200.0 | 664.0(2.2)<br>1764.1 (6.1) | 245.0 (2.2)<br>660.0 (6.0) | 0.00 |
| (2.3) | 307 (3.2)<br>2088 (21.6) | 0.003 | 932.4 (3.3) | 380.0 (3.4)<br>2389.0 (21.6) | 0.00 |
| 8 (45.1)<br>5 (89.7) | 4344 (44.9)<br>8711 (90.1)<br>8019 (82.9) | 0.003 | \$163.2 (21.6)<br>12178.3 (46.1)<br>25700.9 (89.9)<br>23793.5 (83.2)<br>3622.6 (12.7) | \$038.0(45.6)<br>\$911.0(89.7)<br>\$162.0(82.9) | 0.00 |
| (5 (82.7)<br>(5 (13.0) | 1257 (13.0) | 0.007 | 22793.5 (83.2)<br>3622.6 (12.7) | 1375.0(12.4) | 0.00 |
| (2.2)<br>(6.0)<br>(6.0)<br>(7.3)<br>(4(21.7)<br>(4(21.7)<br>(4(21.7)<br>(4(21.7)<br>(5(92.7)<br>(5(92.7)<br>(5(13.0)<br>(7.5)<br>(7.5)<br>(9.5)<br>(9 | 234 (2.4)<br>616 (6.4) | 0.003 | 1860.2 (6.5) | 281.0 (2.5)<br>705.0 (6.4) | 0.00 |
| 19 (41.8)<br>15 (12.3) | 4080 (42.2)<br>1188 (12.3) | 0.009 | 12221.4 (42.8)<br>3605.5 (12.6) | 4754.0(43.0)<br>1378.0(12.5) | 0.00 |
| (1.5) | 149 (1.5)<br>9 (0.1)<br>1263 (13.1) | 0.003 | 469.6 (1.6)<br>26.2 (0.1) | 180.0 (1.6)<br>9.0 (0.1) | 0.00<br>0.01<br>0.01 |
| (1)<br>(4 (13.1)<br>(6 (15.8)<br>(6 (15.7) | 1586 (16.4)<br>1455 (15.7) | 0.009 | 3728.6 (13.0)<br>4585.2 (16.0)<br>10065.7 (35.2) | 1749.0(15.8)<br>1827.0(14.6) | |
| (7.4) | 1814 (18.8)<br>715 (7.4) | 0.004 | \$441.9 (19.0)<br>2186.6 (7.7) | 2066.0(18.7)<br>828.0(7.5) | 0.00<br>0.00 |
| (2.7)<br>(5 (18.3) | 272 (2.8)<br>1749 (18.1) | 0.006 | 813.4 (2.8)<br>5353.3 (18.7) | 297.0 (2.7)<br>1948.0(17.6) | 0.02<br>0.02 |
| (7.4)<br>(0(19.3) | 690 (7.1)<br>1898 (19.6)<br>333 (3.4) | 0.008 | 2136.5 (7.5)<br>6120.2 (21.4)<br>999.1 (3.5)<br>1525.7 (5.3)<br>1492.5 (5.2) | \$19.0 (7.4)<br>2354.0(21.3)<br>261.0 (2.3) | 0.00 |
| (5.6) | 333 (3.4)<br>519 (5.4)<br>508 (5.3) | 0.014 | 999.1 (3.5)<br>1525.7 (5.3) | 361.0 (3.3)<br>583.0 (5.3)<br>557.0 (5.0) | 0.00<br>0.01<br>0.00<br>0.00 |
| (5.4) | \$08 (5.3)<br>1 (0.0)<br>1971 (20.4) | 0.007 | 1.9 (0.0)<br>5712.1 (20.0) | \$57.0 (5.0)<br>1.0 (0.0)<br>2172.0 (19.7) | 0.00 |
| (2-3)<br>(2-7)<br>(2-8)<br>(2-8)<br>(2-1)<br>(2-7)<br>(3-7)<br>(5-6)<br>(5-7)<br>(5 | 6249 (64.6)<br>1120 (11.6) | 0.004 | 18685.4 (65.4)<br>18685.3 (11.7) | 7120.0(64.4)<br>1294.0(11.7) | |
| (5 (18.3)<br>(7 (22.0) | 1721 (17.8)<br>2110 (21.8) | 0.012 | 5104.7 (17.9)<br>6414.6 (22.4) | 1948.0(17.6)<br>2428.0(22.0) | 0.00<br>0.00<br>0.01 |
| (1.4) | 127 (1.4)<br>285 (2.9) | 0.002 | 403.3 (1.4)<br>839.8 (2.9) | 153.0 (1.4)<br>100.0 (2.7) | 0.01<br>0.00<br>0.01 |
| (1.4)<br>(2.8)<br>(4.2)<br>(6(14.6)<br>(5(13.2)<br>(8(24.6) | 188 (4.0)<br>1419 (14.7) | 0.009 | 1161.2 (4.1)<br>4216.2 (14.8) | 429.0 (3.9)<br>1613.0 (14.6) | 0.00 |
| S (13.2)<br>S (24.6) | 1248 (12.9)<br>2393 (24.7) | 0.008 | 3825-3 (13.4)<br>7290-6 (25.5) | 2777.0(25.1) | 0.00 |
| (1.8)<br>(1.0)<br>(5.5) | 387 (4.0)<br>89 (0.9) | 0.011 | 1047.8 (2.7)<br>251.2 (0.9) | 397.0 (3.6)<br>96.0 (0.9) | 0.00 |
| 5 (0.00) | 1 24 (5.3) | 0.011 | 1 26 IN SNI | \$84.0 (5.3)<br>1.34 (0.93) | 0.02 |
| 5 (0.88)<br>19 (17.4)<br>10.0)<br>18 (23.9)<br>21 (59.5)<br>18 (23.9)<br>27 (24.5)<br>10.6)<br>27 (24.5)<br>10.6)<br>27 (21.1)<br>18 (29.2)<br>44 (54.5)<br>12 (26.5)<br>12 (26.5)<br>13 (2.5) | 1.24 (0.91)<br>1633 (16.9)<br>92 (1.0) | 0.013 | 1 26 (0.90)<br>5247.9 (18.4)<br>280.7 (1.0) | 1.24 (0.92)<br>1909.0 (17.3)<br>109.0 (1.0) | 0.02 |
| 18(22.9)<br>11(59.5) | 3223 (33.3)<br>5725 (59.2) | 0.012 | 9690.0 (22.9)<br>17440.8 (61.0) | 1617.0(32.7)<br>6660.0(62.3) | 0.02 |
| (8.3)<br>(7(24.5) | 781 (8.1)<br>2331 (24.1) | 0.009 | 2470.5 (8.6)<br>8110.4 (28.4) | 916.0 (8.3)<br>2992.0 (27.1) | 0.01 |
| (7.6)<br>(7.(71.1) | 47 (0.5)<br>6904 (71.4) | 0.000 | 20429.1 (71.5) | 55.0 (0.5)<br>7879.0 (71.3) | 0.00 |
| 4 (54.5) | 2821 (99.2)<br>5295 (54.8)<br>1450 (35.7)<br>2077 (21.5) | 0.004 | 15753.5 (55.1)<br>16217.4 (15.7) | 6048.0(54.7) | 0.00 |
| (0.8) | 2077 (21.5)<br>878 (9.1) | 0.004 | 10217.4 (35.7)<br>6258.2 (21.9)<br>2715.1 (9.5) | 3912.0(35.4)<br>2386.0(21.6)<br>1043.0(9.4) | 0.00 |
| (2.5) | 878 (9.1)<br>915 (9.5)<br>338 (3.5) | 0.001 | 2715.1 (9.5)<br>2797.0 (9.8)<br>1024.7 (2.6) | 1043.0(9.4)<br>1073.0(9.7)<br>192.0 (8.5) | 0.00 |
| (2.2)<br>(2(25.8) | 217 (2.2)<br>2494 (25.8) | 0.003 | 590.8 (2.1)<br>7659.0 (26.8) | 230.0 (2.1)<br>2882.0 (26.1) | |
| (6 (82.5)<br>(1 (13.0) | 7970 (82.4)<br>1245 (12.9)<br>1644 (17.0)<br>1214 (12.6) | 0.002 | 23786 2 (83.2)<br>3813 4 (13.3)<br>4851 8 (17.0)<br>3536 1 (12.4) | 9132.0(82.7)<br>1467.0(13.3)<br>1917.0(17.3)<br>1342.0(12.1) | 0.01<br>0.01<br>0.00<br>0.00 |
| 17 (16.7)<br>12 (12.5) | 1214 (12.6) | 0.007 | 4851.8 (17.0)<br>3536.1 (12.4)<br>5867.8 (20.5) | 1917.0(17.3)<br>1342.0(12.1) | 0.00 |
| (8(13.5) | 1873 (19.4)<br>1290 (13.3)<br>244 (2.5) | 0.005 | 3957.0 (13.8)<br>685.0 (2.4) | 2183.0(19.8)<br>1517.0(13.7)<br>254.0(2.3) | 0.00 |
| (2.5)<br>(2.2)<br>(2.2)<br>(2.25.8)<br>(4.6)<br>(4.12.0)<br>(7.16.7)<br>(2.12.5)<br>(9.19.4)<br>(8.12.5)<br>(2.4)<br>(9.19.4)<br>( | 2055 (21.3)<br>2956 (30.6) | 0.000 | 6298.1 (22.0)<br>9119.7 (31.9) | 2350.0(21.3)<br>2397.0(30.7) | 0.01 |
| 6 (22.3)<br>1 (9.4) | 2143 (22.2)<br>882 (9.1) | 0.003 | 6698.2 (23.4)<br>2652.3 (9.3) | 2471.0(22.4)<br>1009.0(9.1) | 0.02 |
| (2.5) | 758 (7.8)<br>229 (2.4) | 0.005 | 2450.8 (8.6)<br>631.6 (2.2) | \$00.0 (8.1)<br>237.0 (2.1) | 0.00 |
| 2 (2.18) | 2.20 (2.17) | 0.005 | 2.20 (2.16) | 2.15 (2.15) | 0.01 |
| 7 (0.05) | 0.17 (0.05) | 0.004 | 0.17 (0.05) | 0.17 (0.05) | 0.02 |
| 17 (5.30) | 12.05 (5.12) | 0.021 | 12.37 (5.35) | 12.12 (5.15) | 0.04 |
| 28 (5.40)<br>(4.3)<br>(8.4)<br>(9 (22.8) | 12.17(5.22)<br>401 (4.1)<br>771 (8.0)<br>2158 (92.3) | 0.022 | 12.49 (5.46)<br>1098 D (3.8)<br>2302 2 (8.1)<br>6407 3 (22.4) | 12.24 (5.25)<br>418.0 (3.8)<br>861.0 (7.8) | 0.04<br>0.00 |
| (8.4)<br>19 (22.8) | 271 (8.0)<br>2158 (22.3) | 0.016 | 2302.2 (8.1)<br>6407.3 (22.4) | 861.0 (7.8)<br>2339.0(21.2) | 0.0 |
| 5 (4.42)<br>IB (11.4) | 5.61 (2.88) | 0.01 | 5.83 (5.33) | 5.68 (2.99) | 0.03 |
| HE(11.4)<br>12(43.6)<br>15(90.4) | 1079 (11.2)<br>4223 (43.7)<br>8776 (90.8) | 0.005 | 3315.3 (11.6)<br>12670.7 (44.3) | 1307.0(11.8)<br>4917.0(44.5)<br>10036.0(90.8) | 0.00<br>0.00<br>0.00 |
| 7 (1.19) | 8776 (90.8)<br>0.68 (1.19) | 0.005 | 25992.8 (90.9) | 0.68 (1.18) | 0.00 |
| (0.51) | 0.22 (0.49) | 0.001 | 0.09 (1.27) | 0.22 (0.50) | 0.00 |
| 7 (D.84) | 1.46 (0.81) | 0.012 | 1.49 (0.84) | 1.48 (0.87) | 0.01 |
| (1.11) | 0.41 (1.27) | 0.004 | 0.43 (1.22) | 0.41 (1.26) | 0.01 |
| (0.78) | 1.01(0.00) | 0.001 | 1.02 (0.80) | 1.02 (0.81) | 0.00 |
| (p.20) | 0.03 (0.21)<br>446 (4.6) | 0.012 | 0.03 (0.20)<br>1235.0 (4.7) | 0.03 (0.21)<br>502.0 (4.5) | 0.00 |
| 1 (0.20)<br>(4.6)<br>0 (87.9)<br>3 (13.9)<br>2 (11.8)<br>6 (16.6) | 8523 (88.1) | 0.003 | 25312.1 (88.6) | 9747.0(88.2) | 0.00<br>0.01<br>0.00 |
| 4(13.9)<br>2(11.8) | 1356 (14.0)<br>1157 (12.0)<br>1605 (16.6) | 0.004 | 4123.4 (14.4)<br>3511.3 (12.3) | 1586.0(14.4)<br>1361.0(12.3) | 0.00 |
| (5.0) | 485 (7.0) | 0.001 | 4878.8 (17.1)<br>1483.0 (5.2) | 1892.0(17.1)<br>557.0(5.0) | |
| (5.0)<br>6(22.6)<br>1(16.6)<br>3(21.1) | 2180 (2.5)<br>1614 (16.7)<br>2058 (21.3) | 0.001 | 6464.5 (22.6)<br>4711.3 (16.5)<br>6201.8 (21.7) | 2467.0(22.3)<br>1830.0(16.6)<br>2360.0(21.4) | 0.00 |
| | 227 (2.3) | 0.001 | 476.8 (2.4) | 249.0 (2.3) | 0.00 |
| (5.5) | 546 (5.6) | 0.004 | 1596.7 (5.6) | 644.0 (5.8) | 0.00 |

| Market:<br>Stagliptin - reference | Semaglutide - exposure | Std diff |
|---|---|---|
| ,100 | 2,511 | |
| 8.76 (10.64) | 61.00 (E.64) | 0.547 |
| 1899 (42.5) | 987 (29.2) | 0.351 |
| 2081 (22.9)<br>2932 (22.2) | 386(15.4)<br>565(22.5) | |
| 3543 (28.9)<br>544 (6.0) | 1342 (53.4)<br>218 (8.7) | |
| 1136 (12.5) | 27 (1.1) | 0.703 |
| 859 (9.4)<br>679 (7.5) | 82 (2.2)<br>90 (2.6) | |
| 818 (9.0)<br>835 (9.2) | 128(5.1)<br>185(7.4) | |
| 2673 (29.4)<br>2100 (23.1) | 919 (36.6)<br>1079 (43.0) | |
| 121(1.3)<br>104(1.1) | 23 (0.9)<br>25 (1.0) | 0.039 |
| 232 (2.5)<br>741 (8.1) | 25 (1.0)<br>143 (5.7)<br>285 (11.4) | 0.118 |
| 165 (9.5)<br>1015 (11.2) | 285 (11.4)<br>442 (17.6) | 0.06 |
| 1277 (14.0)<br>146 (10.4) | 478 (19.0)<br>220 (8.8) | 0.115 |
| 621 (6-8)<br>2004 (22-0) | 141 (5.6) | 0.05 |
| 2004 (22.0) | 456 (18.2)<br>456 (18.2) | 0.096 |
| 162 (1.8)<br>1086 (11.9) | 28 (1.5)<br>285 (11.4) | 0.021 |
| 203 (2.2) | 38 (1.5) | 0.053 |
| 612 (6.7)<br>199 (2.2) | 156 (6.2)<br>80 (3.2) | 0.062 |
| 1115 (12.3)<br>1781 (41.5) | 370 (14.7)<br>1164 (46.4) | 0.072 |
| 7957 (87.4)<br>7148 (78.5)<br>1210 (13.3) | 2158 (85.9)<br>2023 (81.0)<br>252 (10.1) | 0.044 |
| 200(2.2) | | 0.037 |
| 195 (4.4)<br>4371 (48.0) | 122 (4.9)<br>1318 (52.5) | 0.024 |
| 612 (6.7)<br>202 (2.2) | 198 (7.9) | 0.045 |
| | 62 (2.5)<br>2 (0.1)<br>287 (1.1.4) | 0.005 |
| 1294 (14.2)<br>1288 (14.2)<br>2285 (26.2) | 2(0.3)<br>287(11.4)<br>269(10.7)<br>548(21.8) | 0.104 |
| 2385 (26.2)<br>1773 (19.5) | 403 (16.0) | 0.00 |
| 715 (7.9)<br>229 (2.5) | 209 (8.3)<br>45 (1.8) | 0.017 |
| 1342 (14.7)<br>455 (5.0) | 286 (11.4) | 0.036 |
| 1621 (17.8)<br>438 (4.8)<br>240 (2.6) | 146 (5.8)<br>581 (23.1)<br>75 (3.0) | 0.132 |
| 240 (2.6) | 67 (2.7)<br>92 (3.7) | 0.002 |
| 2 (0.0)<br>1355 (14.9) | 0 (0.0)<br>284 (11.3) | 0.021 |
| 5169 (56.8) | 1453 (57.9) | 0.021 |
| 908 (10.0)<br>1419 (15.6) | 232 (9.2)<br>330 (13.1) | 0.07 |
| 1490 (16.3)<br>152 (1.7) | 373 (14.9)<br>28 (1.1) | 0.047 |
| 292 (3.2)<br>211 (2.3) | 45 (1.8)<br>44 (1.8) | 0.068 |
| 942 (10.4)<br>880 (9.7) | 242 (9.6)<br>243 (9.7) | 0.024 |
| 1523 (16.7)<br>480 (5.3) | 405 (16.1)<br>33 (1.3) | 0.016 |
| 193 (2.1) | 16 (3.6)<br>160 (6.4) | 0.127 |
| 1.12 (0.86) | 1.28(0.91) | 0.176 |
| 1320 (14.5)<br>113 (1.2) | 645 (17.7)<br>19 (0.8) | 0.068 |
| 1737 (30.1) | 721 (28.7) | 0.03 |
| (010 (55.1)<br>(48 (4.9)<br>(400 (15.4) | 1634 (65.1)<br>178 (7.1)<br>841 (33.6) | 0.091 |
| 28 (0.3) | 10.10.41 | 0.015 |
| 6163 (67.7)<br>2419 (26.6) | 1787 (71.2)<br>729 (29.0) | 0.075 |
| 5207 (57.2)<br>3210 (35.3) | 1426 (56.8)<br>805 (32.1) | 0.009 |
| | 472 (18.8)<br>229 (9.1) | 0.008 |
| 852 (9.4)<br>973 (10.7)<br>166 (4.0) | 278(11.1)<br>112(4.5) | 0.012 |
| 166 (4.0)<br>277 (3.0) | 112 (4.5)<br>61 (2.4)<br>559 (22.3) | 0.038 |
| 2012 (22.1)<br>7025 (77.2) | 2042 (81.3) | 0.102 |
| 1181 (13.0)<br>2045 (22.5) | 389 (15.5)<br>610 (24.3) | 0.072<br>0.043<br>0.063 |
| 1300 (14.3)<br>1567 (17.2) | 305 (12.1)<br>434 (17.3) | 0.002 |
| 1292 (14.2)<br>138 (1.5) | 23 (0.9) | 0.023 |
| 1691 (18.6)<br>2225 (24.5) | 605 (16.1)<br>623 (24.8) | 0.065 |
| 1405 (15.4)<br>759 (8.3) | 382 (15.2)<br>198 (7.9) | 0.006 |
| 547 (6.0) | 165 (6.6)<br>17 (0.7) | 0.023 |
| 258 (2.8)<br>2.10 (2.21) | 1.53 (1.87) | 0.222 |
| | | 0.774 |
| 0.17 (0.05) | 0.16(0.04) | 0.369 |
| 11.06 (4.97) | 11.27 (4.79) | 0.043 |
| 11.18 (5.09)<br>864 (9.5) | 11.39 (4.87)<br>103 (4.1) | 0.041 |
| 1354 (14.9)<br>2831 (21.1) | 216 (8.6)<br>569 (22.7) | 0.196 |
| .30(4.03) | 5.64(5.57) | 0.07 |
| 977 (10.7) | 346 (13.8) | 0.093 |
| 4567 (50.2)<br>7903 (86.8) | 1242 (49.5)<br>2100 (83.6) | 0.091 |
| 1.48 (2.49) | 1.10 (4.29) | 0.096 |
| 0.67 (2.57) | 0.47(1.77) | 0.091 |
| 1.22 (1.18) | 1.39 (1.10) | 0.147 |
| 0.46 (1.58) | 0.40 (1.13) | 0.043 |
| D. 88 (D. 99) | 1.03(0.92) | 0.012 |
| 0.88 (0.99) | 0.03(0.92) | -0.151 |
| 188 (2.1) | 65 (2.6) | 0.06 |
| 1097 (78.0)<br>152 (8.3) | 2084 (83.0)<br>264 (10.5) | 0.127 |
| | 251 (10.0)<br>515 (20.5) | 0.079 |
| 705 (7.7)<br>1549 (17.0) | | |
| 705 (7.7)<br>1549 (17.0)<br>409 (4.5) | 132 (5.3) | 0.02 |
| 1549 [17:0]<br>109 (4:5)<br>1092 [23:0] | 132 (5.3)<br>486 (19.4)<br>601 (23.9) | 0.035 |
| 1549 (17.0)<br>409 (4.5)<br>2092 (23.0)<br>1932 (21.2)<br>1926 (21.2) | 601 (23.9)<br>460 (18.3) | 0.035<br>0.089<br>0.065<br>0.072 |
| 1549 (17.0)<br>109 (4.5)<br>1092 (23.0)<br>1932 (21.2) | 601 (23.9) | 0.035<br>0.069<br>0.065<br>0.072<br>0.032 |
| 549 (17.0)<br>09 (4.5)<br>092 (21.0)<br>932 (21.2)<br>926 (21.2) | 601 (23.9)<br>460 (18.3) | |
| 1549 (17.0)<br>409 (4.5)<br>2092 (23.0)<br>1932 (21.2)<br>1926 (21.2) | 601 (23.9)<br>460 (18.3) | |

| Stagliptin-reference | Semaglutide - exposure | Std diff |
|---|---|---|
| 2,297 | 2,29/ | |
| 63.33 (8.87) | 63.43 (8.54) | 0.011 |
| 912 (39.7) | 907 (19.5) | 0.004 |
| 380(16.5)<br>548(23.9) | 371 (16.2)<br>537 (23.4) | |
| 1185 (51.6) | 1194 (52.0) | |
| 21.02.01 | 27 (1.2) | 0.034 |
| 21 (0.9)<br>87 (2.8) | 12 (2.6) | |
| 88 (3.8)<br>126 (5.5) | 90 (3.9)<br>127 (5.5) | |
| 195 (8.5)<br>854 (37.2) | 182 (7.9)<br>857 (37.3) | |
| 926 (40.3) | 931 (40.5) | |
| 23 (1.0) | 23 (1.0) | 0.000 |
| 22 (1.0)<br>20 (0.9) | 24 (1.0) | 0.000 |
| 137 (6.0) | 137 (6.0) | 0.001 |
| 258 (11.2)<br>361 (15.7) | 253 (11.0)<br>272 (16.2) | 0.007 |
| 413 (18.0) | 625 (18.5)<br>211 (9.2) | 0.014 |
| 217 (9.4)<br>131 (5.8) | 130 (5.7) | 0.000 |
| 432 (18.8)<br>432 (18.8) | 421 (18.3)<br>421 (18.3) | 0.012 |
| 224 (14.1)<br>22 (1.4) | 341 (14.8)<br>35 (1.5) | 0.021 |
| 248 (10.8)<br>47 (2.0) | 255 (11.1)<br>36 (1.6) | 0.03 |
| 145 (6.3)<br>67 (2.9) | 142 (6.2)<br>65 (2.8) | 0.000 |
| 214(12.7) | 327 (14.2) | 0.010 |
| 1976 (86.0) | 1982 (86.3) | 0.000 |
| 1818 (79.1)<br>241 (10.5) | 1847 (80.4)<br>233 (10.1) | 0.031 |
| 89 (2.9)<br>104 (4.5) | 83 (3.6)<br>103 (4.5) | 0.014 |
| 1183 (51.5)<br>123 (7.5) | 1193 (51.9) | 0.009 |
| 61 (2.7) | 59 (2.6) | 0.005 |
| 2 (0.1)<br>252 (11.0) | 59 (2.6)<br>1 (0.0)<br>368 (11.7) | 0.017 |
| 258(11.2)<br>521(22.7) | 246 (10.7)<br>505 (22.0) | 0.017 |
| 282 (16.7) | 377 (16.4) | 0.000 |
| 207 (9.0)<br>43 (1.9) | 192 (8.4)<br>41 (1.8) | 0.000 |
| 274(11.9)<br>138(6.0) | 269 (11.7)<br>125 (5.4) | 0.003 |
| 503 (21.9)<br>72 (3.1) | 523 (22.8)<br>69 (2.0) | 0.021 |
| \$7 (2.5) | \$6 (2.4) | 0.003 |
| 85 (3.7) | 88 (2.8)<br>- | 0.003 |
| 248 (10.8)<br>1318 (57.4) | 260 (11:3)<br>1315 (57.2) | 0.017 |
| 1318 (57.4)<br>213 (9.3)<br>306 (13.3) | 1315 (57.2)<br>213 (9.3)<br>307 (13.4) | 0.000 |
| 306 (13.3)<br>337 (14.7) | 207 (13.4)<br>219 (14.8) | 0.000 |
| 45 (2.0) | 40 (1.1)<br>40 (1.7) | 0.000 |
| 44 (1.9)<br>216 (9.4) | 40 (1.7)<br>223 (9.7) | 0.01 |
| 199 (8.7)<br>368 (16.0) | 222 (9.7)<br>366 (15.9) | 0.01 |
| 26 (1.1) | 366 (15.9)<br>32 (1.4) | 0.002 |
| 15 (0.7)<br>138 (6.0) | 16 (0.7)<br>145 (6.3) | 0.013 |
| 1.26 (0.88) | 1.25 (0.89) 394 (17.2) | 0.009 |
| 16 (0.7) | 394 (17.2)<br>16 (0.7) | 0.001 |
| 677 (29.5) | 652 (28.4) | 0.024 |
| 1492 (ES.O)<br>135 (S.9) | 1472 (64.1)<br>148 (6.4) | 0.018 |
| 582 (29.7)<br>7 (0.3) | 710 (20.5)<br>8 (0.2) | 0.017 |
| 1629 (70.9)<br>656 (28.6) | 1628 (70.9)<br>658 (28.6) | 0.000 |
| 1302 (56.7) | 1105 (54.8) | 0.003 |
| 731 (31.8)<br>450 (19.6) | 744 (32.4)<br>426 (18.5) | 0.012 |
| 199 (8.7) | 206 (9.0) | 0.011 |
| 259 (11.3)<br>99 (4.3)<br>61 (2.7) | 98 (4.3)<br>55 (2.4) | 0.002 |
| 504 (21.9)<br>1891 (82.3) | 502 (21.9)<br>1859 (80.9) | 0.003 |
| 353 (15.4) | 357 (15.5) | 0.001 |
| 578 (25.2)<br>290 (12.6) | 553 (24.1)<br>284 (12.4) | 0.021 |
| 289 (16.9) | 295 (17.2)<br>208 (13.4) | 0.000 |
| 24 (1.0)<br>361 (15.7) | 23 (1.0)<br>275 (16.3) | 0.004 |
| 582 (25.3) | \$70 (24.8) | 0.012 |
| 333 (14.5)<br>186 (8.1) | 351 (15.3)<br>184 (8.0) | 0.022 |
| 141 (6.1) | 152 (6.4)<br>17 (0.7) | 0.00 |
| 1 57 (1 58) | A PER ANN | 0.00 |
| 1.57 (1.88) | 1.55 (1.89) | 0.01 |
| 0.16 (0.04) | 0.16(0.04) | 0.011 |
| 11.20 (4.87) | 11.20 (4.75) | 0.000 |
| 11.31 (4.96) | 11.32 (4.83) | 0.000 |
| 205 (4.6)<br>205 (8.9) | 200 (4.4)<br>206 (9.0) | 0.002 |
| \$41 (23.6) | \$19 (23.5) | 0.003 |
| 5.51 (4.20)<br>291 (12.7)<br>1123 (49.3)<br>1955 (85.1) | 5.59(5.41)<br>300 (13.1) | 0.01 |
| 1123 (49.3) | 300 (12.1)<br>1141 (49.7)<br>1930 (84.0) | 0.003 |
| | | 0.0 |
| 1.09 (2.31) | 1.12 (4.47) | 0.000 |
| 0.48 (1.68) | 0.49(1.83) | 0.001 |
| 1.39 (1.22) | 1.38(1.12) | 0.013 |
| 0.42 (1.21) | 0.41(1.16) | 0.00 |
| 1.03 (0.98) | 1.02 (0.92) | 0.011 |
| 0.02(0.94) | 0.03 (0.21) | 0.011 |
| 0.03 (0.24)<br>60 (2.6)<br>1883 (82.0) | 0.03 (0.21)<br>59 (2.6)<br>1905 (83.0) | 0.011 |
| 1883 (82.0)<br>230 (10.0) | 1905 (83.0)<br>239 (10.4) | 0.020 |
| 217 (9.4) | 228 (9.9) | 0.010 |
| 462 (20.1) | 463 (20.2) | |
| 122 (5.3)<br>446 (19.4) | 120 (5.2)<br>452 (19.7) | 0.004 |
| \$41(23.6) | 561 (24.4)<br>430 (18.7) | 0.018 |
| | 22 (2.1) | |
| 427 (18.6)<br>73 (3.2) | | |
| 427 (18.6)<br>73 (3.2)<br>103 (4.5) | 107 (4.7) | 0.002 |
| 427 (18.6)<br>73 (3.2)<br>103 (4.5) | 107 (4.7) | 0.008 |
| 427 (18.6)<br>72 (3.2)<br>103 (4.5) | 107 (4.7) | 0.008 |

| 1000 | Stagliptin-referen<br>8,861 | scan: Fine stratification cohori<br>ice Semaglutide - exposure<br>2,510 | Stddiff |
|---|---|---|---|
| MATTER M | 3.02 (8.76) | 63.01 (8.44) | 0.002 |
| ALTERNATION ACCOUNTY ACCOUN | 1477.5 (29.2) | 986.0 (39.3) | 0.001 |
| ALTERNATION ACCOUNTY ACCOUN | 1395.0 (15.8)<br>1008.9 (22.7) | 386.0 (15.4)<br>565.0 (22.5) | |
| A. C. A. C | 4676.9 (52.8)<br>779.2 (8.8) | 1341.0 (53.4)<br>218.0 (8.7) | |
| A. C. A. C | 86.9 (1.0)<br>275 8 (2.1) | 27.0 (1.1) | 0.022 |
| A. C. A. C | 294.2 (2.3)<br>431.1 (4.9) | 90.0 (0.6) | |
| A. C. A. C | 664.0 (7.5)<br>2358.8 (27.9) | 185.0 (7.4)<br>919.0 (36.6) | |
| MARCHAN MARCH MARCHAN MARCHA | 3750.4 (42.3) | 1078.0 [42.9] | |
| MARCHAN MARC | 81.6 (0.9) | 23.0 (0.9) | 0.001 |
| 18 1 | 88.8 (1.0)<br>90.2 (1.0) | | 0.001 |
| MATTER M | \$10.4 (\$.8)<br>\$89.5 (11.2) | 143.0 (5.7)<br>285.0 (11.4) | 0.003 |
| MARCHAN MARC | 1467.7 (16.6) | | 0.027 |
| MARCHAN MARC | 785.7 (8.9)<br>516.3 (5.8) | 220.0 (8.8)<br>141.0 (5.6) | 0.004 |
| ## 20 June 19 | | 456.0 (18.2)<br>456.0 (18.2) | 0.004 |
| Teacher Teac | 1321.0 (14.9)<br>128.5 (1.5) | 285.0 (15.3)<br>28.0 (1.5) | 0.012 |
| MARCHAN MARCH MA | | 285.0 (11.4)<br>28.0 (1.5) | 0.017 |
| THE COLUMN THE | 544.0 (6.1) | 156.0 (6.2)<br>80.0 (8.2) | 0.003 |
| MARCHAN MARC | | 370.0 (14.7)<br>1163.0 (46.3) | 0.007 |
| MARCHAN MARC | 7606-2 (85.8)<br>7164-6 (80.9) | 2157.0 (85.9)<br>2032.0 (81.0) | 0.003 |
| MARCHAN MARC | 861.0 (9.7)<br>334.7 (3.8) | 253.0 (10.1)<br>99.0 (3.9) | 0.012 |
| 1922 A. 1922 A | 415.3 (4.7) | 122.0 (4.9) | 0.008 |
| 1.486 | 718.7 (8.1) | 198.0 (7.9) | 0.008 |
| MARCHAN MARC | 4.1 (0.0) | 2.0 (0.1) | 0.013 |
| Tell | 929.3 (10.5) | 269.0 (10.7) | 0.007 |
| MARCHAN MARC | 1435.1 (16.2) | | 0.001 |
| MARTIN | | 45 0 (1 B) | 0.006 |
| MARTIN | 90.4 (10.9)<br>518.0 (5.8) | 146.0 (5.8) | 0.001 |
| MARTINE | 2006-3 (22.6)<br>263.5 (2.0) | 74.0 (2.9) | 0.011 |
| MARCHAEL MARCHAEL SAME | 225.4 (2.5)<br>329.8 (3.7) | 67.0 (2.7)<br>92.0 (3.7) | 0.008 |
| 1841 150 | 985.9 (11.1) | 284.0 (11.3) | 0.006 |
| 1982 | 5153.4 (58.2)<br>821.2 (9.3) | 1452.0 (57.8)<br>232.0 (9.2) | 0.006 |
| March Marc | 1149.3 (13.0)<br>1289.0 (14.5) | 272.0 (12.1) | 0.005 |
| MARCHAN MARC | 91.4(1.0) | 28.0 (1.1) | 0.006 |
| 120 | 166.2 (1.9) | 44.0 (1.8) | 0.009 |
| MARINE M | \$37.3 (9.4)<br>1469.7 (16.6) | 243.0 (9.7) | 0.008 |
| MARINE M | 108.2 (1.2)<br>56.6 (1.6) | 33.0 (1.3)<br>16.0 m (1 | 0.006 |
| MARTINE MART | 557.9 (6.3) | 160.0 (6.4) | 0.003 |
| MARINE 1994 1994 1995 | | | 0.006 |
| Telephone | 64.1 (0.7) | | 0.004 |
| PART | 5764.5 (65.1) | 1634.0 (65.1) | 0.001 |
| MARCHAN MARC | 2973.5 (23.6) | 842.0 (32.5) | 0.001 |
| MARCHAN MARC | 47.1 (0.4)<br>6285.4 (70.9) | 1786.0 (71.2) | 0.005 |
| MARCHAN MARC | 5007.3 (56.5) | 1425.0 (56.8) | 0.005 |
| 1975 1976 | 1619.7 (18.3) | 471.0 (18.8) | 0.013 |
| MARCHAN MARC | 1039.8 (11.7) | 229.0 (9.1)<br>277.0 (11.0) | 0.008 |
| 100 | 290.4 (4.4)<br>206.8 (2.3) | 61.0 (4.5) | 0.004 |
| MARCHAN MARC | 1919.9 (21.7)<br>7237.9 (81.7) | 559.0 (22.3)<br>2041.0 (81.3) | 0.015 |
| MARCHAN MARC | 2168.9 (24.5) | 289.0 (15.5)<br>609.0 (24.3) | 0.013 |
| 100 | 1493.7 (16.9) | 305.0 (12.2)<br>634.0 (17.3) | 0.005 |
| 100 | | | 0.003 |
| 1.0 m. 1 | | 605.0 (16.1)<br>623.0 (24.8) | 0.001 |
| 1.0 m. 1 | 1312.7 (14.8)<br>702.3 (7.9) | 382.0 (15.2)<br>198.0 (7.9) | 0.011 |
| 1201.07 | S6.5 (6.3)<br>S1.3 (0.7) | 165.0 (6.6) | 0.012 |
| 1.50 | | | 0.004 |
| 1.00 | 160.04 | 0.16 (0.04) | 0.00 |
| 1.10 | and the second | 2.40 pc.00) | 0.006 |
| ### AMARIA MARA MAR | | 11.75(6.79) | 0.008 |
| Med. | 157.6 (4.0) | 11.28 (4.87) | 0.003 |
| AMAN AND AMA | 776.0 (8.8)<br>2046.1 (23.1) | 216.0 (8.6)<br>568.0 (22.6) | 0.005 |
| 140 140 140 150 | 5.62 (4.41) | | 0.004 |
| 123.51.56) (55.07.51) (60.00) 120.7(83.4) (70.01) (70.01) (70.01) (70.01) 120.7(83.4) (70.01) | 1242.7 (14.0)<br>1389.8 (49.5) | 345.0 (13.7)<br>1241.0 (49.4) | 0.000 |
| 2235.054) 65.0040 0.000 2203.0540 0.000 2203.0540 0.000 2203.0540 0.000 2204.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.0000 224.0540 0.00000 224.0540 0.00000 224.0540 0.00000 224.0540 0.000000 224.0540 0.0000000000000000000000000000000 | 7443.2 (84.0) | 2099.0 (83.6) | 0.01 |
| 2235.054) 65.0040 0.000 2203.0540 0.000 2203.0540 0.000 2203.0540 0.000 2204.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.0000 224.0540 0.00000 224.0540 0.00000 224.0540 0.00000 224.0540 0.000000 224.0540 0.0000000000000000000000000000000 | 1.07 (2.20) | 1.10 (4.30) | 0.009 |
| 2235.054) 65.0040 0.000 2203.0540 0.000 2203.0540 0.000 2203.0540 0.000 2204.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.000 224.0540 0.0000 224.0540 0.00000 224.0540 0.00000 224.0540 0.00000 224.0540 0.000000 224.0540 0.0000000000000000000000000000000 | 0.48(1.64) | 0.47 (1.77) | 0.002 |
| 2235.054) 65.0045 0.000 2203.078.10 0.001 2203.078.10 0.001 2203.078.10 0.001 2213.078.10 0.001 2214.078.10 0.001 2214.078.10 0.000 2215.078.10 0.000 2215.078.10 0.000 2215.078.10 0.000 2215.078.10 0.000 | 1.40(1.11) | 1.39 (1.10) | 0.006 |
| 732.5 (2.6.) 65.0 (2.6.) 6.000 730.7 (3.4.) (3.01.) (3 | 0.42(1.21) | 0.40 (1.13) | 0.015 |
| 732.5 (2.6.) 65.0 (2.6.) 6.000 730.7 (3.4.) (3.01.) (3 | 1.03 (0.99) | 1.03 (0.92) | 0.001 |
| 984.4 (10.6) 246.0 (10.5) 0.000 0.01 (10.5) 1.000 0.000 0.01 (10.5) 1.51.0 (10.5) 0.000 0.100 0.01 (10.5) 1.51.0 (10.5) 1.000 0.000 0.0000 | 0.03 (0.26) | 0.03 (0.30) | 0.002 |
| 901.8 (10.2) 253.0 (10.0) 0.000 1799.2 (20.1) 535.0 (20.5) 0.000 1799.2 (20.1) 535.0 (20.5) 0.000 1702.7 (20.2) 486.0 (10.4) 0.000 1702.7 (20.2) 486.0 (10.4) 0.000 1702.7 (20.2) 0.000 1509.2 (17.9) 400.0 (10.3) 0.000 1509.2 (17.9) 400.0 (10.3) 0.000 1509.2 (17.9) 400.0 (10.3) 0.000 | | | 0.002 |
| 470,7(5.3) 122.0(5.3) 0.000<br>1702,7(9.2) 486.0(19.4) 0.000<br>1713,6(9.1) 601.0(23.9) 0.000<br>1590,3(9.7.9) 460.0(18.3) 0.01<br>1590,3(9.7.9) 76.0(18.3) 0.01 | 232.5 (2.4)<br>7290.7 (83.4) | | 0.004 |
| 1702.7 (19.2) 486.0 (19.4) 0.004<br>1133.6 (24.1) 691.0 (23.9) 0.001<br>1590.3 (17.9) 460.0 (18.3) 0.01<br>155.2 (2.3) 76.0 (3.0) 0.005 | 901.8 (10.2) | 251.0 (10.0) | 0.006 |
| 1590.3 (17.9) 460.0 (18.3) 0.01<br>255.2 (2.9) 76.0 (3.0) 0.005 | 901.8 (10.2)<br>1799.2 (20.3) | 251.0 (10.0)<br>515.0 (20.5) | 0.005 |
| 255.2 (2.9) 76.0 (3.0) 0.000 | 901.8 (10.2)<br>1799.2 (10.3)<br>470.7 (5.3) | 251.0 (10.0)<br>515.0 (20.5) | 0.002 |
| 3,000 | 901.8 (10.2)<br>1799.2 (20.3)<br>470.7 (5.3)<br>1702.7 (19.2)<br>2133.6 (24.1)<br>1590.3 (17.9) | 251.0 (10.0)<br>515.0 (20.5)<br>132.0 (5.3)<br>486.0 (19.4)<br>601.0 (21.9)<br>460.0 (18.3) | 0.002<br>0.004<br>0.003 |
| | 901.8 (10.2)<br>1799.2 (20.3)<br>470.7 (5.3)<br>1702.7 (19.2)<br>2133.6 (24.1)<br>1590.3 (17.9)<br>255.2 (2.9) | 251.0 (10.0)<br>515.0 (20.5)<br>132.0 (5.3)<br>486.0 (19.4)<br>601.0 (21.9)<br>460.0 (18.3) | 0.002<br>0.004<br>0.003 |
| | 901.8 (10.2)<br>1799.2 (20.3)<br>470.7 (5.3)<br>1702.7 (19.2)<br>2133.6 (24.1)<br>1590.3 (17.9)<br>255.2 (2.9) | 251.0 (10.0)<br>515.0 (20.5)<br>132.0 (5.3)<br>486.0 (19.4)<br>601.0 (21.9)<br>460.0 (18.3) | 0.002<br>0.004<br>0.003 |
| | 901.8 (10.2)<br>1799.2 (20.3)<br>470.7 (5.3)<br>1702.7 (19.2)<br>2133.6 (24.1)<br>1590.3 (17.9)<br>255.2 (2.9) | 251.0 (10.0)<br>515.0 (20.5)<br>132.0 (5.3)<br>486.0 (19.4)<br>601.0 (21.9)<br>460.0 (18.3) | 0.002<br>0.004<br>0.003 |
| | 01.8 (10.2)<br>799.2 (20.3)<br>70.7 (5.3)<br>702.7 (19.2)<br>133.6 (24.1)<br>500.3 (17.9)<br>55.2 (2.9) | 251.0 (10.0)<br>515.0 (20.5)<br>132.0 (5.3)<br>486.0 (19.4)<br>601.0 (21.9)<br>460.0 (18.3) | 0.002<br>0.004<br>0.003 |

| Stagliptin - referen<br>25,643 | edicare: Unadjusted cohort<br>sce Semaglutide - exposure<br>1,147 | 2461 | Stagliptin - refere | edicare: 1:1 matched cohort<br>nce Semaglutide - exposure<br>1,006 | Stddff | Situgliptin - refere<br>24,697 | are: Fine stratifical<br>ice Semaglutide<br>1,142 |
|---|---|---|---|---|---|---|---|
| 5.74 (7.10) | 73.10 (5.93) | 0.403 | 73.29(6.28) | 73.26 (5.97) | 0.004 | 73.12 (6.05) | 73.13 (5.94) |
| 3092 (51.1) | 534 (46.6) | 0.09 | \$30 (48.4) | \$19(47.4) | 0.02 | 11504.9 [46.6] | 533.0 [46.7] |
| 070 [19:8]<br>249 [20:5]<br>1028 [43:0] | 195 (17.0)<br>186 (16.2)<br>504 (43.9)<br>262 (22.8) | | 175 (16.0)<br>204 (18.6)<br>481 (43.9) | 187(17.1)<br>179(16.3) | | 4089.1 (16.6)<br>2998.9 (16.2)<br>10889.4 (44.1) | 195.0 (17.1)<br>185.0 (16.2) |
| 11028 (43.0)<br>1296 (16.8) | 504 (43.9)<br>262 (22.8) | | 481 (43.9)<br>236 (21.5) | 484 (44.2)<br>245 (22.4) | | 10889.4 [44.1]<br>5719.6 (23.2) | \$03.0 [44.0]<br>259.0 [22.7] |
| 6096 [23.8] | 12 (1.0) | 1.21 | 4 (0.4) | 12 (1.1) | 0.086 | 209.7 (1.3) | 11.0 (1.0) |
| 5454 (21.3)<br>4489 (37.5) | 66 (5.8)<br>85 (7.4)<br>413 (36.0) | | 68 (6.2)<br>86 (7.8) | 66 (6.0)<br>85 (7.8) | | 1344.3 (5.4)<br>1819.9 (7.4) | 95.0 (5.8)<br>95.0 (7.4) |
| 4632 (18.1) | \$71 (49.8) | | 536 (48.9) | 532 (48.5) | | 12239.3 (49.6) | 567.0 (49.6) |
| 233 (2.9) | 14(1.2) | 0.03 | 9 (0.8) | 13 (1.2) | 0.037 | 100.9 (1.2) | 14.0 (1.2) |
| 169 (0.7)<br>1116 (4.4) | 4 (0.3)<br>17 (1.5) | 0.044 | 2 (0.2)<br>22 (2.0) | 4 (0.4)<br>17 (1.6) | 0.035 | 86.2 (0.3)<br>362.9 (1.5) | 4.0 (0.4)<br>17.0 (1.5) |
| 3023 (11.8)<br>4279 (16.7) | 231 (20.1) | 0.009 | 124 (11.3)<br>212 (19.3) | 106(9.7)<br>212(19.3) | 0.001 | 2453.6(9.9)<br>4865.6(19.7) | 229.0 (20.1) |
| 2610(10.2)<br>2923(15.3)<br>4303(16.8)<br>1668(6.5) | 206 (18.0)<br>258 (22.5)<br>164 (14.3)<br>67 (5.8) | 0.185 | 181 (16.5)<br>221 (20.2)<br>160 (14.6) | 187 (17.1)<br>233 (21.3)<br>158 (14.4) | 0.027 | \$429.7 (22.0)<br>\$429.5 (14.1) | 255.0 (22.3)<br>154.0 (14.4) |
| 1668 (6.5)<br>5191 (20.2) | 67 (5.8)<br>225 (19.6) | 0.028 | \$6 (5.1) | 66 (6.0)<br>210 (19.2) | 0.04<br>0.059<br>0.059 | 1462.4 (5.9)<br>4836.3 (19.6) | 164.0 (14.4)<br>66.0 (5.8)<br>224.0 (19.6) |
| 5191 (20.2)<br>2205 (8.6) | 225 (19.6)<br>225 (19.6)<br>100 (8.7) | 0.016<br>0.016<br>0.004 | 236 (21.5)<br>236 (21.5)<br>93 (8.5) | 210(19.2)<br>94 (8.6) | 0.059 | 4836.3(19.6)<br>4836.3(19.6)<br>2181.9(8.8) | 224.0 (19.6)<br>100.0 (8.8) |
| 375 (1.5)<br>2461 (9.6) | 19(1.7)<br>84(7.3) | 0.016<br>0.082<br>0.007 | 25 (2.3)<br>82 (7.5) | 18 (1.6)<br>81 (7.4) | 0.046<br>0.003<br>0.021 | 405.5 (1.6)<br>1818.8 (7.4) | 19.0 (1.7)<br>84.0 (7.4) |
| 424 (1.7)<br>1504 (5.9)<br>212 (0.8)<br>2391 (9.3) | 20 [1.7]<br>74 [6.5]<br>10 [0.9]<br>95 [8.3] | 0.007 | 20 (1.8)<br>63 (5.7)<br>8 (2.7)<br>95 (8.7) | 17 (1.6)<br>67 (6.1)<br>10 (0.9)<br>92 (8.4) | 0.021 | 407.8 (1.7)<br>1590.4 (6.4)<br>204.3 (0.4)<br>2070.3 (8.4) | 20.0 (1.8)<br>74.0 (6.5)<br>10.0 (0.9)<br>95.0 (8.3) |
| 212 (0.8)<br>2391 (9.3) | 10 (0.9)<br>95 (8.3) | 0.037 | 8 (0.7)<br>95 (8.7) | 10 (0.9)<br>92 (8.4) | 0.01 | 204.3 (0.8)<br>2070.3 (8.4) | 95.0(8.3) |
| 9186 (35.8)<br>19249 (75.1) | 467 (40.7)<br>823 (72.6) | 0.054 | 436 (29.8)<br>806 (73.5) | 425 (29.7)<br>796 (72.6) | 0.002 | 9949.4 (40.3)<br>17964.9 (72.7) | 463.0 (40.5)<br>830.0 (72.7) |
| 14941 (58.3)<br>4333 (16.9) | 645 (56.2)<br>165 (14.4) | 0.041 | 644 (58.8)<br>166 (15.1) | 608 (55.5)<br>158 (14.4) | 0.021<br>0.006 | 13844.1 (56.1)<br>3531.1 (14.3) | 641.0 (56.1)<br>165.0 (14.4) |
| 1855 (7.2)<br>18008 (50.7) | 27 (2.4)<br>70 (6.1)<br>571 (49.8) | 0.015<br>0.045<br>0.045 | 25 (2.3)<br>57 (5.2)<br>525 (48.8) | 67 (6.1)<br>528 (49.1) | 0.04 | 1512.1 (6.1)<br>12208 1 (49.4) | 69.0 (6.0)<br>567.0 (49.6) |
| 4228 (16.5)<br>385 (1.5) | 70 (6.1)<br>571 (49.8)<br>169 (14.7)<br>20 (1.7) | 0.048 | 161 (14.7)<br>12 (1.1) | 164 (15.0)<br>19 (1.7) | 0.008 | 1624.2 (14.7)<br>417.7 (1.7) | 168.0 (14.7)<br>20.0 (1.8) |
| 31 (0.1)<br>4439 (17.3) | 1 (0.1)<br>169 (14.7) | 0.01 | 2 (0.2)<br>162 (14.8) | 1 (0.1)<br>163 (14.9) | 0.025<br>0.003<br>0.048 | 23.5 (0.1)<br>3580.9 (14.5) | 1.0 (0.1) |
| 4822 (18.8)<br>8817 (34.4) | 187 (16.3)<br>276 (22.8) | 0.066 | 199 (18.2)<br>375 (34.2) | 179(16.3)<br>261(32.9) | 0.04E<br>0.027 | 4040.4 (16.4)<br>8135.2 (32.9) | 186.0 (16.3)<br>273.0 (32.7) |
| 4532 (17.7)<br>1624 (6.3)<br>852 (3.3) | 188 (16.4)<br>60 (5.2) | 0.034<br>0.047<br>0.031 | 179 (16.3)<br>51 (4.7)<br>34 (3.1) | 180 (16.4)<br>56 (5.1) | 0.027<br>0.002<br>0.021<br>0.022 | 1982.1 (16.1)<br>1247.4 (5.1) | 186.0 (16.3)<br>60.0 (5.3) |
| 852 (3.3)<br>3891 (15.2)<br>1394 (5.4) | 32 (2.8)<br>162 (14.1)<br>51 (4.4) | 0.031 | 34 (3.1)<br>163 (14.9)<br>52 (4.7) | 20 (2.7)<br>151 (13.8)<br>51 (4.7) | 0.022<br>0.031<br>0.004 | 715.3 (2.9)<br>2472.4 (14.1)<br>1099.1 (4.5) | 32.0 (2.8)<br>162.0 (14.2)<br>51.0 (4.5) |
| 2794 (10.9) | 167 (14.6) | 0.11 | 144 (13.1) | 155(14.1) | 0.029 | 3537.8(14.3) | 165.0 (14.4) |
| 1213 (4.7)<br>614 (2.4)<br>1921 (7.5) | 35 (3.1)<br>32 (2.8)<br>49 (4.3) | 0.025 | 33 (3.0)<br>25 (2.3)<br>58 (5.3) | 35 (3.2)<br>30 (2.7)<br>47 (4.3) | 0.029 | 723.7 (2.9)<br>685.8 (2.8)<br>1044.0 (4.2) | 35.0 (3.1)<br>32.0 (2.8)<br>49.0 (4.3) |
| 1921 (7.5)<br>2 (0.0)<br>1820 (15.2) | 0 (0.0) | 0.012 | 122 (12.1) | 179/11/0 | 0.011 | 2842.2(11.5) | 133.0 (11.6) |
| 13114 (51.1) | 625 (54.5)<br>67/5 (0 | 0.102<br>0.067<br>0.016 | 569 (51.9)<br>67 (5.1) | 589 (53.7)<br>61 /5 (0 | 0.011<br>0.027<br>0.023 | 13418.6 (54.3)<br>1379.6 (5.6)<br>4054.1 (16.4) | 620.0 (54.3)<br>66.0 (5.8) |
| 4128(16.1)<br>4906(19.1) | 134 (11.7)<br>625 (54.5)<br>67 (5.8)<br>190 (16.6)<br>216 (18.8) | 0.013 | 67 (6.1)<br>210 (19.2)<br>210 (19.2) | 177 (16.1)<br>202 (18.4) | 0.079 | 4054.1 (16.4)<br>4657.5 (18.9) | 189.0 (16.5)<br>215.0 (18.8) |
| 421 (1.6)<br>82 (0.3) | 11(1.0) | 0.05 | 10 (0.9) | 10 (0.9)<br>1 (0.1) | 0.001 | 218.6 (0.9)<br>20.9 (0.1) | 11.0 (1.0)<br>1.0 (0.1) |
| 1192 (4.6)<br>2566 (10.0) | 50(4.4)<br>115(10.0) | 0.014 | 46 (4.2)<br>112 (10.2) | 67 (6.2)<br>107 (9.8) | 0.005 | 1060.0 (4.3)<br>2455.1 (9.9) | \$0.0 (4.4)<br>114.0 (10.0) |
| 2092 (8.2) | 70(6.1)<br>181 (15.8)<br>14 (3.0)<br>16 (1.4)<br>25 (2.2) | 0.08 | 64 (5.8) | 68 (6.2)<br>171 (15.6) | 0.015 | 1510.6(6.1) | 68.0 (6.0) |
| 4877 (19.0)<br>1614 (6.3)<br>532 (2.1)<br>302 (1.2) | 34(3.0)<br>16(1.4) | 0.052 | 167 (15.2)<br>36 (3.2)<br>15 (1.4)<br>24 (2.2) | 171 (15.6)<br>14 (3.1)<br>15 (1.4)<br>23 (2.1) | 0.01 | 3810.3 (15.4)<br>764.6 (3.0)<br>319.6 (1.3)<br>489.8 (2.0) | 179.0 (15.7)<br>34.0 (3.0)<br>16.0 (1.4)<br>25.0 (2.2) |
| | | 0.078 | | | 0.006 | | |
| 1.17 (D.84)<br>4225 (16.5) | 1.33 (0.93)<br>273 (23.8) | 0.177 | 1.32 (0.88)<br>250 (22.8) | 1.31 (0.92)<br>251 (22.9) | 0.002 | 1.31 (0.89)<br>5825.1 (23.6) | 1.32 (0.92)<br>271.0 (23.7) |
| 417 (1.6)<br>9429 (36.8) | 14 (1.2)<br>402 (35.0) | 0.036 | 8 (0.7)<br>377 (34.4) | 14 (1.3)<br>387 (35.3) | 0.019 | 291.8 (1.2)<br>8647.2 (35.0) | 299.0 (34.9)<br>245.0 (65.2) |
| 1538 (6.0)<br>2157 (8.4) | 402 (35.0)<br>748 (65.2)<br>92 (8.1)<br>260 (22.7)<br>12 (1.0) | 0.082 | 736 (67.2)<br>83 (7.6)<br>217 (19.8)<br>8 (9.7)<br>786 (7.7) | 86 (7.8)<br>224 (20.4) | 0.01 | 1992.8 (8.1) | 93.0 (8.1) |
| 112 (0.4)<br>17644 (68.8) | 12 (1.0)<br>826 (72.0) | 0.071 | 8 (0.7)<br>786 (71.7) | 10 (0.9)<br>789 (72.0) | 0.02 | 233.0 (0.9)<br>17729.1 (71.8) | 256.0 (22.4)<br>11.0 (1.0)<br>823.0 (72.1) |
| 17544 (68.8)<br>6945 (27.1)<br>15562 (60.7) | 826 (72.0)<br>324 (28.2)<br>701 (61.1) | 0.07<br>0.026<br>0.009 | 786 (71.7)<br>319 (29.1)<br>676 (61.7) | 789 (72.0)<br>308 (28.1)<br>669 (61.0) | 0.022 | 17729.1 (71.8)<br>7017.4 (28.4)<br>14993.1 (60.7) | \$22.0 (28.2)<br>697.0 (61.0) |
| 9595 (37.4)<br>6795 (26.5) | 396 (34.5)<br>310 (27.0) | 0.05<br>0.012<br>0.054 | 296 (26.1)<br>290 (26.5) | 382 (34.9)<br>297 (27.1) | 0.014<br>0.003 | 8635.5 (35.0)<br>6658.2 (27.0) | 296.0 (34.7)<br>308.0 (27.0) |
| 2291 (8.9)<br>2959 (11.5)<br>1092 (4.3)<br>1001 (3.9) | 121 (10.5)<br>137 (11.9)<br>44 (2.8)<br>37 (3.2) | 0.054 | 115 (10.5)<br>102 (9.3)<br>42 (2.8)<br>25 (3.2) | 116(10.6)<br>131(12.0)<br>42(2.8)<br>16(2.3) | 0.003 | 3590.9(10.5)<br>3949.6(11.9)<br>938.4 (3.8)<br>780.6 (3.2) | 120.0 (10.5)<br>135.0 (11.8) |
| 1092 (4.3)<br>1001 (3.9)<br>6462 (25.2) | 84 (3.8)<br>37 (3.2) | 0.022 | 42 (3.8)<br>35 (3.2)<br>270 (24.6) | 42 (3.8)<br>36 (3.3) | 0.001 | 938.4 (3.8)<br>780.6 (3.2)<br>6231.2 (25.2) | 44.0 (3.9)<br>37.0 (3.2)<br>290.0 (25.4) |
| 20202 (79.8) | 291 (25.4)<br>932 (81.3) | 0.004 | 888 (81.0) | 280 (25.5)<br>487 (80.9) | 0.021 | 20020.1 (81.1) | 928.0 (81.3) |
| 3179(12.4)<br>4999(19.5) | 194 (16.9)<br>221 (19.3) | 0.006 | 177 (16.1)<br>220 (20.1) | 175 (16.0)<br>214 (19.5) | 0.014 | 4111.5(16.6)<br>4779.6(19.4) | 292.0 (16.8)<br>219.0 (19.2) |
| 4640(18.1)<br>4496(17.5)<br>3498(13.6) | 189 (16.5)<br>210 (18.3)<br>122 (10.6)<br>32 (2.8) | 0.02 | 210 (19.2)<br>215 (11.4) | 180(16.4)<br>199(18.2)<br>119(10.9) | 0.026 | 3978.1(16.1)<br>4587.7(18.6)<br>2640.1(10.7) | 210.0 (18.4)<br>210.0 (18.4) |
| 710 (2.8)<br>5385 (21.0) | 246 (21.4) | 0.001 | 28 (2.5)<br>256 (23.4) | 31 (2.8)<br>232 (21.2) | 0.037 | 671.8 (2.7)<br>5315.2 (21.5) | 32.0 (2.8)<br>245.0 (21.5) |
| 7452 (29.1)<br>4802 (18.7) | 339 (29.6)<br>243 (21.2) | 0.011 | 329 (30.0)<br>227 (20.7) | 325 (29.7)<br>228 (20.8) | 0.008 | 7328.2 (29.7)<br>5212.8 (21.1) | 237.0 (29.5)<br>242.0 (21.2) |
| 2674 (10.4)<br>1638 (6.4) | 118 (10.3)<br>83 (7.2) | 0.005 | 118 (10.8)<br>68 (6.2) | 114(10.4)<br>79(7.2) | 0.012 | 2560.8(10.4)<br>1752.6(7.1) | \$1.0 (10.3)<br>\$1.0 (7.1) |
| 1377 (5.4) | 39 (3.4) | 0.094 | 37 (3.4) | 37 (3.4) | 0.001 | \$29.9 (3.4) | 38.0 (3.3) |
| 2.13 (2.21) | 0.19 (0.05) | 0.158 | 0.19(0.05) | 0.19 (0.05) | 0.012 | 0.19 (0.05) | 0.19 (0.05) |
| 0.20 (0.06)<br>11.35 (4.78) | 11.93(4.72) | 0.123 | 0.19 (0.05)<br>11.91 (4.84) | 0.19 (0.05)<br>11.84 (4.67) | 0.013 | 0.19 (0.05) | 11.91 (4.70) |
| 11.46 (4.87) | 12.07 (4.82) | 0.125 | 12.05 (4.97) | 11.98 (4.78) | 0.015 | 12.05 (5.10) | 12.05 (4.81) |
| 2663 (10.4)<br>3901 (15.2) | 67 (5.8) | 0.167 | 72 (6.6)<br>116 (10.6) | 65 (5.9)<br>114 (10.4) | 0.026<br>0.006<br>0.036 | 1434.4 (5.8)<br>2484.4 (10.1) | 67.0 (5.9)<br>117.0 (10.2) |
| 7513 (29.3) | 118 (10.3)<br>247 (21.5) | 0.179 | 221 (20.2) | 237 (21.6) | 0.036 | 5241.6(21.2) | 246.0 (21.5) |
| 5.28 (7.52)<br>1223 (12.6) | 6.63 (7.56)<br>187 (16.3) | 0.046 | 6.78 (10.94)<br>171 (15.6) | 6.30 (5.76)<br>164 (15.0) | 0.055 | 6.50 (8.69)<br>1994.2 (16.2) | 6.54 (7.11)<br>184.0 (16.1) |
| 12276 (47.9)<br>21170 (82.6) | \$16 (45.0)<br>920 (80.2) | 0.058 | 489 (44.6)<br>859 (78.4) | 484 (44.2)<br>877 (80.0) | 0.009 | 11011.3 (44.6)<br>19818.8 (80.2) | \$12.0 (44.8)<br>915.0 (80.1) |
| 0.99 (2.25) | 0.85 (2.17) | 0.065 | 0.83 (1.75) | 0.85 (2.20) | 0.011 | 0.83 (1.90) | 0.85 (2.17) |
| 0.31 (0.83) | 0.34 (1.48) | 0.023 | 0.35 (1.43) | 0.29 (0.77) | 0.05 | 0.23 (1.24) | 0.34 (1.48) |
| 1.46 (1.33) | 1.55 (0.92) | 0.076 | 1.54 (1.15) | 1.52 (0.90) | 0.011 | 1.55 (1.32) | 1.54 (0.92) |
| 0.55 (0.12) | 0.61 (5.51) | 0.013 | 0.45 (1.20) | 0.61 (5.63) | 0.041 | 0.60 (4.10) | 0.61(5.52) |
| 1.01 (1.01) | 1.13 (0.95) | 0.123 | 1.09 (1.15) | 1.10 (0.85) | 0.007 | 1.13 (1.41) | 1.13 (0.93) |
| 0.05 (0.47)<br>876 (3.4) | 0.04 (0.35)<br>40 (0.5) | 0.022 | 0.03 (0.23)<br>43 (2.9) | 0.04 (0.35)<br>38 (3.5) | 0.027 | 0.04 (0.47)<br>853.7 (3.5) | 0.04 (0.35)<br>40.0(2.5) |
| 22833 (89.0)<br>2185 (8.5) | 40 (2.5)<br>1049 (91.5)<br>93 (8.1)<br>87 (7.6) | 0.081 | 998 (91.1)<br>95 (8.7) | 1000 (91.2)<br>91 (8.3) | 0.006 | 22616.2 (91.6)<br>2020.6 (8.2) | 1045.0(91.5)<br>93.0(8.1) |
| 2040 (8.0)<br>3722 (14.5) | 87 (7.6)<br>215 (18.7) | 0.014 | 94 (8.6)<br>200 (18.2) | 85 (7.8)<br>200 (18.2) | 0.03 | 1891.5 (7.7)<br>4601.5 (18.6) | 87.0(7.6)<br>212.0(18.6) |
| 1058 (4.1) | 48 (4.2) | 0.003 | 41(3.9) | 45 (4.1) | 0.009 | 1022.0(4.1) | 47.0 (4.1) |
| 11162 (43.5)<br>5013 (19.5)<br>6464 (25.2)<br>937 (3.7) | \$09 (44.4)<br>\$91 (34.1)<br>\$61 (22.8)<br>\$8 (3.3) | 0.017 | 484 (44.2)<br>352 (32.1)<br>247 (22.5)<br>36 (3.3) | 45 (4.1)<br>476 (43.4)<br>368 (33.6)<br>255 (23.3)<br>37 (3.4) | 0.015<br>0.031<br>0.017 | 10904.2 (44.2)<br>8435.8 (34.2)<br>5621.7 (22.8)<br>815.2 (3.3) | \$06.0 (44.2)<br>288.0 (24.0)<br>260.0 (22.8)<br>28.0 (3.3) |
| 5464 (25.2)<br>927 (2.7)<br>1017 (4.0) | 261 (22.8)<br>28 (2.3)<br>57 (5.0) | 0.057 | 247 (22.5)<br>36 (2.2)<br>45 (4.1) | 255 (23.3)<br>27 (3.4)<br>56 (5.1) | 0.005 | \$621.7(22.8)<br>815.2(3.3)<br>1268.6(5.1) | 260.0 (22.8)<br>28.0 (3.3)<br>57.0 (5.0) |
| 19535 (76.6) | 921 (80.3) | 0.049 | 45 (4.1)<br>897 (81.8) | 56 (5.1)<br>878 (80.1) | 0.048 | 19852.9 (80.4) | 918.0 (80.4) |
| 1157 (4.5) | 51 (4.4)<br>89 (7.8) | | 47 (4.3)<br>21 (6.5) | 49 (4.5)<br>87 (7.9) | | 1121.4 (4.5) | 50.0 (4.4)<br>99.0 (7.8) |
| 854 (3.3)<br>1332 (5.2)<br>6578 (25.7) | 24 (2.1)<br>62 (5.4)<br>283 (24.7) | 1 1 | 26(2.4) | 24 (2.2)<br>58 (5.3)<br>273 (24.9) | - | \$13.5 (2.1)<br>1315.5 (5.3)<br>6073.9 (24.6) | 24.0 (2.1)<br>61.0 (5.3)<br>281.0 (24.6) |

| Stagliptin - reference<br>1,096 | Semaglutide - exposure<br>1,096 | Stddff | Sitagliptin - reference<br>24,697 |
|---|---|---|---|
| 73.2916.281 | 73.26 (5.97) | 0.004 | 73.12 (6.05) |
| 530 (48.4) | | | 11504.9 [46.6] |
| 530 (48.4) | \$19(47.4) | 0.064 | 11504.9 [46.6] |
| 175 (16.0) | 187 (17.1) | | 4089.1 (16.6) |
| 481 (43.9) | 484 (44.2) | | 10889.4 (44.1) |
| 236 (21.5) | 246 (22.4) | 0.086 | \$719.6(23.2) |
| (2.4) | 12 (1.1) | | 109.7 (1.3) |
| 68 (5.2)<br>86 (7.8) | \$5 (7.8) | | 1819.9(7.4) |
| 602 (26.7)<br>536 (46.5) | 401 (36.6)<br>532 MB 51 | | 12220 2 (95.4) |
| | 101(100) | | |
| 1.00.00 | 120.20 | 0.027 | 200.00.00 |
| 2 (0.2) | 4 (0.4) | 0.035 | 86.2 (0.3) |
| 22 (2.0) | 17 (1.6) | 0.035 | 362.9 (1.5)<br>3453.639.61 |
| 124 (11.3)<br>212 (19.3) | 212 (19:3)<br>187 (17:1) | 0.001 | 4865.6(19.7)<br>4364.4(17.7) |
| 181 (16.5)<br>221 (20.2) | 187 (17.1)<br>233 (21.3) | 0.015 | 4364.4(17.7)<br>5439.7(22.0) |
| 160 (14.6)<br>56 (5.1) | 158 (14.4)<br>66 (6.0) | 0.005 | 3480.5 (14.1)<br>1462.4 (5.9) |
| 236 (21.5) | 210(19.2) | 0.059 | 4836.3 (19.6) |
| 236 (21.5) | 210(19.2) | 0.059 | 4836.3 (19.6) |
| 25 (2.3) | 18 (1.6) | 0.046 | 406.5 (1.6) |
| 12 (7.5)<br>20 (1.8) | 81 (7.4)<br>17 (1.6) | 0.003<br>0.021<br>0.015 | 1818.8 (7.4) |
| 20 (1.8)<br>53 (5.7) | 17 (1.6)<br>67 (6.1)<br>10 (0.9)<br>92 (8.4)<br>435 (39.7)<br>796 (72.6) | 0.015 | 407.8 (1.7)<br>1599.4 (6.4)<br>204.3 (0.8)<br>2073.3 (8.4)<br>9949.4 (40.3)<br>17964.9 (72.7) |
| 1 (0.7)<br>35 (8.7) | 10 (0.9)<br>92 (0.4) | 0.02 | 204.3 (0.8) |
| (36 (29.8)<br>106 (73.5) | 435 (39.7) | 0.002 | 9949.4 (40.3) |
| 564 (SB.B) | | 0.056 | |
| 544 (58.8)<br>166 (15.1)<br>15.17 31 | 158 (14.4)<br>26 (2.4) | 0.021 | 3531.1 (14.3)<br>579.7 (2.3) |
| 25 (2.3)<br>57 (5.2) | 67 (6.1) | 0.04 | 1512.1 (6.1) |
| 535 (48.8)<br>161 (14.7) | \$38(49.1) | 0.005 | 12208.1 (49.4)<br>1624.2 (14.7) |
| 12(1.1) | 164 (15.0) | 0.054 | 417.7 (1.7) |
| 2 (0.2) | 1 (0.1) | 0.025 | 23.5 (0.1)<br>2580.9(14.5) |
| 2 (0.2)<br>162 (14.8)<br>199 (18.2)<br>375 (34.2) | 179(16.3) | 0.048 | 4040.4 (16.4) |
| 179 (16.3) | 361(32.9)<br>180(16.4) | 0.027 | 8135.2(32.9)<br>3982.1(16.1) |
| 179 (16.3)<br>51 (4.7) | \$6 (5.1) | 0.021 | 1247.4 (5.1) |
| 34 (3.1)<br>163 (14.9) | 30 (2.7)<br>151 (13.8) | 0.022<br>0.031<br>0.004 | 715.3 (2.9)<br>3473.4 (14.1) |
| 52 (4.7) | \$1 (4.7) | | 1099.1(4.5) |
| 144 (13.1)<br>33 (3.0) | 155 (14.1)<br>35 (8.2) | 0.029<br>0.011<br>0.029 | 1537.8(14.3)<br>723.7 (2.9) |
| 25 (2.3)<br>58 (5.3) | 30 (2.7)<br>47 (4.3) | 0.029 | 685.8 (2.8)<br>1044.0 (4.2) |
| | | 0.011 | |
| 133 (12.1)<br>569 (51.9)<br>67 (6.1)<br>210 (19.2) | 129(11.8)<br>589(52.7)<br>61(5.6)<br>177(16.1) | 0.037 | 2842.2(11.5)<br>12418.6 (54.3)<br>1279.65.6)<br>4054.1(16.4) |
| 67 (6.1) | 61 (5.6) | 0.023 | 1379.4 (5.6) |
| 210 (19.2) | 177 (16-1)<br>202 (18-4) | 0.079 | 4054.1(16.4)<br>4657.5(18.9) |
| 10 (0.9) | 10 (0.9)<br>1 (0.1) | 0.001 | 218.6 (0.9)<br>20.9 (0.1) |
| 0 (0.0)<br>46 (4.2) | 1 (0.1)<br>47 (4.3) | 0.005 | 20.9 (0.1)<br>1060.0(4.3) |
| 112 (10.2) | 107 (9.8) | 0.015 | 2455.1(9.9) |
| 64 (S.B)<br>167 (15.2) | 68 (6.2)<br>171 (15.6) | 0.01 | 1510.6(6.1)<br>3810.3(15.4) |
| 36(3.3) | 24 (2.1) | 0.01 | 744.6 (3.0) |
| 15 (1.4)<br>24 (2.2) | 15 (1.4)<br>23 (2.1) | 0.001 | 489.8 (2.0) |
| 1.32 (0.88) | 1.31 (0.92) | 0.016 | 1.31 (0.89) |
| 250 (22.8) | 251(22.9) | 0.002 | \$825.1(23.6) |
| 1 (0.7)<br>277 (24.4) | 14 (1.3)<br>287 (35.3) | 0.055 | 291.8 (1.2)<br>8647.2 (25.0) |
| 277 (24.4)<br>736 (67.2) | 387 (35.3)<br>708 (64.6) | 0.019 | 8647.2 (25.0)<br>16073.7 (65.1) |
| 83 (7.6)<br>217 (19.8) | 86 (7.8)<br>224 (20.4) | 0.016 | 1992.8 (8.1)<br>5333.5 (21.6) |
| 1 (2.7) | 10 (0.9) | 0.02 | |
| 786 (71.7)<br>319 (29.1) | 789(72.0)<br>208(28.1) | 0.022<br>0.023<br>0.027 | 17729.1 (71.8)<br>7017.4 (28.4)<br>14993.1 (90.7)<br>8625.3 (25.0)<br>6658.2 (27.0)<br>2590.9 (10.5)<br>7949.4 (11.9) |
| 576 (61.7) | 669(61.0)<br>382(34.9)<br>297(27.1)<br>116(10.6)<br>131(12.0) | 0.013 | 14993.1 (60.7) |
| 576 (61.7)<br>396 (36.1)<br>290 (36.5)<br>115 (10.5)<br>102 (9.3) | 297(27.1) | 0.014 | 6658.2 (27.0) |
| 115 (10.5) | 116(10.6) | 0.003 | 2590.9(10.5)<br>2949.6(11.9) |
| (2 (3.8)<br>35 (3.2) | | 0.001 | |
| 15 (3.2)<br>270 (24.6) | 36 (3.3)<br>280 (25.5) | 0.005 | 780.6 (3.2)<br>6231.2 (25.2) |
| 188 (81.0) | \$87 (80.9) | 0.002 | 20020.1 (81.1) |
| 177 (16.1)<br>230 (20.1) | 175(16.0)<br>214(19.5) | 0.014 | 4111.5(16.6)<br>4779.6(19.4) |
| 190 (17.3) | 180(16.4)<br>199(18.2) | 0.024 | 1978.1(16.1)<br>4587.7(18.6) |
| 210 (19.2)<br>125 (11.4) | 119(10.9) | 0.017 | 2640.1(10.7) |
| 28 (2.5)<br>256 (23.4) | 31 (2.8)<br>232 (21.2) | 0.037 | 671.8 (2.7)<br>5315.2 (21.5) |
| 329 (30.0) | 325 (29.7) | 0.008 | 7328 2729 71 |
| 118 (10.8) | 228(20.8)<br>114(10.4) | 0.012 | 5212.8(21.1)<br>2560.8(10.4) |
| 68 (6.2)<br>37 (3.4) | 79 (7.2)<br>37 (3.4) | 0.04 | 1752.6 (7.1)<br>829.9 (3.4) |
| 1.84 (2.01) | 1.81 (1.91) | 0.012 | 3.80 (3.97) |
| 0.19 (0.05) | 0.19 (0.05) | 0.007 | 0.19 (0.05) |
| 11.91(4.84) | 11.84 (4.67) | 0.013 | 11.91 (5.00) |
| 17 05 (4 97) | 11 98 (4 76) | 0.015 | 12.05.5.100 |
| 12.05 (4.97)<br>72 (6.6)<br>116 (10.6) | 11.98 (4.78)<br>45 (5.9)<br>114 (10.4) | 0.026 | 12.05 (5.10)<br>1434.4 (5.8)<br>2484.4 (10.1) |
| 116 (10.6)<br>221 (20.2) | 114(10.4)<br>237(21.6) | 0.006 | 2484.4 (10.1)<br>5241.6 (21.2) |
| 5.78 (10.94)<br>171 (15.6) | 6.30 (5.76)<br>164 (15.0) | 0.055 | 6.50 (8.69)<br>1994.2 (16.2) |
| 489 (44.6) | 484 (44.2) | 0.009 | 11011.3 (44.6) |
| 859 (78.4) | 877 (80.0) | 0.04 | 19818.8 (80.2) |
| 0.83 (1.75) | 0.85 (2.20) | 0.011 | 0.83 (1.90) |
| 2.35 (1.43) | 0.29 (0.77) | 0.05 | 0.33 (1.24) |
| F40.10 | 1 53 50 000 | 0.0** | 1777033 |
| | a. ea (0.90) | 0.011 | 1.55 (1.42) |
| 0.45 (1.20) | 0.61 (5.63) | 0.041 | 0.60 (4.10) |
| 1.09 (1.15) | 1.10 (0.85) | 0.007 | 1.11(1.41) |
| 0.03 (0.23) | 0.04 (0.35) | 0.027 | 0.04 (0.47) |
| (2 (2.9) | 28 (2.5) | 0.027 | 853.7 (8.5) |
| 998 (91.1) | 1000 (91.2)<br>91 (8.3) | 0.006 | 22616.2 (91.6)<br>2020.6 (8.2) |
| | | 0.01 | 1891.5(7.7) |
| 94(8.6) | 85 (7.8) | 0.001 | 4601.5 (18.6) |
| 74 (8.6)<br>200 (18.2) | 85 (7.8)<br>200 (18.2) | | 1022.0(4.1) |
| 94 (8.4)<br>200 (18.2)<br>43 (3.9) | 85 (7.8)<br>200 (18.2)<br>45 (4.1) | 0.009 | |
| 152 (12.1) | 85 (7.8)<br>200 (18.2)<br>45 (4.1)<br>476 (43.4)<br>168 (33.6) | 0.009<br>0.015<br>0.031 | 10904.2 (44.2)<br>8435.8 (34.2) |
| 247 (22.5) | 268(22.6)<br>255(23.3) | 0.009<br>0.015<br>0.031<br>0.017 | 8435.8 (34.2)<br>5621.7 (22.8) |
| 352 (32.1) | 161(33.6) | 0.031 | \$435.8 (34.2) |
| 352 (32.1)<br>247 (32.5)<br>36 (3.3)<br>45 (4.1) | 368 (33.6)<br>355 (23.3)<br>37 (3.4)<br>56 (5.1) | 0.031 | 8425.8 (24.2)<br>5621.7 (22.8)<br>815.2 (3.3)<br>1268.6 (5.1) |
| 352 (32.1)<br>247 (22.5)<br>36 (3.3)<br>45 (4.1)<br>897 (81.8)<br>47 (4.3) | 268 (23.6)<br>255 (23.3)<br>27 (2.4)<br>56 (5.1)<br>878 (80.1)<br>49 (4.5) | 0.031 | 8435.8 (34.2)<br>5631.7 (22.8)<br>815.2 (3.3)<br>1268.4 (5.1)<br>19852.9 (80.4)<br>1123.4 (6.5) |
| 352 (32.1)<br>247 (32.5)<br>36 (3.3)<br>45 (4.1) | 368 (33.6)<br>355 (23.3)<br>37 (3.4)<br>56 (5.1) | 0.031 | 8425.8 (24.2)<br>5621.7 (22.8)<br>815.2 (3.3)<br>1268.6 (5.1) |

| | Fine stratification cohort | |
|---|---|---|
| Situgliptin - reference<br>4,697 | Semaglutide - exposure<br>1,142 | Std diff |
| | | 0.001 |
| 1304.9 [46.6] | p.4.4.0 [46.7] | 0.002 |
| 089.1(16.6)<br>998.9(16.2) | 195.0 (17.1)<br>185.0 (16.2) | = |
| 0889.4 (44.1)<br>719.6/23.21 | 503.0 (44.0)<br>250.0 (22.7) | |
| | | 0.031 |
| 09.7 (1.3)<br>244.2 (5.4) | 11.0 (1.0)<br>66.0 (5.8) | |
| 819.9 (7.4)<br>983.9 (36.4) | 85.0 (7.4)<br>413.0 (36.2) | |
| 2239.3 [49.6] | 567.0 (49.6) | |
| | | L., |
| 00.9 (1.2)<br>6.2 (0.3) | 14.0 (1.2)<br>4.0 (0.4) | 0.001 |
| 62.9 (1.5)<br>453.6(9.9) | 17.0(1.5) | 0.002 |
| 865.6 (19.7)<br>364.4 (17.7) | 229.0 (20.1) | 0.009 |
| 439.7 (22.0) | 255.0 (22.3) | 0.007 |
| 480.5 (14.1)<br>462.4 (5.9) | 164.0 (14.4)<br>66.0 (5.8) | 0.006 |
| 462.4 (5.9)<br>836.3 (19.6)<br>836.3 (19.6) | 224.0 (19.6)<br>224.0 (19.6) | 0.001 |
| 181.9(8.8) | 224.0 (19.6)<br>100.0 (8.8) | 0.003 |
| 09.5 (1.6)<br>818.8 (7.4) | 84.0 (7.4) | 0.001 |
| 07.8 (1.7)<br>590.4 (6.4) | 20.0 (1.8)<br>74.0 (6.5) | 0.008 |
| 04.3 (D.B) | 10.0 (0.9) | 0.005 |
| 949.4 (40.3) | 463.0 (40.5) | 0.005 |
| 7964.9 (72.7)<br>3844.1 (56.1) | 830.0 (72.7)<br>641.0 (56.1) | 0.001 |
| 531.1(14.3) | 165.0 (14.4)<br>27.0 (2.4) | 0.004 |
| 18 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 69.0 (6.0) | 0.003 |
| 2208.1 (49.4)<br>624.2 (14.7) | 567.0 (49.6)<br>168.0 (14.7) | 0.004 |
| 17.7 (1.7)<br>3.5 (0.1) | 10.0 (1.8)<br>1.0 (1.1)<br>1.67.0 (14.6)<br>186.0 (16.3)<br>173.0 (32.7) | 0.005 |
| 590.9(14.5) | 167.0 (14.6) | 0.004 |
| 135.2 (32.9) | 273.0 (32.7) | 0.006 |
| 982.1(16.1)<br>247.4(5.1) | 186.0 (16.3)<br>60.0 (5.3) | 0.004 |
| 15.3 (2.9) | 32.0 (2.8)<br>162.0 (14.2) | 0.006 |
| 099.1(4.5) | 162.0 (14.2)<br>51.0 (4.5) | 0.001 |
| 247.8(14.3)<br>23.7(2.9) | 165.0 (14.4)<br>35.0 (3.1) | 0.004 |
| 85.8 (2.8)<br>044.0(4.2) | 32.0 (2.8)<br>49.0 (4.3) | 0.002 |
| 643 3/01 F | | 200 |
| 842.2 (11.5)<br>3418.6 (54.3) | 122.0 (11.6)<br>620.0 (54.2) | 0.004 |
| 842.2(11.5)<br>3418.6 (54.3)<br>379.6 (5.6)<br>054.1 (16.4)<br>657.5 (18.9) | 66.0 (5.8)<br>189.0 (16.5) | 0.008 |
| | 215.0 (18.8) | 0.001 |
| 0.9 (0.1) | 1.0 (0.1) | 0.001 |
| 0.9 (0.1)<br>060.0 (4.3)<br>455.1 (9.9) | 50.0 (4.4)<br>114.0 (10.0) | 0.004 |
| 510.6(6.1) | 68.0 (6.0)<br>179.0 (15.7) | 0.007 |
| 44.6 (2.0) | 179.0 (15.7)<br>34.0 (3.0) | 0.002 |
| 455.1(9.9)<br>510.6(6.1)<br>810.3(15.4)<br>44.6(2.0)<br>19.6(1.3)<br>89.8(2.0) | 16.0 (1.4)<br>25.0 (2.2) | 0.009 |
| .31 (0.89) | 1.32 (0.92) | 0.014 |
| 31 (0.89)<br>825 1(23.6)<br>825 1(23.6)<br>647.2 (35.0)<br>647.2 (35.0)<br>647.2 (35.0)<br>922.8 (8.1)<br>323.5 (21.6)<br>321.0 (3.9)<br>7728.1 (71.8) | 1.32 (0.92)<br>271.0 (23.7)<br>14.0 (1.2) | 0.003 |
| 91.8 (1.2)<br>647.2 (35.0) | 14.0 (1.2)<br>399.0 (34.9)<br>345.0 (65.2) | 0.002 |
| 6073.7 (65.1)<br>992.8 (8.1) | 745.0 (65.2)<br>93.0 (8.1) | 0.003 |
| 333.5 (21.6)<br>33.0 m si | 256.0 (22.4) | 0.02 |
| 7729.1 (71.8) | 823.0 (72.1) | 0.006 |
| 017.4 (28.4)<br>4993.1 (60.7) | 322.0 (28.2)<br>697.0 (61.0) | 0.005 |
| 625.5 (35.0) | 296.0 (34.7)<br>208.0 (27.0) | 0.006 |
| 7736.101.8) 0174.028.4) 4893.110.7) 4893.110.7) 483.120.7) 483.120.7) 983.611.9) 983.611.9) 984.62.1) 180.60.2) 180.60.2) 181.2(5.2) 180.60.2) 181.1(6.1) | 120.0 (10.5)<br>135.0 (11.8) | 0.001 |
| 28.4 (3.8) | 44.0 (3.9) | 0.003 |
| 90.6 (3.2)<br>231.2 (25.2) | 27.0 (3.2)<br>290.0 (25.4) | 0.005 |
| 0020.1 (81.1) | 928.0 (81.3) | 0.00S |
| 779.6(19.4) | 219.0 (19.2) | 0.004 |
| 978.1 (16.1)<br>587.7 (18.6) | 219.0 (19.2)<br>189.0 (16.5)<br>210.0 (18.4) | 0.012 |
| 71.8 (2.7) | 121.0 (10.6)<br>32.0 (2.8) | 0.003 |
| 315.2(21.5) | 245.0 (21.5) | 0.002 |
| 212.8(21.1) | 237.0 (29.5)<br>242.0 (21.2) | 0.002 |
| 560.8(10.4)<br>752.6(7.1) | 118.0 (10.2)<br>81.0 (7.1) | 0.001 |
| 29.9 (3.4) | 38.0 (3.3) | 0.002 |
| .80 (1.97) | 1.80 (1.91) | 0.004 |
| 19 (0.05) | 0.19 (0.05) | 0.003 |
| 1.91 (5.00) | 11.91 (4.70) | 0.002 |
| 100 (0.10) | 1205 (400) | 2.00 |
| 2 US (5.10)<br>434.4 (5.8) | 12.05 (4.81)<br>67.0 (5.9) | 0.001 |
| 484.4(10.1)<br>241.6(21.2) | 117.0 (10.2)<br>246.0 (21.5) | 0.006 |
| romen. | erecon. | 200 |
| .50 (8.69)<br>994.2 (16.2) | 9-36 (7.11)<br>184.0 (16.1) | 0.002 |
| | \$12.0 (64.8)<br>915.0 (80.1) | 0.005 |
| 1011.3 (44.6)<br>9818.8 (80.2) | | |
| 1011.3 (44.6)<br>9818.8 (80.2) | 0.65 (2.17) | 0.000 |
| 1011.3 (44.6)<br>9818.8 (80.2)<br>(83 (1.90) | 0.85 (2.17) | 0.009 |
| 10113 (44.6)<br>9818.8 (80.2)<br>183 (1.90) | 0.85 (2.17)<br>0.34 (1.48) | 0.009 |
| 1011.3 (44.6)<br>9818.8 (80.2)<br>(83 (1.90)<br>(33 (1.24) | 0.85 (2.17)<br>0.34 (1.48)<br>1.54 (0.92) | 0.009 |
| 1011.3 (44.6)<br>9818.8 (80.7)<br>83 (1.90)<br>33 (1.24)<br>35 (1.32) | 0.85 (2.17)<br>0.34 (1.48)<br>1.54 (0.92)<br>0.61(5.52) | 0.009<br>0.01<br>0.003<br>0.001 |
| 1011.3 [44.6]<br>9818.8 [90.7]<br>(83 [1.90]<br>(23 [1.24]<br>(55 [1.27])<br>(60 [4.10]<br>(12 [1.41]) | 0.85 (2.17)<br>0.34 (1.48)<br>1.54 (0.92)<br>0.61 (5.52)<br>1.13 (0.93) | 0.009<br>0.01<br>0.003<br>0.001 |
| 1011.3 (44.6)<br>9818.8 (90.7)<br>(81 (1.90)<br>132 (1.24)<br>.55 (1.22)<br>.60 (4.10)<br>.13 (1.41) | 0.85 (2.17)<br>0.34 (1.48)<br>1.54 (0.52)<br>0.61 (5.52)<br>1.12 (0.93) | 0.009<br>0.01<br>0.003<br>0.001 |
| 1011.2 (44.5)<br>9318.8 (80.7)<br>133 (1.90)<br>132 (1.24)<br>135 (1.32)<br>140 (4.10)<br>131 (1.41)<br>140 (1.64)<br>151 (1.41) | 9.85 (2.17)<br>9.34 (1.48)<br>1.54 (9.92)<br>9.61 (5.52)<br>1.13 (9.93)<br>9.04 (9.15)<br>40.2(2.5) | 0.009<br>0.01<br>0.003<br>0.001<br>0.007 |
| 1091.3 (44.6)<br>991.6 (10.9)<br>1.33 (1.24)<br>.55 (1.27)<br>.60 (4.10)<br>.11 (1.41)<br>.12 (1.41)<br>.13 (1.41)<br>.14 (1.41)<br>.15 (1.41)<br>.15 (1.41)<br>.16 (1.41)<br>.17 (1.41) | 0.85 (2.17)<br>9.34 (1.48)<br>1.54 (0.92)<br>1.61 (5.52)<br>1.12 (0.93)<br>3.04 (0.35)<br>40.9 (1.5)<br>104.0 (1.91)<br>104.0 (1.91) | 0.009<br>0.01<br>0.003<br>0.001<br>0.007<br>0.002<br>0.002<br>0.002 |
| 1091.3 [44.4]<br>991.8 [109.7]<br>182 [109]<br>132 [1.24]<br>135 [1.37]<br>140 [1.37]<br>141 [1.41]<br>1 | 0.85 (2.17)<br>0.34 (1.48)<br>1.54 (0.92)<br>0.61 (5.52)<br>1.12 (0.92)<br>0.04 (0.35)<br>0.04 (0.35)<br>1.04 (0.915) | 0.009<br>0.01<br>0.001<br>0.001<br>0.002<br>0.002<br>0.002<br>0.002<br>0.002 |
| 10913 (H-4.5)<br>99188 (B0.7)<br>182 (2.90)<br>132 (2.24)<br>132 (2.24)<br>135 (2.27)<br>136 (4.10)<br>137 (2.27)<br>137 (2.27)<br>137 (2.27)<br>138 (2.27)<br>139 (2.27)<br>1 | 9.85 (2.17)<br>9.34 (1.48)<br>1.54 (9.52)<br>9.61 (5.57)<br>1.13 (9.52)<br>9.04 (9.35)<br>49.9(2.5)<br>10.94 (9.15)<br>10.94 (9.15 | 0.009<br>0.01<br>0.001<br>0.007<br>0.002<br>0.002<br>0.002<br>0.002 |
| 1011.3 (4.4) 0318.8 (8.7) 131(1.90) 131(1.90) 131(1.24) 155(1.32) 156(1.32) 154(1.31) | 5.85 (2.17) 3.34 (1.48) 1.54 (9.52) 3.61 (5.12) 3.61 (5.12) 3.64 (9.15) 4.76 (9.15) 3.76 (9.15) 3.76 (9.15) 3.76 (9.15) 3.76 (9.15) 3.77 (9.15) 3.77 (9.15) 3.77 (9.15) 3.77 (9.15) 3.77 (9.15) | 0.009 0.01 0.001 0.001 0.001 0.002 0.002 0.002 0.002 0.001 0.002 |
| 10913 (H4.4) 09188 (B.7) 183 (1.90) 183 (1.90) 183 (1.90) 183 (1.90) 183 (1.90) 183 (1.90) 183 (1.90) 185 (1.9 | 3 85 (2.17) 3 34 (1.48) 154 (9.57) 54 (5.17) 54 (5.17) 54 (5.17) 119 (3.91) 100 (3.91) 100 (3.91) 17.0 (2.61) 17.0 (2.61) 17.0 (3.61) 17.0 (3.61) 18.0 (3.11) 18.0 (3.11) 18.0 (3.11) 18.0 (3.11) 18.0 (3.11) 18.0 (3.14) | 0.009 0.01 0.001 0.001 0.002 |
| 10913 (44.4) 10913 (44.4) 10914 (19.7) 131 (1.24) 135 (1.32) 146 (4.10) 137 (1.41) 146 (3.47) 157 (3.9) 147 (3.9) 148 (3.9) 158 (3.9) 159 (3.9) 169 (3.9) 169 (3.9) 179 (3.9) 189 (3.9) 18 | 3-85 (3.17) 3-86 (1.46) 3-86 (1.46) 3-86 (1.47) 3-86 ( | 0.009 0.01 0.003 0.003 0.007 0.007 0.002 0.003 |
| 1911 3 (44.4)<br>9114 4 (92.2)<br>133 (1.90)<br>134 (1.24)<br>134 (1.24)<br>135 (1.31)<br>136 (1.31)<br>137 (1.31) | 3-85 (2.17) 3-86 (1.46) 1-56 (0.52) 8-61 (1.57) 1-16 (0.52) 1-16 (0.52) 1-16 (0.53) 4-0 (1.5) 1-16 (0.53) 1-16 (0.54) 1-16 (0 | 0.009 0.01 0.003 0.003 0.007 0.007 0.002 |
| 1931.144.61 931.149.61 1331.144.61 931.149.71 1331.149 13 | 3.85 (3.17) 3.86 (1.48) 1.84 (3.52) 3.41 (3.52) 3.42 (3.52) 3.43 (3.52) 3.44 (3.52) 3.45 | 0.000<br>0.01<br>0.001<br>0.001<br>0.002 |
| 190.1144.6) 191.1144.6) 191.11 | 2.85 (2.17) 2.86 (1.46) 2.86 (1.87) 2.86 (1.87) 2.86 (1.87) 2.17 ( | 0.009 0.01 0.003 0.001 0.007 0.007 0.002 |

| Covariates | Source |
|---|---|
| Region | If region not available, from State, https://www2.census.gov/geo/pdfs/maps-data/maps/reference/us_regdiv.pdf |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://hcup- |
| | us.ahrq.gov/datainnovations/ICD-10CaseStudyonOpioid-RelatedIPStays042417.pdf, |
| Drug abuse or dependence | https://stacks.cdc.gov/view/cdc/59394, https://pubmed.ncbi.nlm.nih.gov/34134872/ |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, |
| | https://espace.curtin.edu.au/bitstream/handle/20.500.11937/34117/19233_downloaded_stream_325.pdf?isAllo |
| Alcohol abuse or dependence | wed=y&sequence=2 |
| Underweight or normal weight | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Overweight | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Obese | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Severe Obese | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| Unspecified obesity | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ |
| | Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic- |
| | packages/browse?at=refs%2Fheads%2Fcder_mpl2p_wp015, |
| | https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic- |
| | packages/browse?at=refs%2Fheads%2Fcder_sir_wp002, https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| | https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/, |
| Smoking | https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/ |
| 50 L 10 L 10 L 10 L | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| Diabetic retinopathy | https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Dishatia na una sastiu. | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| Diabetic neuropathy | https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Diabetic nephropathy | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, |
| | https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, https://www.health.mil/Reference- |
| Disheta with was sifted as 10 mg | Center/Publications/2016/03/01/Diabetes-Mellitus, http://www.icd9data.com/2014/Volume1/240-279/249- |
| Diabetes with unspecified complication | 259/250/default.htm, https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11- |
| Diabetes with other ophthalmic manifestations | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion |
| | Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, |
| | https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus, |
| Disheter with peripheral size-ulate and dis-ulate- | http://www.icd9data.com/2014/Volume1/240-279/249-259/250/default.htm, |
| Diabetes with peripheral circulatory disorders | https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11- |
| Diabetic foot + Lower extremity amputation | Investigator review of codes based on: (modified codes) https://pubmed.ncbi.nlm.nih.gov/36102675/ |
| Skin infections | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion |
| | Investigator review of codes based on: the paper then used ICD9/ICD10 website to expand it, |
| Fractile durfunction | https://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-N53/N52-, |
| Erectile dysfunction | https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/ |
| Hynoglycemia | Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ |
| Hypoglycemia | IICCho://haniiiea:ucn:uiiii:liiii:80x/22042102/ |

Hyperglycemia, DKA, HONK

Hypertension

Hyperlipidemia

Atrial fibrillation
Acute MI
Old MI
Coronary atherosclerosis
History of CABG/PTCA
Previous cardiac procedure
Cerebrovascular procedure
Ischemic stroke
PVD diagnosis or surgery
CKD stage 3-4

Other cardiac dysrhythmia

Cardiomyopathy

Valve disorders COPD

Asthma

Obstructive sleep apnea

Investigator review of codes based on:

Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/, https://pubmed.ncbi.nlm.nih.gov/38262528/HONK: https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnovation/DEF/DKA.pdf

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4910677/

algorithm (any care setting, any diagnosis position)

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

 $https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconcepts cardiology 1.pdf, ICD9\ to\ ICD10\ conversion$ 

 $Investigator\ review\ of\ codes\ based\ on:\ https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at=refs\%2Fheads\%2Fcder\_mpl2p\_wp015$ 

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://pubmed.ncbi.nlm.nih.gov/38440888/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp009 Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/

Pneumonia Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/ CKD 1-2 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/ Acute renal disease (AKI) Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, Nephrotic syndrome https://www.cms.gov/icd10m/FY2024-nprmversion41.0-fullcode-cms/fullcode cms/P2401.html Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e29ab67-7a7d-4621-Hypertensive nephropathy 9af3-81bd071bbc67/mmc1.pdf, https://www.icd10data.com/ICD10CM/Codes/I00-I99 Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637. https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion Other renal conditions https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinelanalytic-packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, Modified algorightm from Liver disease https://pubmed.ncbi.nlm.nih.gov/34256144/, Modified CCW algorithm Modified CCW algorithm Hypothyroidism Osteoarthritis Modified CCW algorithm https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder mpl2p wp009 Fractures https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder mpl2p wp015, Falls https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp010 https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Osteoporosis packages/browse?at=refs%2Fheads%2Fcder sir wp002, CCW Algorithms Depression https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms https://pubmed.ncbi.nlm.nih.gov/35043165/ Anxiety Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-and-diagnostic-codes-Sleep disorder 3014779 https://pubmed.ncbi.nlm.nih.gov/35043165/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Dementia packages/browse?at=refs%2Fheads%2Fcder mpl2p wp015 Delirium https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/ COVID https://pubmed.ncbi.nlm.nih.gov/34913208/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/ Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5256065/, https://www.drugs.com/drug-class/antidiabetic-Number of antidiabetic drugs agents.html, https://www.ncbi.nlm.nih.gov/books/NBK279141/ Investigator review of codes based on: https://www.drugs.com, ACE + ARBs https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Thiazide

Investigator review of codes based on: https://www.drugs.com, Beta blockers https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Calcium channel blockers https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Loop diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Other diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes based on: https://www.drugs.com, Nitrates https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ HF drugs (Digoxin + Entresto + Ivabadrine) Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using class I and class II as class 2 is beta blockers and class 4 is Anti-arrhythmics calcium channel blockers) Investigator review of codes based on: https://www.copdfoundation.org/Learn-More/I-am-a-Person-with-COPD/asthma meds COPD/Treatments-Medications.aspx, https://getasthmahelp.org/medications-list.aspx Investigator review of codes based on: https://www.drugs.com, https://www.heart.org/en/health-Statins topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-medications Investigator review of codes based on: https://www.drugs.com, https://www.heart.org/en/health-Other lipid-lowering drugs topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-medications Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK537062/ Antiplatelet agents Investigator review of codes based on: https://www.drugs.com, https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559 Oral anticoagulants Investigator review of codes based on: https://www.drugs.com, **NSAIDs** https://www.ncbi.nlm.nih.gov/books/NBK547742/ Investigator review of codes based on: https://www.drugs.com, https://www.aaaai.org/tools-for-the-public/drug-Oral corticosteroids guide/oral-corticosteroid-medications Investigator review of codes based on: https://www.drugs.com, **Bisphosphonates** https://www.ncbi.nlm.nih.gov/books/NBK470248/ Investigator review of codes based on: https://www.drugs.com, https://pubmed.ncbi.nlm.nih.gov/31643200/#:~:text=They%20can%20also%20be%20informally,%2C%20codeine Opioids %2C%20oxycodone%2C%20hydrocodone%2C Investigator review of codes based on: https://www.drugs.com, Anti-depressants https://www.ncbi.nlm.nih.gov/books/NBK538182/ Gabapentnoids GABAPENTIN, PREGABALIN Investigator review of codes based on: https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-06/Benzodiazepenes-2020.pdf, https://www.ncbi.nlm.nih.gov/books/NBK470159/ Benzodiazepines Investigator review of codes based on: https://www.drugs.com Anxiolytics/hypnotics Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/, https://go.drugbank.com/drugs/DB00382

Dementia meds

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-evaluation-and-management-visitcomplexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-Office visits officeoutpatient-evaluation-and-management-em-visits-fact-sheet.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-**Endocrinologist visit** enrollment-and-certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-Cardiologist visits enrollment-and-certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Internal medicine/family medicine visits Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleId=57326, https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/, https://www.aapc.com/codes/coding-newsletters/my-cardiology-coding-alert/cpt-answer-5-common-ecg-coding-Electrocardiograms questions-175952-article Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/, https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56625&ver=27&, https://www.medicalbillgurus.com/echocardiogram-cpt-Echocardio code/ HbA1c tests received Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Glucose tests ordered Lipid tests ordered Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Creatinine tests ordered Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=59040&ver=4, https://static.cigna.com/assets/chcp/pdf/coveragePolicies/medical/mm 0300 coveragepositioncriteria bone min Bone mineral density test eral density measurement.pdf Basic or comprehensive metabolic blood chem test Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56448&ver=16&bc=0, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm Mammogram Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, http://www.icd9data.com/2012/Volume1/V01-V91/V70-Pap smear V82/V72/default.htm, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-PSA packages/browse?at=refs%2Fheads%2Fcder sir wp002 Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy packages/browse?at=refs%2Fheads%2Fcder sir wp002 Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder sir wp002, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleId=54767&DocID=A54767

Investigator review of codes, Flu vaccine/Pnemococcal vaccine

Telemedicine
Heart failure
TIA
Ankle-brachial index<0.9
Microalbuminuria/proteinuria

DUAL status for medicare ED visit (Medicare) ED visit (Optum)

ED visit (Marketscan)
Hernia (negative control)
Lumbar radiculopathy (negative control)

Cataract surgery (negative control)

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/,

https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-fact-sheet, https://www.aafp.org/family-physician/practice-and-career/getting-paid/coding/coding-telehealth-audio-virtual-digital-visits.html

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Investigator review of codes based on: https://www.cms.gov/medicare-medicaid-coordination/medicare-and-medicaid-coordination/medicare-medicaid-coordination/medicare-medicaid-coordination-gff Revenue center codes: 0450, 0451, 0452, 0456, 0459, 0981; Place of service: 23

Place of service: 23

Service sub-category codes: 10120, 10220, 10320, 10420, 10520, 12220, 20120, 20220, 21120, 21220, 22120, 22320, 30120, 30220, 30320, 30420, 30520, 30620, 31120, 31220, 31320, 31420, 31520, 31620; Place of service: 23

https://pmc.ncbi.nlm.nih.gov/articles/PMC11320168/#note-ZOI240844-1-s https://pmc.ncbi.nlm.nih.gov/articles/PMC11320168/#note-ZOI240844-1-s

https://pubmed.ncbi.nlm.nih.gov/32828874/, https://pubmed.ncbi.nlm.nih.gov/29433851/, https://pubmed.ncbi.nlm.nih.gov/29075781/, https://pubmed.ncbi.nlm.nih.gov/34935591/ and https://pubmed.ncbi.nlm.nih.gov/23993357/ and department ICD-9 to ICD-10 conversion


BYPASS CORONARY ARTERY, TWO ARTERIES FROM RIGHT INTERNAL MAMMARY WITH NONAUTOLOGOUS TISSUE


DILATION OF INTRACRANIAL ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES,


NONDISPLACED FRACTURE OF OLECRANON PROCESS WITHOUT INTRAARTICULAR EXTENSION OF UNSPECIFIED


UNSPECIFIED FRACTURE OF UPPER END OF LEFT RADIUS, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE IIIA,


NONDISPLACED FRACTURE OF HEAD OF RIGHT RADIUS, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE IIIA,


NONDISPLACED FRACTURE OF HEAD OF UNSPECIFIED RADIUS, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE


NONDISPLACED FRACTURE OF NECK OF RIGHT RADIUS, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE IIIA,


NONDISPLACED FRACTURE OF NECK OF UNSPECIFIED RADIUS, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE


OTHER FRACTURE OF UPPER END OF LEFT RADIUS, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE IIIA, IIIB, OR


NONDISPLACED TRANSVERSE FRACTURE OF SHAFT OF LEFT ULNA, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE


DISPLACED OBLIQUE FRACTURE OF SHAFT OF RIGHT ULNA, SUBSEQUENT ENCOUNTER FOR CLOSED FRACTURE WITH


DISPLACED OBLIQUE FRACTURE OF SHAFT OF UNSPECIFIED ULNA, SUBSEQUENT ENCOUNTER FOR CLOSED


NONDISPLACED TRANSVERSE FRACTURE OF SHAFT OF LEFT RADIUS, SUBSEQUENT ENCOUNTER FOR CLOSED


DISPLACED OBLIQUE FRACTURE OF SHAFT OF UNSPECIFIED RADIUS, SUBSEQUENT ENCOUNTER FOR CLOSED


NONDISPLACED OBLIQUE FRACTURE OF SHAFT OF LEFT RADIUS, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE


DISPLACED SPIRAL FRACTURE OF SHAFT OF RADIUS, UNSPECIFIED ARM, SUBSEQUENT ENCOUNTER FOR OPEN


OTHER FRACTURE OF SHAFT OF RADIUS, UNSPECIFIED ARM, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE I


UNSPECIFIED PHYSEAL FRACTURE OF LOWER END OF ULNA, UNSPECIFIED ARM, SUBSEQUENT ENCOUNTER FOR


SALTER-HARRIS TYPE III PHYSEAL FRACTURE OF LOWER END OF ULNA-HARRIS TYPE III PHYSEAL FRACTURE OF LOWER


SALTER-HARRIS TYPE III PHYSEAL FRACTURE OF UPPER END OF RADIUS, UNSPECIFIED ARM, SUBSEQUENT


SALTER-HARRIS TYPE IV PHYSEAL FRACTURE OF UPPER END OF RADIUS, UNSPECIFIED ARM, SUBSEQUENT


SALTER-HARRIS TYPE I PHYSEAL FRACTURE OF LOWER END OF RADIUS, UNSPECIFIED ARM, SUBSEQUENT


SALTER-HARRIS TYPE II PHYSEAL FRACTURE OF LOWER END OF RADIUS, UNSPECIFIED ARM, SUBSEQUENT


SALTER-HARRIS TYPE IV PHYSEAL FRACTURE OF LOWER END OF RADIUS, LEFT ARM, SUBSEQUENT ENCOUNTER FOR


SALTER-HARRIS TYPE I PHYSEAL FRACTURE OF UPPER END OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR


SALTER-HARRIS TYPE I PHYSEAL FRACTURE OF LOWER END OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR


SALTER-HARRIS TYPE II PHYSEAL FRACTURE OF LOWER END OF UNSPECIFIED FEMUR, SEQUELA-HARRIS TYPE III


NONDISPLACED MIDCERVICAL FRACTURE OF LEFT FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE


DISPLACED FRACTURE OF BASE OF NECK OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE


UNSPECIFIED FRACTURE OF HEAD OF RIGHT FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE IIIA, IIIB,


UNSPECIFIED TROCHANTERIC FRACTURE OF RIGHT FEMUR, SUBSEQUENT ENCOUNTER FOR CLOSED FRACTURE WITH


DISPLACED INTERTROCHANTERIC FRACTURE OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN


DISPLACED SUBTROCHANTERIC FRACTURE OF RIGHT FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE I


NONDISPLACED SUBTROCHANTERIC FRACTURE OF LEFT FEMUR, INITIAL ENCOUNTER FOR OPEN FRACTURE TYPE IIIA,


NONDISPLACED TRANSVERSE FRACTURE OF SHAFT OF LEFT FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE


DISPLACED OBLIQUE FRACTURE OF SHAFT OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE


DISPLACED SPIRAL FRACTURE OF SHAFT OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR CLOSED FRACTURE


NONDISPLACED SPIRAL FRACTURE OF SHAFT OF LEFT FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE


NONDISPLACED COMMINUTED FRACTURE OF SHAFT OF LEFT FEMUR, SUBSEQUENT ENCOUNTER FOR CLOSED


DISPLACED SEGMENTAL FRACTURE OF SHAFT OF RIGHT FEMUR, INITIAL ENCOUNTER FOR OPEN FRACTURE TYPE I OR


NONDISPLACED UNSPECIFIED CONDYLE FRACTURE OF LOWER END OF UNSPECIFIED FEMUR, SUBSEQUENT


NONDISPLACED FRACTURE OF LATERAL CONDYLE OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN


DISPLACED SUPRACONDYLAR FRACTURE WITHOUT INTRACONDYLAR EXTENSION OF LOWER END OF RIGHT FEMUR,


NONDISPLACED SUPRACONDYLAR FRACTURE WITHOUT INTRACONDYLAR EXTENSION OF LOWER END OF LEFT


NONDISPLACED SUPRACONDYLAR FRACTURE WITH INTRACONDYLAR EXTENSION OF LOWER END OF UNSPECIFIED


UNSPECIFIED FRACTURE OF UNSPECIFIED FEMUR, SUBSEQUENT ENCOUNTER FOR OPEN FRACTURE TYPE I OR II WITH


SALTER-HARRIS TYPE III PHYSEAL FRACTURE OF LOWER END OF RIGHT FEMUR, SUBSEQUENT ENCOUNTER FOR


SALTER-HARRIS TYPE IV PHYSEAL FRACTURE OF LOWER END OF RIGHT FEMUR, SUBSEQUENT ENCOUNTER FOR


WEDGE COMPRESSION FRACTURE OF T5-T6 VERTEBRA, SUBSEQUENT ENCOUNTER FOR FRACTURE WITH DELAYED


UNSPECIFIED FRACTURE OF T5-T6 VERTEBRA, INITIAL ENCOUNTER FOR CLOSED FRACTURE-HARRIS TYPE IV PHYSEAL


Generic

FENTANYL CITRATE IN DEXTROSE 5% IN WATER/PF RX

Opioids

Oral Oral Oral Oral

Oral Oral

Oral Oral Oral Oral Oral

FENTANYL CITRATE/BUPIVACAINE HCL IN 0.9 % SODIUM CHLORIDE/PF RX Opioids Generic FENTANYL Opioids CITRATE/DROPERIDOL RX Generic Opioids FENTANYL CITRATE/PF RX Generic FENTANYL CITRATE/ROPIVACAINE HCL/SODIUM CHLORIDE Opioids 0.9%/PF RX Generic Opioids FENTANYL HCL RX Generic Opioids HYDROMORPHONE HCL RX Generic HYDROMORPHONE HCL IN Opioids 0.9 % SODIUM CHLORIDE Generic HYDROMORPHONE HCL IN 0.9 % SODIUM CHLORIDE/PF RX Opioids Generic HYDROMORPHONE HCL IN Opioids DEXTROSE 5 %-WATER/PF Generic HYDROMORPHONE HCL IN Opioids STERILE WATER/PF Generic HYDROMORPHONE HCL/BUPIVACAINE HCL IN Opioids 0.9% SODIUM CHLORIDE/PF RX Generic Opioids APOMORPHINE HCL Generic Opioids HYDROMORPHONE HCL/PF RX Generic HYDROMORPHONE HCL/ROPIVACAINE IN 0.9 % Opioids SODIUM CHLORIDE/PF Generic Opioids LEVORPHANOL TARTRATE RX Generic Opioids MEPERIDINE HCL Generic MEPERIDINE HCL IN 0.9 % Opioids SODIUM CHLORIDE Generic MEPERIDINE HCL IN 0.9 % Opioids SODIUM CHLORIDE/PF Generic MEPERIDINE HCL/ATROPINE Opioids SULFATE Generic Opioids MEPERIDINE HCL/PF RXGeneric MEPERIDINE Opioids HCL/PROMETHAZINE HCL RX Generic Opioids METHADONE HCL RX Generic METHADONE HYDROCHLORIDE IN 0.9 % Opioids SODIUM CHLORIDE RX Generic Opioids MORPHINE SULFATE RX Generic MORPHINE SULFATE IN 0.9 Opioids % SODIUM CHLORIDE Generic MORPHINE SULFATE IN 0.9 Opioids % SODIUM CHLORIDE/PF Generic MORPHINE SULFATE IN SODIUM CHLORIDE, ISO-Opioids OSMOTIC/PF RXGeneric MORPHINE SULFATE Opioids LIPOSOMAL/PF RX Generic MORPHINE SULFATE/DEXTROSE 5 % IN Opioids WATER Generic

MORPHINE SULFATE/DEXTROSE 5%-RX Opioids WATER/PF Generic MORPHINE SULFATE/NALTREXONE HCL RX Opioids Generic Opioids MORPHINE SULFATE/PF RX Generic Opioids OPIUM TINCTURE RXGeneric OPIUM/BELLADONNA Opioids ALKALOIDS RX Generic Opioids OXYMORPHONE HCL RX Generic PENTAZOCINE Opioids HCL/ACETAMINOPHEN RX Generic Opioids PENTAZOCINE HCL/ASPIRIN RX Generic PENTAZOCINE Opioids HCL/NALOXONE HCL RXGeneric Opioids PENTAZOCINE LACTATE RX Generic Opioids TAPENTADOL HCL RX Generic ACETAMINOPHEN WITH CODEINE PHOSPHATE RX Opioids Generic ASPIRIN/CODEINE PHOSPHATE Opioids Generic BUTALBITAL/ACETAMINOPH EN/CAFFEINE/CODEINE Opioids PHOSPHATE RX Generic RX Opioids CODEINE PHOSPHATE Generic CODEINE PHOSPHATE/BUTALBITAL/A Opioids SPIRIN/CAFFEINE RX Generic RXOpioids CODEINE SULFATE Generic CODEINE/ASPIRIN/SALICYLA MIDE/ACETAMINOPHEN/CA Opioids FFEINE Generic Opioids HYDROCODONE BITARTRATE RX Generic **HYDROCODONE** BITARTRATE/ACETAMINOPH Opioids EN Generic HYDROCODONE BITARTRATE/ACETAMINOPH **EN/DIETARY SUPPLEMENT** Opioids #11 Generic **HYDROCODONE** Opioids BITARTRATE/ASPIRIN RX Generic HYDROCODONE/IBUPROFE Opioids Ν Generic IBUPROFEN/OXYCODONE Opioids HCL RX Generic Opioids OXYCODONE HCL RX Generic OXYCODONE RXOpioids HCL/ACETAMINOPHEN Generic Opioids OXYCODONE HCL/ASPIRIN RX Generic OXYCODONE HCL/OXYCODONE Opioids TEREPHTHALATE/ASPIRIN RX Generic Opioids OXYCODONE MYRISTATE RX Generic OXYCODONE/ASPIRIN RX Opioids Generic TRAMADOL HCL RX Opioids Generic TRAMADOL Opioids HCL/ACETAMINOPHEN RX Generic TRAMADOL HCL/DIETARY SUPPLEMENT, MISC. CB.11 RX

Generic

Opioids


mergency Room

OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF A NEW PATIENT, WHICH REQUIRES THESE 3 KEY COMPONENTS: A PROBLEM FOCUSED HISTORY; A PROBLEM FOCUSED EXAMINATION; STRAIGHTFORWARD MEDICAL DECISION MAKING. COUNSELING AND/OR COORDINATION OF CARE WITH OTHER PHYSICIANS, OTHER QUALIFIED HEALTH CARE PROFESSIONALS, OR AGENCIES ARE PROVIDED CONSISTENT WITH THE NATURE OF THE PROBLEM(S) AND THE PATIENT'S AND/OR FAMILY'S NEEDS. USUALLY, THE PRESENTING PROBLEM(S) ARE SELF LIMITED OR MINOR. TYPICALLY, 10 MINUTES ARE SPENT FACE-TO-FACE WITH THE PATIENT AND/OR


| OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF A NEW PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND STRAIGHTFORWARD MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 15-29 MINUTES OF TOTAL TIME IS SPENT ON THE DATE OF THE ENCOUNTER. | No inpatient confinement claim |
|---|---|
| OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF A NEW PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND LOW LEVEL OF MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 30-44 MINUTES OF TOTAL TIME IS SPENT ON THE DATE OF THE | |
| ENCOUNTER. OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF A NEW PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND MODERATE LEVEL OF MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 45-59 MINUTES OF TOTAL TIME IS SPENT ON THE DATE OF THE FNCOLUTER. | No inpatient confinement claim No inpatient confinement claim |
| OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF A NEW PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND HIGH LEVEL OF MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 60-74 MINUTES OF TOTAL TIME IS SPENT ON THE DATE OF THE | · |
| ENCOUNTER. OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF AN ESTABLISHED PATIENT THAT MAY NOT REQUIRE THE PRESENCE OF A PHYSICIAN OR OTHER QUALIFIED HEALTH CARE PROFESSIONAL | No inpatient confinement claim No inpatient confinement claim |
| OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF AN ESTABLISHED PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND STRAIGHTFORWARD MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 10-19 MINUTES OF TOTAL TIME IS SPENT ON THE DATE OF THE ENCOUNTER. | No inpatient confinement claim |
| OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF AN ESTABLISHED PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND LOW LEVEL OF MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 20-29 MINUTES OF TOTAL TIME IS SPENT ON THE | · |
| DATE OF THE ENCOUNTER. OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF AN ESTABLISHED PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND MODERATE LEVEL OF MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 30-39 MINUTES OF TOTAL TIME IS SPENT ON THE | No inpatient confinement claim |
| DATE OF THE ENCOUNTER. OFFICE OR OTHER OUTPATIENT VISIT FOR THE EVALUATION AND MANAGEMENT OF AN ESTABLISHED PATIENT, WHICH REQUIRES A MEDICALLY APPROPRIATE HISTORY AND/OR EXAMINATION AND HIGH LEVEL OF MEDICAL DECISION MAKING. WHEN USING TIME FOR CODE SELECTION, 40-54 MINUTES OF TOTAL TIME IS SPENT ON THE | No inpatient confinement claim |
| DATE OF THE ENCOUNTER. | No inpatient confinement claim |

| | | NUCC Taxonomy |
|---|---|---|
| Endocrinologist visit | 207RE0101X | Code 1 |
| Endocrinologist visit | 207RE0101X | NUCC Taxonomy<br>Code 2<br>Provider category |
| Cardiologist visit | 0400 | code Provider category |
| Cardiologist visit | 0401 | code Provider category |
| Cardiologist visit | 0402 | code Provider category |
| Cardiologist visit | 0403 | code<br>Provider category |
| Cardiologist visit | 0404 | code<br>Provider category |
| Cardiologist visit | 0405 | code<br>Provider category |
| Cardiologist visit | 0407 | code<br>Provider category |
| Cardiologist visit | 0408 | code<br>Provider category |
| Cardiologist visit | 0409 | code<br>Provider category |
| Cardiologist visit | 0410 | code<br>Provider category |
| Cardiologist visit | 0411 | code<br>Provider category |
| Cardiologist visit | 0412 | code<br>Provider category |
| Cardiologist visit | 0416 | code<br>Provider category |
| Cardiologist visit | 1108 | code<br>Provider category |
| Cardiologist visit | 1123 | code<br>Provider category |
| Cardiologist visit | 1135 | code<br>Provider category |
| Cardiologist visit | 1162 | code<br>Provider category |
| Cardiologist visit | 1212 | code<br>Provider category |
| Cardiologist visit | 1582 | code<br>Provider category |
| Cardiologist visit | 1629 | code<br>Provider category |
| Cardiologist visit | 1728 | code<br>Provider category |
| Cardiologist visit | 1856 | code<br>Provider category |
| Cardiologist visit | 1947 | code<br>Provider category |
| Cardiologist visit | 2653 | code<br>Provider category |
| Cardiologist visit | 2810 | code<br>Provider category |
| Cardiologist visit | 3073 | code<br>Provider category |
| Cardiologist visit | 3137 | code<br>Provider category |
| Cardiologist visit | 3249 | code<br>Provider category |
| Cardiologist visit | 3534 | code |

| Cardiologist visit | 4113 | Provider category code |
|---|---|---|
| Cardiologist visit | 4163 | Provider category code |
| Cardiologist visit | 4622 | Provider category code |
| Cardiologist visit | 4644 | Provider category code |
| Cardiologist visit | 5726 | Provider category code |
| Cardiologist visit | 5742 | Provider category code |
| Cardiologist visit | 5761 | Provider category code |
| Cardiologist visit | 5771 | Provider category code |
| Cardiologist visit | 6593 | Provider category code |
| Cardiologist visit | 6616 | Provider category<br>code |
| Cardiologist visit | 6887 | Provider category<br>code<br>Provider category |
| Cardiologist visit | 7034 | code Provider category |
| Cardiologist visit | 7749 | code<br>NUCC Taxonomy |
| Cardiologist visit | 207RC0000X | Code 1 NUCC Taxonomy |
| Cardiologist visit | 207RC0000X | Code 2 Provider category |
| Internal medicine/family medicine visit | 0334 | code<br>Provider category |
| Internal medicine/family medicine visit | 0335 | code<br>Provider category |
| Internal medicine/family medicine visit | 0336 | code<br>Provider category |
| Internal medicine/family medicine visit | 0337 | code<br>Provider category |
| Internal medicine/family medicine visit | 0338 | code<br>Provider category |
| Internal medicine/family medicine visit | 0339 | code<br>Provider category |
| Internal medicine/family medicine visit | 0340 | code<br>Provider category |
| Internal medicine/family medicine visit | 0341 | code<br>Provider category |
| Internal medicine/family medicine visit | 0342 | code<br>Provider category |
| Internal medicine/family medicine visit | 1133 | code<br>Provider category |
| Internal medicine/family medicine visit | 1419 | code<br>Provider category |
| Internal medicine/family medicine visit | 1673 | code<br>Provider category |
| Internal medicine/family medicine visit | 1697 | code<br>Provider category |
| Internal medicine/family medicine visit | 1860 | code<br>Provider category |
| Internal medicine/family medicine visit Internal medicine/family medicine visit | 1864<br>2050 | code<br>Provider category<br>code |
| internal medicine/laminy medicine visit | 2030 | code |

| | | Drouider entegen |
|------------------------------------------|------|---------------------------|
| Internal medicine/family medicine visit | 2280 | Provider category code |
| Internal medicine/family medicine visit | 2302 | Provider category code |
| Internal medicine/family medicine visit | 2313 | Provider category code |
| median medicine, idinity medicine visit | 2313 | Provider category |
| Internal medicine/family medicine visit | 2314 | code |
| Internal medicine/family medicine visit | 2373 | Provider category code |
| Internal medicine/family medicine visit | 2610 | Provider category code |
| Internal medicine/family medicine visit | 2842 | Provider category code |
| Internal medicine/family medicine visit | 3268 | Provider category code |
| Internal medicine/family medicine visit | 3755 | Provider category code |
| Internal medicine/family medicine visit | 4641 | Provider category code |
| Internal medicine/family medicine visit | 4876 | Provider category code |
| internal medicine/laminy medicine visit | 4870 | Provider category |
| Internal medicine/family medicine visit | 5724 | code |
| Internal medicine/family medicine visit | 5736 | Provider category code |
| | | Provider category |
| Internal medicine/family medicine visit | 5829 | code<br>Provider category |
| Internal medicine/family medicine visit | 5991 | code<br>Provider category |
| Internal medicine/family medicine visit | 5998 | code |
| Internal medicine/family medicine visit | 0308 | Provider category code |
| internal medicine, family medicine visit | 0308 | Provider category |
| Internal medicine/family medicine visit | 0311 | code |
| Internal medicine/family medicine visit | 0312 | Provider category code |
| Internal medicine/family medicine visit | 0313 | Provider category code |
| Internal medicine/family medicine visit | 0314 | Provider category code |
| | | Provider category |
| Internal medicine/family medicine visit | 0316 | code<br>Provider category |
| Internal medicine/family medicine visit | 0317 | code<br>Provider category |
| Internal medicine/family medicine visit | 0318 | code |
| Internal medicine/family medicine visit | 0319 | Provider category code |
| Internal medicine/family medicine visit | 0326 | Provider category code |
| • | | Provider category |
| Internal medicine/family medicine visit | 0327 | code<br>Provider category |
| Internal medicine/family medicine visit | 0329 | code |
| Internal medicine/family medicine visit | 0330 | Provider category code |
| • | 3330 | Provider category |
| Internal medicine/family medicine visit | 0331 | code<br>Provider category |
| Internal medicine/family medicine visit | 0332 | code |

| Internal medicine/family medicine visit | 0333 | Provider category code |
|---|---|---|
| Internal medicine/family medicine visit | 1046 | Provider category code |
| Internal medicine/family medicine visit | 1113 | Provider category code |
| Internal medicine/family medicine visit | 1127 | Provider category code |
| Internal medicine/family medicine visit | 1643 | Provider category code |
| Internal medicine/family medicine visit | 1646 | Provider category code |
| Internal medicine/family medicine visit | 1694 | Provider category<br>code<br>Provider category |
| Internal medicine/family medicine visit | 1721 | code Provider category |
| Internal medicine/family medicine visit | 1785 | code Provider category |
| Internal medicine/family medicine visit | 1832 | code<br>Provider category |
| Internal medicine/family medicine visit | 1865 | code Provider category |
| Internal medicine/family medicine visit | 1927 | code<br>Provider category |
| Internal medicine/family medicine visit | 2068 | code<br>Provider category |
| Internal medicine/family medicine visit | 2189 | code<br>Provider category |
| Internal medicine/family medicine visit | 2219 | code<br>Provider category |
| Internal medicine/family medicine visit | 2233 | code<br>Provider category |
| Internal medicine/family medicine visit | 2286 | code<br>Provider category |
| Internal medicine/family medicine visit | 2340 | code<br>Provider category |
| Internal medicine/family medicine visit | 2354 | code<br>Provider category |
| Internal medicine/family medicine visit | 2378 | code<br>Provider category |
| Internal medicine/family medicine visit | 2403 | code<br>Provider category |
| Internal medicine/family medicine visit | 2574 | code<br>Provider category |
| Internal medicine/family medicine visit Internal medicine/family medicine visit | 2614<br>2615 | code<br>Provider category |
| Internal medicine/family medicine visit | 2628 | code<br>Provider category<br>code |
| Internal medicine/family medicine visit | 2644 | Provider category<br>code |
| Internal medicine/family medicine visit | 2790 | Provider category |
| Internal medicine/family medicine visit | 2835 | Provider category code |
| Internal medicine/family medicine visit | 2978 | Provider category code |
| Internal medicine/family medicine visit | 2996 | Provider category code |
| Internal medicine/family medicine visit | 3122 | Provider category code |

| Internal medicine/family medicine visit | 3777 | Provider category code |
|---|---|---|
| Internal medicine/family medicine visit | 3787 | Provider category code |
| Internal medicine/family medicine visit | 4362 | Provider category code |
| Internal medicine/family medicine visit | 4645 | Provider category code |
| Internal medicine/family medicine visit | 4648 | Provider category code |
| Internal medicine/family medicine visit | 5063 | Provider category code |
| Internal medicine/family medicine visit | 5683 | Provider category code |
| Internal medicine/family medicine visit | 5696 | Provider category code |
| Internal medicine/family medicine visit | 5706 | Provider category<br>code |
| Internal medicine/family medicine visit | 5732 | Provider category<br>code |
| Internal medicine/family medicine visit | 5774 | Provider category<br>code<br>Provider category |
| Internal medicine/family medicine visit | 5781 | code<br>Provider category |
| Internal medicine/family medicine visit | 5994 | code<br>Provider category |
| Internal medicine/family medicine visit | 6000 | code<br>Provider category |
| Internal medicine/family medicine visit | 7017 | code<br>Provider category |
| Internal medicine/family medicine visit | 7592 | code<br>Provider category |
| Internal medicine/family medicine visit | 7777 | code<br>Provider category |
| Internal medicine/family medicine visit | 7792 | code<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207Q00000X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QA0000X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QA0401X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QA0505X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QB0002X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QG0300X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit | 207QH0002X | Code 1<br>NUCC Taxonomy |
| Internal medicine/family medicine visit Internal medicine/family medicine visit | 207QS0010X<br>207QS1201X | Code 1<br>NUCC Taxonomy<br>Code 1 |
| Internal medicine/family medicine visit | 207Q31201X<br>207Q00000X | NUCC Taxonomy<br>Code 2 |
| Internal medicine/family medicine visit | 207Q00000X<br>207QA0000X | NUCC Taxonomy<br>Code 2 |
| Internal medicine/family medicine visit | 207QA0401X | NUCC Taxonomy<br>Code 2 |
| Internal medicine/family medicine visit | 207QA0505X | NUCC Taxonomy<br>Code 2 |
| . , | • | |


| ECHOCAR | IRDIOGRAPHY, TRANSESOPHAGEAL (TEE) FOR GUIDANCE OF A TRANSCATHETER INTRACARDIAC OR GREAT |
|---|---|
| VESSEL(S) | S) STRUCTURAL INTERVENTION(S) (EG,TAVR, TRANSCATHETER PULMONARY VALVE REPLACEMENT, MITRAL |
| VALVE RE | EPAIR, PARAVALVULAR REGURGITATION REPAIR, LEFT ATRIAL APPENDAGE OCCLUSION/CLOSURE, |
| VENTRIC | CULAR SEPTAL DEFECT CLOSURE) (PERI-AND INTRA-PROCEDURAL), REAL-TIME IMAGE ACQUISITION AND |
| DOCUME | ENTATION, GUIDANCE WITH QUANTITATIVE MEASUREMENTS, PROBE MANIPULATION, INTERPRETATION, |
| AND REP | PORT, INCLUDING DIAGNOSTIC TRANSESOPHAGEAL ECHOCARDIOGRAPHY AND, WHEN PERFORMED, |


GENERAL HEALTH PANEL THIS PANEL MUST INCLUDE THE FOLLOWING: COMPREHENSIVE METABOLIC PANEL

| DIGITIZATION OF FILM RADIOGRAPHIC IMAGES WITH COMPUTER ANALYSIS FOR LESION DETECTION, OR COMPUTER |
|---|
| ANALYSIS OF DIGITAL MAMMOGRAM FOR LESION DETECTION, AND FURTHER PHYSICIAN REVIEW FOR |
| INTERPRETATION, DIAGNOSTIC MAMMOGRAPHY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY |

